# **Clinical Study Protocol**

# **Title Page**

| | I |
|---|---|
| Clinical Study Protocol Title: | A Phase II, Multicenter, Open Label Study of<br>Bintrafusp alfa (M7824) Monotherapy in<br>Participants with HMGA2-expressing Triple<br>Negative Breast Cancer |
| Study Number: | MS200647_0020 |
| Protocol Version: | 06 July 2021 / Version 2.0 |
| Merck Compound Number: | M7824 |
| Study Phase: | Phase II |
| Short Title: | Bintrafusp alfa in HMGA2-expressing Triple<br>Negative Breast Cancer |
| Coordinating Investigator: | PPD , PPD |
| | PPD |
| Sponsor Name and Legal Registered Address: | Sponsor: Affiliates of Merck KGaA, Darmstadt, Germany |
| Audi ess. | For all countries, except the US and Canada: Merck Healthcare KGaA, Darmstadt, Germany An affiliate of Merck KGaA, Darmstadt, Germany Frankfurter Str. 250 64293 Darmstadt, Germany |
| | In the US and Canada: EMD Serono Research & Development Institute, Inc. An affiliate of Merck KGaA, Darmstadt, Germany 45A Middlesex Turnpike Billerica, MA, 01821, USA |
| Regulatory Agency Identifying Numbers: | EudraCT: 2019-004833-18 |

## **Protocol Amendment Summary of Changes**

## **Protocol History**

| Version Number | Туре | Version Date |
|----------------|-------------------|--------------|
| 1.0 | Original Protocol | 11-Jul-2019 |
| 2.0 | Global Amendment | 06-Jul-2021 |

## Protocol Version 2.0 (06-Jul-2021)

This amendment is substantial based on the criteria in Article 10(a) of Directive 2001/20/EC of the European Parliament and the Council of the European Union.

#### **Overall Rationale for the Amendment**

The primary purpose of this amendment is to update the risk classification.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Title Page | Revised "Amendment Number" row<br>Removed "Medical Responsible" field<br>Removed "Protocol Version",<br>"Replaces Version", "Approval Date",<br>and "Medical Monitor Contact<br>Information" rows | To be consistent with current Sponsor protocol template (Version 15) |
| 1.3 Schedule of Activities | <ul> <li>Text updated to clarify limited disease history information to be collected at prescreening</li> <li>Text is updated to clarify Intervention Period window of ±3 days is not applicable for tumor evaluations</li> </ul> | To clarify study procedures. |
| 2.3 Benefit/Risk<br>Assessment | Text updated to address risk reclassification | The risk reclassification was based on indepth analysis of a pooled safety dataset of N = 765 participants who received bintrafusp alfa monotherapy at 1200 mg Q2W. |
| 5. Study Population<br>Appendix 2 | Edits related to informed consent procedure | To be consistent with current Sponsor protocol template (Version 15) |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 6.9 Management of<br>Adverse Events of<br>Special Interest<br>Appendix 4 | Risk reclassification has been done and the list of events has been updated accordingly | |
| 6.9.1 Infusion-related<br>Reactions Including<br>Hypersensitivity | Infusion-related reactions are reclassified from "important identified risk" to "identified risk" for bintrafusp alfa | The risk reclassification was based on in- |
| 6.9.1, Table 5. Treatment<br>Modification of Bintrafusp<br>alfa for Symptoms of<br>Infusion Related<br>Reactions Including<br>Immediate<br>Hypersensitivity | Additional details of treatment modifications for severe or life-threatening reactions have been added. | depth analysis of a pooled safety dataset of N = 765 participants who received bintrafusp alfa monotherapy at 1200 mg Q2W as reflected in Investigator's Brochure, V7.0. |
| 6.9.2 Immune-related<br>Adverse Events | Risk reclassification has been done and the list of events has been updated accordingly | |
| 6.9.3. TGF-β Inhibition<br>Mediated Skin Reactions | Skin Adverse Events have been renamed as TGF-β Inhibition Mediated Skin Reactions | |
| 6.9.4 Anemia | Term "treatment-related anemia<br>events" has been revised to "anemia"<br>and reclassified from "important<br>potential risk" to "important identified<br>risk" for bintrafusp alfa | |
| 6.9.5 Bleeding Events | Bleeding events are reclassified from<br>"potential risk" to "important identified<br>risk" for bintrafusp alfa | |
| 6.9.6.1 Impaired Wound<br>Healing | The risk name "Alterations in Wound Healing or Repair of Tissue Damage" has been changed to "Impaired Wound Healing" | |
| 7.3 Lost to Follow-up | Edits are done related to Lost to Follow-up information | To be consistent with current Sponsor protocol template (Version 15) |
| 8.1 Efficacy Assessments and Procedures | Text has been updated to suggest caution in diagnosis of disease progression based solely on nodal enlargement within 8 weeks of coronavirus vaccination. | To clarify study procedures. |

Note: Minor changes have been performed throughout the protocol to address consistency pertaining to major changes made in the protocol or to add further clarity and precision.

#### - Confidential -

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its subsidiaries. It is intended for restricted use only and may not – in full or part – be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany, or its subsidiary. Copyright © 2021 by Merck KGaA, Darmstadt, Germany, or its subsidiary. All rights reserved.

# **Table of Contents**

| Title Page | 1 |
|---|---|
| Table of Contents | 4 |
| 1 | Protocol Summary8 |
| 1.1 | Synopsis8 |
| 1.2 | Schema11 |
| 1.3 | Schedule of Activities |
| 2 | Introduction |
| CC | |
| 2.2 | Background |
| 2.3 | Benefit/Risk Assessment |
| 3 | Objectives and Endpoints |
| 4 | Study Design31 |
| 4.1 | Overall Design |
| 4.2 | Scientific Rationale for Study Design |
| 4.3 | Justification for Dose |
| 4.4 | End of Study Definition |
| 5 | Study Population |
| 5.1 | Inclusion Criteria |
| 5.2 | Exclusion Criteria |
| 5.3 | Lifestyle Considerations |
| 5.4 | Screen Failures |
| 6 | Study Intervention(s) |
| 6.1 | Study Intervention(s) Administration |
| 6.2 | Study Intervention(s) Preparation, Handling, Storage, and Accountability |
| 6.3 | Measures to Minimize Bias: Study Intervention Assignment and Blinding |
| 6.3.1 | Study Intervention Assignment |
| 6.3.2 | Blinding41 |
| 6.4 | Study Intervention Compliance41 |
| 6.5 | Concomitant Therapy42 |
| 6.5.1 | Permitted Medicines |

| 6.5.2 | Prohibited Medicines | 43 |
|---|---|---|
| 6.5.3 | Other Interventions | 43 |
| 6.6 | Dose Selection and Modification. | 44 |
| 6.7 | Study Intervention After the End of the Study | 44 |
| 6.8 | Special Precautions | 44 |
| 6.9 | Management of Adverse Events of Special Interest | 46 |
| 6.9.1 | Infusion-related Reactions Including Hypersensitivity | 47 |
| 6.9.2 | Immune-related Adverse Events | 49 |
| 6.9.3 | TGF-β Inhibition Mediated Skin Reactions | 51 |
| 6.9.4 | Anemia | 52 |
| 6.9.5 | Bleeding Events | 53 |
| 6.9.5.1 | Mucosal/Non-Tumor Bleeding | 54 |
| 6.9.5.2 | Tumor Bleeding | 54 |
| 6.9.6 | Other Potential Risks | 54 |
| 6.9.6.1 | Impaired Wound Healing | 54 |
| 6.9.6.2 | Embryofetal Toxicity | 54 |
| 7 | Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal | 55 |
| 7.1 | Discontinuation of Study Intervention | 55 |
| 7.1.1 | Temporary Discontinuation | 56 |
| 7.1.2 | Rechallenge | 56 |
| 7.1.2.1 | Reinitiation | 56 |
| 7.1.3 | Treatment Beyond Progression | 57 |
| 7.1.3.1 | Treatment Beyond Initial Progression | 57 |
| 7.1.3.2 | Treatment Beyond Confirmed Progression | 57 |
| 7.1.3.3 | Continuation of Study Intervention After Local Treatment of Disease Progression | 57 |
| 7.2 | Participant Discontinuation/Withdrawal from the Study | 58 |
| 7.3 | Lost to Follow-Up | 58 |
| 8 | Study Assessments and Procedures | 59 |
| 8.1 | Efficacy Assessments and Procedures | 59 |
| 8.2 | Safety Assessments and Procedures | 60 |
| 8.2.1 | Physical Examinations | 61 |

| 8.2.2 | Vital Signs61 |
|---|---|
| 8.2.3 | Electrocardiograms |
| 8.2.4 | Clinical Safety Laboratory Assessments |
| 8.3 | Adverse Events and Serious Adverse Events |
| 8.3.1 | Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information |
| 8.3.2 | Method of Detecting Adverse Events and Serious Adverse Events63 |
| 8.3.3 | Follow-up of Adverse Events and Serious Adverse Events63 |
| 8.3.4 | Regulatory Reporting Requirements for Serious Adverse Events64 |
| 8.3.5 | Pregnancy |
| 8.4 | Treatment of Overdose |
| 8.5 | Pharmacokinetics |
| 8.6 | Pharmacodynamics |
| 8.7 | Pharmacogenetics |
| 8.8 | Biomarkers |
| 8.9 | Immunogenicity Assessments |
| C | CCI |
| 9.1 | Statistical Hypotheses |
| 9.2 | Sample Size Determination69 |
| 9.3 | Populations for Analyses |
| 9.4 | Statistical Analyses |
| 9.4.1 | Efficacy Analyses |
| 9.4.2 | Safety Analyses |
| 9.4.3 | Other Analyses |
| 9.4.4 | Sequence of Analyses |
| 10 | References |
| 11 | Appendices |
| Appendix 1 | Abbreviations |
| Appendix 2 | Study Governance |
| Appendix 3 | Contraception89 |
| Appendix 4 | Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting91 |
| Appendix 5 | The Recommendations for irAE Management95 |

| Appendix 6 | Clinical Laboratory Tests |
|---|---|
| Appendix 7 | Prohibited Traditional Chinese Medicines |
| Appendix 8 | Pharmacogenetics |
| Appendix 9 | Protocol Amendment History |
| Appendix 10 | Sponsor Signature Page |
| Appendix 11 | Coordinating Investigator Signature Page |
| Appendix 12 | Principal Investigator Signature Page140 |
| List of Tables | |
| Table 1 | Schedule of Activities |
| Table 2 | Bintrafusp alfa Pharmacokinetic, Immunogenicity Sampling25 |
| Table 3 | Study Objectives and Endpoints30 |
| Table 4 | Study Intervention40 |
| Table 5 | Treatment Modification of Bintrafusp alfa for Symptoms of Infusion-Related Reactions Including Hypersensitivity48 |
| Table 6 | Evaluation Guidance of Suspected Anemia Adverse Events53 |
| Table 7 | Pharmacokinetic Parameters 66 |
| Table 8 | Biomarkers Overview |
| Table 9 | Confidence Intervals for Different Objective Response Rates70 |
| Table 10 | Analysis Populations |
| Table 11 | Statistical Analysis Methods for Efficacy Analysis |
| Table 12 | Safety Endpoints and Statistical Analysis Methods74 |
| Table 13 | Protocol-Required Clinical Laboratory Assessments |
| List of Figures | |
| Figure 1 | Study Design Diagram |
| Figure 2 | Bintrafusp alfa in Participants with TNBC by HMGA2 Expression in Study EMR200647-001 - Best Change in Target Lesions from Baseline Assessed by Investigator |

## 1 Protocol Summary

## 1.1 Synopsis

**Protocol Title:** A Phase II, Multicenter, Open Label Study of Bintrafusp alfa (M7824) Monotherapy in Participants with HMGA2-expressing Triple Negative Breast Cancer

**Short Title:** Bintrafusp alfa in HMGA2-expressing Triple Negative Breast Cancer

#### **Rationale:**

Triple negative breast cancer (TNBC) is an aggressive subtype of breast cancer that is defined by the lack of protein expression of estrogen receptor, lack of protein expression of the progesterone receptor, and the absence of human epidermal growth factor receptor 2 (HER2) protein overexpression. Of the estimated 1 million cases of breast cancer diagnosed annually worldwide, more than 170,000 are TNBC. The prognosis with standard chemotherapy has been poor and recent studies using checkpoint inhibitor monotherapy in previously treated TNBC patients have also been disappointing. However, interest in using immunotherapy in TNBC is growing since the recent encouraging data of the programmed death-ligand 1 (PD-L1) inhibitor atezolizumab in combination with nab-paclitaxel, in treatment-naïve PD-L1 positive TNBC became available, which led to the first immunotherapy approval in this disease.

Bintrafusp alfa monotherapy has shown promising clinical activity in participants with TNBC in the expansion cohort of the Phase I Study EMR200647-001. In Study EMR200647-001, a retrospective analysis signaled the potential for bintrafusp alfa to have considerable efficacy specifically in TNBC participants with tumors expressing high levels of High Mobility Group AT-Hook 2 (HMGA2), a molecule downstream of the transforming growth factor- $\beta$  (TGF- $\beta$ ) signaling pathway.

The purpose of this study is to prospectively investigate and confirm this efficacy signal in tumors expressing high levels of HMGA2.

## **Objectives and Endpoints:**

| Objectives | Endpoints (Outcome Measures) |
|---|---|
| Primary | |
| To evaluate clinical efficacy of bintrafusp alfa in<br>participants with TNBC with high HMGA2<br>expression, based on ORR | Confirmed objective response according to RECIST 1.1 assessed by an IRC |
| Secondary | |
| To evaluate clinical efficacy of bintrafusp alfa<br>based on DOR | DOR according to RECIST 1.1 assessed by an IRC |
| To evaluate clinical efficacy of bintrafusp alfa<br>based on DRR | Durable response of at least 6 months assessed by an IRC |
| To evaluate clinical efficacy based on PFS | PFS according to RECIST 1.1 assessed by an IRC |
| To evaluate ORR, DOR, DRR, and PFS by<br>Investigator read | Objective response, DOR, DRR, and PFS according to<br>RECIST 1.1 as assessed by the Investigator |
| To evaluate clinical efficacy based on OS | • OS |
| To evaluate clinical safety of bintrafusp alfa | Occurrence of TEAEs and treatment-related AEs including AEs of special interest |
| To characterize the PK profile of bintrafusp alfa | The concentration observed immediately at the end of infusion (C <sub>EOI</sub> ) of bintrafusp alfa |
| | The concentration observed immediately before next dosing (corresponding to predose or trough concentration [Ctrough] for multiple dosing) of bintrafusp alfa |
| To characterize the immunogenicity of bintrafusp alfa | Immunogenicity of bintrafusp alfa as measured by ADA assay from Screening through Safety Follow-up Visit up to 28 days after last treatment |

ADA=antidrug antibody, AE=adverse event, DOR=duration of response, DRR=durable response rate, HMGA2=High Mobility Group AT-Hook 2, IRC=Independent Review Committee, ORR=objective response rate, OS=overall survival, PFS=progression-free survival, PK=pharmacokinetic, RECIST 1.1=Response Evaluation Criteria in Solid Tumors Version 1.1, TEAE=Treatment-emergent adverse event, TNBC=Triple negative breast cancer.

### **Overall Design:**

This is a Phase II, multicenter, single-arm, open label study to evaluate bintrafusp alfa monotherapy in participants with TNBC who express high levels of HMGA2 as determined by a centralized reverse transcriptase-polymerase chain reaction (RT-PCR) test with predefined cutoff. Participants must have progressed during or after first-line of chemotherapy.

The study plans to enroll approximately 29 eligible participants globally with competitive enrollment.

## The study includes:

- Prescreening (a Prescreening informed consent form will be used for HMGA2 biomarker analysis and collection of baseline clinical history). Positive HMGA2 test results on tumor tissue is required to enter formal study Screening.
- Up to 28-day Screening period.
- Treatment with bintrafusp alfa at a dose of 1200 mg intravenously once every 2 weeks until confirmed progressive disease (PD), unacceptable toxicity, study withdrawal, or death.
- In the case of PD, treatment may continue past the initial determination of PD or confirmed PD if the participant's performance status has remained at least stable, and if in the opinion of the Investigator, the participant will benefit from continued treatment and if other criteria are fulfilled as outlined in the protocol.
- In the case of stable disease, partial response, or complete response, treatment should be continued until the end of 24 months. If the Investigator believes that a participant will benefit from treatment beyond 24 months, it may be permissible after discussion with the Medical Monitor and the Sponsor Medical Responsible.
- Safety Follow-up will continue until 12 weeks after the last dose of bintrafusp alfa. The 12-week Safety Follow-up is allowed to be conducted via telephone calls or patient chart reviews unless there is medical necessity requiring a clinical visit.
- Long-term Follow-up for progression and survival should be performed every 12 weeks after the Safety Follow-up according to the Schedule of Activities. Long-term Follow-up should be performed by patient chart reviews or telephone calls unless a clinical visit is indicated.

## **Number of Participants:**

The planned total sample size is 29 female participants to address the primary and other efficacy objectives, safety assessments, and evaluation of the clinical utility of the RT-PCR-based assay for HMGA2.

Assuming a true objective response rate of 30%, the probability to observe a lower bound of the exact 95% confidence interval above 10% (the benchmark for clinically non-relevant effect) would be 81% when analyzing 29 participants.

## **Study Intervention Groups and Duration:**

The planned maximum study duration for a participant is estimated to be up to 24 months (in certain instances, this duration may be lengthened if it is in the best interest of the participant to continue further treatment). This includes a 28-day Screening period (decision will be made in this period for participants' study inclusion if all eligibility criteria are met); a treatment duration until confirmed PD, unacceptable toxicity, study withdrawal or death occurs, a 28-day Safety Follow-up Visit, a 12-week Safety Follow-up phone call after the last dose of bintrafusp alfa, and a Long-term Follow-up (performed every 12 weeks after the Safety Follow-up).

## **Involvement of Special Committee(s): Yes**

The Independent Review Committee (IRC) will be involved in the study. The role of the IRC will be to review radiographic image findings, physical findings, and other clinical data for the determination of the best overall response (objective response) and date of disease progression for each participant. The full membership, mandate, and processes of the IRC will be detailed in the IRC charter.

## 1.2 Schema

This is a Phase II, multicenter, single-arm, open label study to evaluate bintrafusp alfa monotherapy in participants with TNBC expressing high levels of HMGA2 and who have progressed during or after first-line of chemotherapy.

Figure 1 Study Design Diagram



DOR=duration of response, DRR=durable response rate, HMGA2=High Mobility Group AT-Hook 2, IV=intravenous, N=number of participants, OS=overall survival, PFS=progression-free survival, Q2W=every 2 weeks.

### 1.3 Schedule of Activities

The Schedule of Activities is provided in Table 1. The bintrafusp alfa pharmacokinetic and immunogenicity sampling time points are provided in Table 2.

Table 1Schedule of Activities

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventio<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | reatment Safety | | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within 7 Days of | (± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| | Administrative Procedures | | | | | | | | | | | | | | | | |
| Written<br>informed<br>consent | Xª | Х | | | | | | | | | | | | | | | Screening tests performed as part of routine care prior to informed consent signed will be accepted if they are within 28-day Screening window (see Section 5.4). a: Prescreening ICF will be used to determine the main study eligibility criteria ahead of full Screening procedures (see Section 4.1). |
| Inclusion/<br>exclusion<br>criteria/<br>Enrollment (if<br>eligible) | | X | Х | | | | | | | | | | | | | | , |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioi<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | ety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat<br>ment | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | of or Within 7 Days of | (± 5 Days)<br>After Last | (± 2<br>Weeks) | 12<br>Weeks | |
| | | Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | Treatment | After Last<br>Treatment | (± 2<br>Weeks) | |
| Demographic<br>data | X | Xp | | | | | | | | | | | | | | | See Appendix 2. b: Demographic data collected during Prescreening should be verified and updated (if indicated) at Screening Visit. |
| Medical history | Xc | X | | | | | | | | | | | | | | | See Appendix 2. c: Part of the Disease History should be collected during Prescreening. The remaining Disease History and the full Medical History should be collected only if the participant passes prescreening. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventio<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | ety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | of or Within 7 Days of | (± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | After Last<br>Treatment | After Last | (± 2 | |
| Prior<br>anticancer<br>drug/radio<br>therapy<br>/procedures for<br>baseline visit | X | Xq | | | | | | | | | | | | | | | Prior anticancer procedures and therapies should at least include prior therapy, prior diagnosis of premalignant lesions and treatments, surgical resection and recurrence, and details on anticancer treatments, treatment duration, and treatment responses. d: Prior therapy collected during Prescreening should be verified and updated (if indicated) at Screening Visit. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | vention<br>(± 3 da | | d | | | End-of-<br>Treatment<br>Visit | | ety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to<br>Treat | V1<br>W1 | V2<br>W3 | V3<br>W5 | V4<br>W7 | V5<br>W9 | V6<br>W11 | V7<br>W13 | V8<br>W15 | V9<br>W17 | Until | On the Day of or Within | 28 Days<br>(± 5 Days) | 12 Weeks<br>(± 2 | Every<br>12 | |
| | | ment<br>Assign<br>ment | | D15 | D29 | D43 | D57 | | D85 | D99 | D113 | PD | 7 Days of Decision to Discontinue | After Last<br>Treatment | Weeks)<br>After Last<br>Treatment | | |
| Documentation of concomitant medication and procedures | | X | X | X | X | X | X | Х | Х | X | X | Q2W | X | X | Xe | | e: The 12-week Safety Follow-up and Long-term Follow-up may be conducted via telephone calls or patient chart reviews as necessary unless there is medical necessity requiring. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | vention<br>(± 3 da | n Perio<br>lys) | od | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | to<br>Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within<br>7 Days of | (± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| | | | | | | | | Tumo | r Biops | sies/Ar | chival 1 | Tissue C | Collection | | | | |
| Tumor tissue collection <sup>f</sup> | X | Xţ | | Xf | | | | | | | | | Xf | | | | See Section 8.8. Archival or fresh tumor tissue during Prescreening period is required for HMGA2 testing (see Section 4.1 and 8.8). f: Optional fresh biopsies during Screening, at W3 and End-of-Treatment Visit (excluding bone biopsies) may be tested for CCI biomarkers (see Section 8.8). Tissue from unscheduled procedures may also be submitted. |
| | | | 1 | 1 | | 1 | | | ntrafus | p alfa | | dminist | ration | | | | |
| Bintrafusp alfa administration | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Q2W | | | | | See Section 4.1 for treatment duration. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioi<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 20 Davis | 12 Weeks | Every | |
| | | to<br>Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within<br>7 Days of | 28 Days<br>(± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| | | | | | | | | | S | afety A | ssessr | nents | | | | | |
| Documentation of AEs | Xa | X | X | X | X | X | X | X | X | X | X | Q2W | X | X | Xh | | See Section 8.3 and Appendix 4 for definition of AE reporting period and follow-up. g: During Prescreening, only AEs associated with study procedures should be recorded. h: The 12-week Safety Follow-up and Long-term Follow-up may be conducted via telephone calls or patient chart reviews as necessary unless there is medical necessity requiring a clinical visit. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioi<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | ety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within 7 Days of | (± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| Physical<br>examination | | Х | X | X | X | X | X | X | X | X | X | Q2W | X | Х | | | Complete PE to be performed at Screening; subsequent focused examinations to be performed as described in Section 8.2.1. |
| Skin<br>assessment | | Х | | | | Х | | | Х | | | Q6W | Х | Х | | | See Section Error! R eference source not found. for skin assessment. |
| Vital signs | | Х | X | Х | X | Х | X | Х | Х | Х | Х | Q2W | Х | X | | | Including weight and height (height at Screening only). See Section 8.2.2. |
| ECOG PS | | Х | Χ | | | | | | | | | | | | | | |
| 12-lead ECG | | X | | | | 1 | 2-lea | d ECG | will be | repeate | ed if clir | ically in | dicated | | | | See Section 8.2.3. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | vention<br>(± 3 da | n Perio<br>ıys) | od | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | of or Within 7 Days of | (± 5 Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | Decision to After Last 4 ter Last (± 2 | | | | | | | | | | | | | |
| | | | | Laboratory Assessments | | | | | | | | | | | | | |
| Virology<br>serology<br>(HIV) | | | | As | s clinio | cally i | ndica | ted in p | articipa | ints with | n a histo | ory of HI | V infection | | | | HIV testing is not mandatory. Any HIV history should be indicated in medical history. If a test is performed at any point in Screening or while on study, a site must consent the participant for HIV testing as per local standard guidance (see Inclusion Criteria 9). |
| Virology<br>serology (HBV<br>and HCV) | | Х | | As | clinio | cally i | ndicat | ted in p | articipa | ınts witl | n a histo | ory of HE | BV or HCV infe | ction | | | |



| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioı<br>(± 3 da | | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat<br>ment | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | of or Within<br>7 Days of | (± 5 Days)<br>After Last | (± 2<br>Weeks) | 12<br>Weeks | |
| | | Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | FD | Decision to<br>Discontinue | Treatment | After Last<br>Treatment | (± 2<br>Weeks) | |
| Hematology | | X | X | X | X | X | X | | X | | X | Q4W | X | X | | | See Appendix 6 for details on blood tests. Samples must also be drawn prior to study intervention administration and results of selected laboratory tests (see Appendix 6) must be reviewed within 3 days prior to dosing. |
| Biochemistry | | X | X | X | X | X | X | | X | | X | Q4W | Х | X | | | Biochemistry is listed in Appendix 6. Samples must be drawn prior to study intervention administration and results of selected laboratory tests (see Appendix 6) must be reviewed within 3 days prior to dosing. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventio<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>_to | | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day of or Within | 28 Days | 12 Weeks<br>(± 2 | Every<br>12 | |
| | | Treat<br>ment | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | 7 Days of | (± 5 Days)<br>After Last | Weeks) | Weeks | |
| | | Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | . 5 | Decision to Discontinue | Treatment | ATTORISET | ` | |
| Urinalysis | | × | | | | | | | As clir | nically i | ndicate | d | | | | | Routine urinalysis at the Screening Visit. If the urinalysis is abnormal, then a culture should be performed. |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioi<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 00 D | 12 Weeks | Every | |
| | | to<br>Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within<br>7 Days of | (I o Days) | (± 2<br>Weeks) | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| β-hCG pregnancy test | | X | × | | × | | × | | X | | X | Q4W | | X | Xi | | β-hCG should be determined from serum at Screening and from a urine or serum sample thereafter. Results of the most recent pregnancy test should be available prior to dosing of study intervention. If a confirmation of a participant's postmenopausal status is necessary, FSH and estradiol tests will be performed at Screening. i: Participants may go to local laboratory to perform pregnancy test. Clinical visit is not required. |
| T4 and TSH | | Х | | | | Х | | | Х | | | Q6W | | Х | | | |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | ventioi<br>(± 3 da | n Perio<br>lys) | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat<br>ment | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until<br>PD | of or Within<br>7 Days of | (± 5 Days)<br>After Last | (± 2<br>Weeks) | 12<br>Weeks | |
| | | Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to Discontinue | Treatment | After Last<br>Treatment | (± 2<br>Weeks) | |
| | | | | | | | | | <b>+</b> T | umor | Assess | ments | | | | | |
| Tumor<br>evaluation<br>/staging (CT<br>scan/MRI/other<br>established<br>methods) | | X | | | | | × | | | | X | Q8W<br>up to<br>12<br>months,<br>then<br>Q12W | | | χi | | See Section 8.1. j: For participants discontinuing treatment due to reason other than PD, perform tumor evaluation Q8W until 12 months (e.g.W49), then Q12W until confirmed PD or study discontinuation. The window for tumor evaluation is ± 7 days. The Intervention Period window of (± 3 days) is not applicable for tumor evaluations. |
| Subsequent<br>anticancer<br>therapy (any<br>line) | | | | | | | | | | | | | | X | X | X | |
| Survival<br>follow-up | | | | | | | | | | | | | | | | Х | |

| | Pre<br>scree<br>ning | Scree<br>ning | | | | | | vention<br>(± 3 da | | d | | | End-of-<br>Treatment<br>Visit | | fety<br>up Visit | Long-<br>term<br>Follow-<br>up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments & Procedures | | Day -28<br>to | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | | On the Day | 28 Days | 12 Weeks | Every | |
| | | Treat | W1 | W3 | W5 | W7 | W9 | W11 | W13 | W15 | W17 | Until | of or Within 7 Days of | (± 5 Days) | | 12<br>Weeks | |
| | | ment<br>Assign<br>ment | D1 | D15 | D29 | D43 | D57 | D71 | D85 | D99 | D113 | PD | Decision to<br>Discontinue | After Last<br>Treatment | After Last<br>Treatment | (± 2 | |
| | | • | | • | • | | • | | PK, | , ADA a | and Bio | marker | | | | | |
| PK and ADA sampling | | | | | | | | See | Table 2 | 2 for Pk | ( and A | DA samp | oling times | | | | |
| Whole blood<br>for pharmaco-<br>genetics | | | X | | | | | | | | | | | | | | Whole blood sample for participants who provide separate informed consent. This sample can be collected at any other visit if missed in this visit. |
| Liquid biopsy<br>(plasma) | | | X | X | | | | | | X | | Q12W | X | | | | Liquid biopsy (plasma) for genetic profiling including TMB analysis will be collected within 2 hours prior to study intervention infusion as scheduled. |

ADA=antidrug antibody, AE=adverse events, β-hCG=β-human chorionic gonadotropin, CT=computed tomography, D=Day, ECG=electrocardiogram, ECOG PS=Eastern Cooperative Oncology Group performance status, FSH=follicle-stimulating hormone, HBV=hepatitis B virus, HCV=hepatitis C virus, HIV=Human immunodeficiency virus, HMGA2=High Mobility Group AT-Hook 2, ICF= informed consent form, MRI=magnetic resonance imaging, PD=progressive disease, PE=physical examination, PK=pharmacokinetics, Q2W=every 2 weeks; Q4W=every 4 weeks, Q6W=every 6 weeks, Q8W=every 8 weeks, Q12W=every 12 weeks, T4=free thyroxine, TMB= Tumor mutational burden, TSH=thyroid-stimulating hormone, V=visit, W=Week.



Table 2 Bintrafusp alfa Pharmacokinetic, Immunogenicity Sampling

| | Screening /<br>Baseline<br>Assessments | | | | ntion Perio<br>3 days) | od | | End-of-<br>Treatment<br>Visit | Safety Fol | low-up Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | V1 | V2 | V3 | V4 | V7 | | | | | |
| | | W1 | W3 | W5 | W7 | W13 | Until | On the Day of or Within | | 12 Weeks | |
| Bintrafusp<br>alfa<br>Measure | Day -28 to<br>First<br>Treatment | | | | D43<br>Pre/End<br>Infusion | | Progression<br>Pre/End | 7 Days of Decision to Discontinue | After Last | (± 2 weeks)<br>After Last | Notes |
| Blood<br>sample for<br>PK | | X/X | X/- | X/X | X/- | X/- | X/-<br>Q6W up<br>to/including<br>W25, then<br>Q12W | X | X | | Samples for PK analysis to be taken before (pre) infusion (as close to the start of the infusion as possible), immediately after the completion of infusion (as close to the completion as possible but no later than 30 minutes post end of infusion). The predose sample should still be drawn even if dosing is ultimately deferred at the study visit. The exact time of each draw must be recorded. |
| Blood<br>sample for<br>ADA | | X/- | X/- | X/- | X/- | X/- | X/-<br>Q6W up<br>to/including<br>W25, then<br>Q12W | Х | Х | | Predose ADA samples to be collected prior to study intervention infusions. The exact time of each draw must be recorded. |

ADA=antidrug antibody, D=day, PK=pharmacokinetics, Q6W=every 6 weeks, Q12W=every 12 weeks, V=visit, W=Week.



### 2 Introduction

Bintrafusp alfa (M7824) is a first-in-class, bifunctional fusion protein that combines an anti-programmed death-ligand 1 (anti-PD-L1) antibody and the soluble extracellular domain of the human transforming growth factor- $\beta$  (TGF- $\beta$ ) receptor as a TGF- $\beta$  neutralizing "trap" into a single molecule. Bintrafusp alfa is the recommended international nonproprietary name for M7824.

Bintrafusp alfa is intravenously administered at 1200 mg every 2 weeks.

Complete information on the chemistry, pharmacology, efficacy, and safety of bintrafusp alfa is detailed in the Investigator's Brochure (IB).





#### 2.2 **Background**

Bintrafusp alfa is a first-in-class, intravenously administered bifunctional fusion protein that combines an anti-PD-L1 antibody and the soluble extracellular domain of the human TGF-B receptor as a TGF-β neutralizing "trap". Bintrafusp alfa is designed to simultaneously target 2 pathways that have independent and complementary immunosuppressive functions in the tumor microenvironment. PD-L1 signaling plays a key role in the immunosuppressive network that dampens T-cell activity and TGF-β functions as an autocrine or paracrine signal within the local tumor microenvironment, where it promotes tumor progression. Bintrafusp alfa has been investigated in the Phase I Study, EMR200647-001, for treatment of several cancers, including TNBC (Spira 2019).

In breast cancer, several studies showed that TGF-β overexpression is related to a worse outcome (Gorsch 1992, Desruisseau 2006). TGF-β within the breast tumor microenvironment is also known to facilitate cancer metastasis (Padua 2008). The loss of TGF-βRII expression has been linked to tumor progression and metastasis, principally in HER2-negative patients (Gobbi 2000).

Approximately 20% of TNBC tumors express PD-L1, although expression is predominantly localized to the tumor-infiltrating lymphocytes (Mittendorf 2014). Importantly, in the TNBC cohort of the Phase I Study of the anti-PD-L1 drug, atezolizumab, higher PD-L1 expression correlated with improved response to treatment and survival (Emens 2019). Similarly, in the recent IMpassion130 study of nab-paclitaxel ± atezolizumab in advanced, treatment-naïve TNBC, 40.9% of participants were determined to be PD-L1 positive and median overall survival (OS) was significantly improved in participants who received chemotherapy plus atezolizumab versus chemotherapy and placebo (25.0 months versus 18.0 months), highlighting the significant contribution of PD-L1 blockade for these participants (Schmid 2018, Schmid 2019).

Bintrafusp alfa has shown promising clinical activity in participants with TNBC in the expansion cohort of the Phase I Study EMR200647-001 (Spira 2019). As of 15 October 2019, participants (n= 33) with heavily pretreated TNBC (54.5% of participants had ≥ 4 prior regimens) received a median of 3 (range 1 to 24) doses of bintrafusp alfa (1200 mg every 2 weeks). Responses as assessed by Investigator occurred in 4 participants; 3 of 4 responses were confirmed by Independent Review Committee (IRC), while the fourth was considered stable disease (SD). The objective response rate (ORR) for these 4 responses was 12.1% (95% confidence interval [CI]: 3.4, 28.2) and disease control was achieved in a total of 5 participants (15.2% [95% CI: 5.1, 31.9]) per Investigator. The median OS was 7.8 months (95% CI: 2.1, 12.8). PD-L1 expression in tumor cells or in the tumor microenvironment was not associated with response to treatment. Bintrafusp alfa was well tolerated, with a safety profile consistent with expectations in this heavily pretreated, advanced TNBC cohort.

In an exploratory analysis of RNAseq data from tumor samples in the TNBC participants, high expression of HMGA2 was associated with response to bintrafusp alfa (Figure 2). A total of 5 TNBC participants in the cohort experienced disease control and had high HMGA2 expression; of these participants, 4 had a partial response (PR) and 1 had SD. One of these participants with a PR had high levels of HMGA2 expression, but low quality RNAseq data, precluding the result from being included in the formal biomarker assessment. However, even excluding that 1 participant, there was a 32.0-fold higher mean expression of HMGA2 in the participants who experienced disease control compared with those who had progressive disease (PD). Using an HMGA2 cutoff defining high expression as the lowest HMGA2 expression in a participant experiencing PR, there were 3 additional participants in the cohort of 33 participants considered to have high HMGA2 (total 8/33, 24%). Of these 3 additional participants, 2 had PD and 1 was non-evaluable as a best response. In summary, 8 participants had high levels of HMGA2 expression, 5 of which experienced disease control, including 4 PRs (ORR in HMGA2 50%, disease control rate 62.5%). As per The Cancer Genome Atlas, approximately 12% of patients with TNBC are projected to have high HMGA2 expression using a comparable cutoff.

HMGA2 is downstream of the TGF- $\beta$  signaling pathway and is known to be a key regulator of epithelial mesenchymal transformation (Thuault 2006). Classically, HMGA2 is associated with poor prognosis, including in breast cancer (Wu 2016). The clinical activity observed in the TNBC cohort in Study EMR200647-001 suggests that participants expressing high levels of HMGA2 might particularly benefit from treatment with a bifunctional molecule which targets TGF- $\beta$  and PD-L1, such as bintrafusp alfa (Locke 2019a).

Based on the biological rationale and promising clinical activity of bintrafusp alfa in TNBC and manageable safety profile in participants with various cancer types (refer to the bintrafusp alfa IB), this study is designed to further investigate bintrafusp alfa in participants with TNBC expressing high levels of HMGA2.

## 2.3 Benefit/Risk Assessment

At the time of study initiation the identified and potential risks with bintrafusp alfa monotherapy were manageable and no new safety signals emerged in the Phase I studies (EMR200647-001, MS200647-0008) compared with therapies targeting PD-L1 or TGF- $\beta$ . The following have been identified as important identified risks for bintrafusp alfa: immune-related adverse events (irAEs; immune-related pneumonitis, immune-related hepatitis, immune-related colitis, immune-related nephritis and renal dysfunction, immune-related endocrinopathies [thyroid disorders, adrenal insufficiency, Type 1 diabetes mellitus, pituitary disorders], immune-related rash and other irAEs [myositis, myocarditis, encephalitis]), TGF- $\beta$  inhibition mediated skin reactions, anemia, and bleeding adverse events. The overall incidence and severity for irAEs is found to be consistent across bintrafusp alfa studies and similar to the known safety profile of approved anti-PD-L1 agents (Brahmer 2018). Infusion-related reactions (IRRs) are classified as identified risk for the treatment with bintrafusp alfa. Infusion-related reactions observed with bintrafusp alfa were similar to those seen with monoclonal antibodies. At the time of study initiation, the overall bintrafusp alfa related IRRs were observed to be < 5%; they were typically low-grade (Grade 1/2) severity and did not require permanent treatment discontinuation.

Dermatologic AEs related to TGF- $\beta$  inhibition (including keratoacanthomas [KA] and cutaneous squamous cell cancers) are an important identified risk with bintrafusp alfa not seen with other programmed death-1 (PD-1)/PD-L1 antibodies. These lesions were previously observed in participants with genetic mutations in the TGF- $\beta$  receptor (i.e., Ferguson-Smith syndrome), and participants treated with the TGF- $\beta$  targeting agent fresolimumab (Goudie 2011, Morris 2014). At the time of study initiation in the Phase I studies, these treatment-emergent TGF- $\beta$  inhibition mediated skin reactions were observed in approximately 11% of participants, were well managed with simple excision (or spontaneous resolution) and did not require any participant to discontinue treatment (refer to IB). The risk of these lesions with bintrafusp alfa was considered manageable, especially in the context of encouraging clinical activity in several tumor types.

No additional/new safety signals emerged in the TNBC cohort of Study EMR200647-001 compared with other tumor types (Spira 2019).

In consideration of the following items, the benefit/risk assessment is considered favorable to conduct this study of bintrafusp alfa in participants with high expressing HMGA2 TNBC:

- The high unmet medical need and absence of an efficacious standard of care for patients with TNBC who have progressed after their first line of chemotherapy.
- The bifunctional mode of action of bintrafusp alfa, targeting 2 complementary and nonredundant signaling pathways within the tumor immune microenvironment.
- The consideration that bintrafusp alfa targets TGF-β (demonstrated in preclinical studies as well as pharmacodynamically in Phase I dose-escalation participants), and that HMGA2 is downstream of the TGF-β signaling pathway (see Section 2.1 and Section 2.2).
- The signal for considerable clinical activity of bintrafusp alfa in participants in Study EMR200647-001 with TNBC expressing high levels of HMGA2 (50% ORR, 62.5% disease control rate) (Locke 2019b).
- The manageable safety profile of bintrafusp alfa observed in the Phase I studies, including TNBC participants.

More detailed information about the known and expected benefits and risks and reasonably expected AEs of bintrafusp alfa may be found in Section 4.2 and the current IB.

Based on the available nonclinical and clinical data to date, the conduct of the study, as specified in this protocol, is considered justifiable.

#### 3 **Objectives and Endpoints**

#### Table 3 **Study Objectives and Endpoints**

| Objectives | Endpoints (Outcome Measures) |
|---|---|
| Primary | |
| To evaluate clinical efficacy of bintrafusp alfa in<br>participants with TNBC with high HMGA2<br>expression, based on ORR | Confirmed objective response according to RECIST 1.1 assessed by an IRC |
| Secondary | |
| To evaluate clinical efficacy of bintrafusp alfa<br>based on DOR | DOR according to RECIST 1.1 assessed by an IRC |
| To evaluate clinical efficacy of bintrafusp alfa<br>based on DRR | Durable response of at least 6 months assessed by an IRC |
| To evaluate clinical efficacy based on PFS | PFS according to RECIST 1.1 assessed by an IRC |
| To evaluate ORR, DOR, DRR, and PFS by<br>Investigator read | Objective response, DOR, DRR, and PFS according to<br>RECIST 1.1 as assessed by the Investigator |
| To evaluate clinical efficacy based on OS | • OS |
| To evaluate clinical safety of bintrafusp alfa | Occurrence of TEAEs and treatment-related AEs including AEs of special interest |

| Objectives | Endpoints (Outcome Measures) |
|---|---|
| To characterize the PK profile of bintrafusp alfa | The concentration observed immediately at the end of infusion (C <sub>EOI</sub> ) of bintrafusp alfa |
| | <ul> <li>The concentration observed immediately before next<br/>dosing (corresponding to predose or trough<br/>concentration [Ctrough] for multiple dosing) of bintrafusp<br/>alfa</li> </ul> |
| To characterize the immunogenicity of bintrafusp alfa | <ul> <li>Immunogenicity of bintrafusp alfa as measured by ADA<br/>assay from Screening through Safety Follow-up Visit up<br/>to 28 days after last treatment</li> </ul> |
| CCI | |

ADA=antidrug antibody, AE=adverse event, DOR=duration of response, DRR=durable response rate, HMGA2=High Mobility Group AT-Hook 2, ir=immune-related, IRC=Independent Review Committee, ORR=Objective response rate, OS=overall survival, PD-L1=programmed death-ligand 1, PFS=progression-free survival, PK=pharmacokinetic, RECIST 1.1=Response Evaluation Criteria in Solid Tumors Version 1.1, TEAE=Treatment-emergent adverse event, TMB=tumor mutational burden, TNBC=triple negative breast cancer.

## 4 Study Design

## 4.1 Overall Design

This is a Phase II, multicenter, single-arm, open label study to evaluate bintrafusp alfa monotherapy in participants with TNBC who express high levels of HMGA2 as determined by a centralized reverse transcriptase-polymerase chain reaction (RT-PCR) test with predefined cutoff. Participants must have progressed during or after first-line of chemotherapy.

The primary objective is to evaluate the clinical efficacy of bintrafusp alfa based on the ORR as assessed by an IRC. The key secondary objectives are duration of response (DOR), durable response rate (DRR), progression-free survival (PFS), OS, and safety. Tumor response evaluations based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) (Eisenhauer 2009) will be performed every 8 weeks until 12 months after the first administration of bintrafusp alfa and then every 12 weeks until confirmed disease progression, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study.

The study plans to enroll approximately 29 eligible participants globally with competitive enrollment.

The study includes:

- Prescreening (a Prescreening informed consent form [ICF] will be used for HMGA2 biomarker analysis and collection of baseline clinical history). Positive HMGA2 test results on tumor tissue is required to enter formal study Screening (see Table 1).
- Up to 28-day Screening period.
- Treatment with bintrafusp alfa at a dose of 1200 mg intravenously once every 2 weeks until confirmed PD, unacceptable toxicity, study withdrawal, or death.
- In the case of PD, treatment may continue past the initial determination of PD or confirmed PD, if the participant's performance status (PS) has remained at least stable, and if in the opinion of the Investigator, the participant will benefit from continued treatment and if other criteria are fulfilled as outlined in the protocol (see Section 7.1.3).
- In the case of SD, PR, or complete response (CR), treatment should be continued until the end of 24 months. If the Investigator believes that a participant will benefit from treatment beyond 24 months, it may be permissible after discussion with the Medical Monitor and the Sponsor Medical Responsible.
- Safety Follow-up will continue until 12 weeks after the last dose of bintrafusp alfa. The 12-week Safety Follow-up is allowed to be conducted via telephone calls or patient chart reviews, unless there is medical necessity requiring a clinical visit.
- Long-term Follow-up for progression and survival should be performed every 12 weeks after the Safety Follow-up according to the Schedule of Activities (Table 1). Long-term Follow-up should be performed by patient chart reviews or telephone calls unless a clinical visit is indicated.

The overall study design is shown in Figure 1. A detailed Schedule of Activities is provided in Section 1.3.

# 4.2 Scientific Rationale for Study Design

This study investigates participants with TNBC and high HMGA2 expression who have progressed during or after first-line of chemotherapy (see Section 2). The inclusion criteria for TNBC is based upon American Society of Clinical Oncology (ASCO)/College of American Pathologists guidelines (Hammond 2010a, Hammond 2010b, Wolff 2013). The decision to enroll participants with high HMGA2 expression is based on encouraging signals from a Phase I Study with bintrafusp alfa in TNBC participants (see Section 2.2). HMGA2 expression will be determined by a centralized RT-PCR assay with predefined cutoff and appropriate regulatory status.

A single-arm design is considered justified given the overall low activity of immunotherapy monotherapy in chemotherapy-experienced TNBC participants (see Section 9.2), and the aim of this study is to further explore the efficacy signal observed in the biomarker-positive population.

Standard endpoints will be used to assess efficacy. The primary objective is the confirmed ORR as assessed by an IRC according to RECIST 1.1, and the key secondary endpoints include DOR, DRR, PFS, OS, and safety.

The sample size of 29 participants is based on the preliminary signals of substantial efficacy (see Section 9.2) and includes an opportunity to assess this efficacy after the first 15 participants (see Section 9.2 and Section 9.4.4) as well as an opportunity to assess if the preselection biomarker tends to show predictive properties related to clinical activity as anticipated. In a future amendment, further cohorts may be added if the biomarker is validated as identifying participants who will clinically benefit from bintrafusp alfa to further explore additional participants who may benefit and/or may be extended to support registration intent.

#### 4.3 **Justification for Dose**

The recommended Phase II dose (RP2D) for bintrafusp alfa is 1200 mg administered as an intravenous infusion once every 2 weeks. The selection of RP2D is based on the available clinical data from the Phase I studies EMR200647-001 and MS200647-0008, including safety/tolerability, pharmacokinetics (PK), and pharmacodynamics (PD-L1 target occupancy in peripheral blood mononuclear cell and TGF-β plasma concentrations), as well as efficacy in second-line non-small cell lung cancer cohorts from the Study EMR200647-001. The selection of RP2D is also supported by population pharmacokinetic (PopPK) and exposure-response modeling and simulation.

Refer to the IB for the complete and detailed data and analysis for dose justification.

#### 4.4 **End of Study Definition**

A participant has completed the study if he/she has completed all study parts, including the last visit or the last scheduled procedure shown in Section 1.3.

The end of the study is defined as the date of completion of 24 months of follow-up after the accrual of the last participant. After the stipulated end of study, Survival Follow-up may continue until the last participant has died or at the discretion of the Sponsor.

The Sponsor may terminate the study at any time once access to study intervention for participants still benefiting is provided via a rollover study, expanded access, marketed product, or another mechanism of access as appropriate.

#### 5 **Study Population**

The criteria in Section 5.1 and Section 5.2 are designed to enroll only participants, who are appropriate for the study; thereby, ensuring the study fulfills its objectives. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a participant is suitable for this study.

Prospective approval of protocol deviations to inclusion and exclusion criteria, also known as protocol waivers or exemptions, is not permitted.

Before performing any study assessments that are not part of the participant's routine medical care, the Investigator will confirm that the participant or the participant's legal representative (where allowed by local laws and regulations) has provided written informed consent, as indicated in Appendix 2.

## 5.1 Inclusion Criteria

Participants are eligible to be included in the study only if all the following criteria apply:

### Age

1. Are  $\geq$  18 years of age at the time of signing the informed consent (Main ICF).

### **Type of Participant and Disease Characteristics**

- 2. Are participants with histologically or cytologically confirmed TNBC. Absence of HER2, estrogen receptor, and progesterone receptor expression must be documented:
- HER2 negativity is defined as either of the following by local laboratory assessment:
  - o In situ hybridization non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), or
  - o Immunohistochemistry (IHC) 0 or IHC 1+ (if more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the Medical Monitor to establish eligibility of the participant).
- Estrogen receptor and progesterone receptor negativity are defined as < 1% of cells expressing hormonal receptors via IHC analysis.
- Participants must have received at least one line of systemic therapy for metastatic disease and have progressed on the line of therapy immediately prior to study entry. There is no limit to the number of prior therapies.
- Participants may prescreen for HMGA2 expression while on preceding treatment, however screening should only occur if in the opinion of the Investigator, the participant would likely be eligible for study within 6 months. For enrollment, participant must have progressed during or after prior line of systemic treatment, and a 28-day washout period is required. Enrollment for the study is competitive, therefore a result of HMGA2 high tumor expression as determined by central testing prior to participant being eligible does not guarantee a slot until formally entering the screening procedures, indicated by signing the Main ICF.
- 3. Measurable disease according to RECIST 1.1 at Screening in the opinion of the Investigator.
- 4. Availability of either archival tumor tissue or fresh core or excisional biopsy of a tumor lesion (primary or metastatic, excluding bone biopsies) is mandatory to determine HMGA2 expression level prior to enrollment. Fine needle aspirates are not acceptable. Tumor material must be suitable for biomarker assessment as described in the Laboratory Manual. If an archival sample is submitted during Prescreening for HMGA2 testing, a fresh tumor biopsy during the Screening period is additionally encouraged if feasible for exploratory biomarker analysis.
- 5. HMGA2 high tumor expression is required. If a tumor specimen is assessed as not evaluable for HMGA2 expression by the central laboratory, another sample may be submitted to assess for HMGA2 high status. The status of tumor HMGA2 expression (high versus not high) will be determined by a centralized RT-PCR assay with predefined cutoff

(documented in the applicable documentation submitted to the Food and Drug Administration [FDA]) and with appropriate regulatory status.

- 6. Have Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1 at study entry and Day 1 of treatment with bintrafusp alfa.
- 7. Life expectancy > 12 weeks as judged by the Investigator at study start.
- 8. Have adequate organ function:
  - Adequate hematological function defined by absolute neutrophil count  $\geq 1.5 \times 10^9 / L$ , platelet count  $\geq 100 \times 10^9$ /L, and hemoglobin (Hgb)  $\geq 9$  g/dL.
  - Adequate hepatic function defined by a total bilirubin level  $\leq$  the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels  $< 1.5 \times ULN$ . For participants with liver involvement in their tumor, AST  $< 5.0 \times ULN$ . ALT  $\leq 5.0 \times \text{ULN}$ , and bilirubin  $\leq 3.0 \times \text{ULN}$  are acceptable.
  - Adequate renal function defined by creatinine  $\leq 1.5 \times \text{ULN}$  or calculated creatinine clearance (CrCL) ≥ 30 mL/min for participant with creatinine > 1.5 × ULN (glomerular filtration rate can also be used).

Note: CrCL should be calculated per institutional standard. If no local guideline is available, CrCL should be calculated using the Cockcroft-Gault Method:

- $CrCL = ([140\text{-age}] \times \text{weight [kg}] \times [0.85 \text{ for females only}])/(72 \times \text{creatinine}).$
- Adequate coagulation function defined as international normalized ratio or prothrombin time < 1.5× ULN unless the participant is receiving anticoagulant therapy and activated partial thromboplastin time  $\leq 1.5 \times \text{ULN}$  unless the participant is receiving anticoagulant therapy.
- 9. Participants with known human immunodeficiency virus (HIV) infections are in general eligible if the following criteria are met (FDA Guidance on Cancer Clinical Trial Eligibility, March 2019):
  - If clinically indicated participants must be stable on antiretroviral therapy (ART) for at least 4 weeks and agree to adhere to ART. If not clinically indicated, consult study Medical Monitor.
  - Participants with HIV infection should have no evidence of documented multidrug resistance that would prevent effective ART.
  - Have an HIV viral load of < 400 copies/mL at Screening. c.
  - Have CD4+ T-cell (CD4+) counts  $\geq 350 \text{ cells/}\mu\text{L}$ .
  - For patients with a history of an AIDS-defining opportunistic infection within the last 12 months, patients may be eligible only after consultation and agreement with the study Medical Monitor.
  - If prophylactic antimicrobial drugs are indicated, patient may still be considered eligible f. upon agreement with the study Medical Monitor.

- 10. Participants with hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infections are in general eligible if the following criteria are met (FDA Guidance on Cancer Clinical Trial Eligibility, March 2019):
  - Patients with serologic evidence of chronic HBV infection must have an HBV viral load below the limit of quantification and be on a stable dose of antiviral therapy.
  - Patients with a history of HCV infection should have completed curative antiviral b. treatment and require HCV viral load below the limit of quantification.
  - Patients on concurrent HCV treatment should have HCV below the limit of c. quantification.

#### Sex

#### 11. Are female or male:

- a. A female is eligible if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
- Not a woman of childbearing potential (WOCBP).

OR

- If a WOCBP, use a highly effective contraceptive method (i.e., with a failure rate of < 1% per year), preferably with low user dependency, as described in Appendix 3 for the following time periods:
  - o Before the first dose of the study intervention(s), if using hormonal contraception:
    - Has completed at least one 4-week cycle of an oral contraception pill and either had or has begun her menses.

OR

- Has used a depot contraceptive or extended-cycle oral contraceptive for at least 28 days and has a documented negative pregnancy test using a highly sensitive assay.
- o During the intervention period.
- o After the study intervention period (i.e., after the last dose of study intervention is administered) for at least 2 months.

The Investigator evaluates the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

Have a negative serum or highly sensitive urine pregnancy test, as required by local regulations, within 24 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required.

Additional requirements for pregnancy testing during and after study intervention are in Section 8.2.4.
The Investigator reviews the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female with an early undetected pregnancy.

b. Males with TNBC may also screen for this study.

Male participants are eligible to participate if they agree to the following during the intervention period and for at least 4 months after the last dose of study intervention:

• Refrain from donating sperm

PLUS, either

• Abstain from intercourse with a female

OR

- Use a male condom:
  - When having sexual intercourse with a WOCBP, who is not currently pregnant, and advise her to use a highly effective contraceptive method with a failure rate of < 1% per year, as described in Appendix 3, since a condom may break or leak.
  - o When engaging in any activity that allows for exposure to ejaculate.

#### **Informed Consent**

12. Capable of giving signed informed consent, as indicated in Appendix 2, which includes compliance with the requirements and restrictions listed in the Main ICF and this protocol.

### 5.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions**

- 1. Participants with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention are excluded. Participants with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 4 weeks, and are not using steroids for at least 7 days prior to the start of study intervention. Brain lesions, if present, should not be selected as target lesions, but should be assessed as non-target lesions.
- 2. Has interstitial lung disease OR has had a history of pneumonitis that has required oral or intravenous steroids.
- 3. Receipt of any organ transplantation, including stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
- 4. Previous malignant disease (other than the target malignancy to be investigated in this study) within the last 3 years, except:

- a. Participants with a history of superficial/noninvasive bladder cancer, or basal or squamous cell carcinoma in situ previously treated with curative intent are NOT excluded.
- b. Endoscopically resected early gastrointestinal cancers limited to mucosal layer (esophageal, gastric, and colorectal) that are without recurrence in > 1 year are allowed.
- c. Participants with other localized malignancies treated with curative intent should be discussed with the Medical Monitor. Further biopsy/evaluations may be required prior to allowing enrollment if there are any concerns of a non-TNBC cancer recurrence.

Any questions regarding these criteria should be discussed with Medical Monitor.

- 5. Significant acute or chronic infections including but not limited to:
  - a. Participants with active tuberculosis (history of exposure or history of positive tuberculosis test; plus presence of clinical symptoms, physical, or radiographic findings).
  - b. Active bacterial or fungal infection requiring systemic therapy (except as indicated, discuss alternative scenarios with the Medical Monitor).
- 6. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, except:
  - a. Participants with diabetes Type 1, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
  - b. Participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg of prednisone or equivalent per day.
  - c. Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intraocular, or inhalation) is acceptable.
- 7. Known severe hypersensitivity (Grade ≥ 3 National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v5.0]) to investigational product (bintrafusp alfa) or any components in its formulation, any history of anaphylaxis, or recent, within 5 months, history of uncontrollable asthma.
- 8. Persisting Grade > 1 NCI-CTCAE v5.0 toxicity (except alopecia and vitiligo) related to prior therapy; however, sensory neuropathy Grade ≤ 2 is acceptable.
- 9. Clinically significant cardiovascular/cerebrovascular disease including: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia. Participants with history of bleeding diathesis or recent major bleeding events considered by the Investigator as high risk for investigational drug treatment are also excluded.
- 10. Severe and/or clinically relevant acute or chronic diseases which, in the opinion of the Investigator, might impair the participant's tolerance for the study or ability to consistently participate in study procedures.

### **Prior/Concomitant Therapy**

- 11. Has received prior cancer treatment with any other immunotherapy or checkpoint inhibitors, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-cell lymphocyte-associated antigen-4, or any other immune-modulating monoclonal antibody (e.g., any other antibody or drug specifically targeting T-cell co-stimulation, checkpoint pathways, or immune-suppressive pathways [e.g., TGF-β]).
- 12. Concurrent treatment with prohibited drugs (see Section 6.5.2).
- 13. Systemic therapy with immunosuppressive agents within 7 days before the start of study intervention; or use of any investigational drug within 28 days before the start of study intervention.
- 14. Has received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted.

#### **Prior/Concurrent Clinical Study Experience**

15. Participants, who received chemotherapy, radiation therapy (with the exception of palliative radiotherapy delivered in a normal organ-sparing technique), or biological therapy (e.g., antibodies) within 4 weeks, or who have been treated with small molecule therapeutics or investigational agents within 4 weeks prior to starting bintrafusp alfa or who have not recovered from the side effects of such therapy (except for alopecia or potentially neuropathy).

#### **Other Exclusions**

- 16. Major surgery within 28 days before the start of study intervention (diagnostic biopsy, for example, is not considered major surgery).
- 17. Pregnancy or breast feeding.
- 18. Known active alcohol or drug abuse.

## 5.3 Lifestyle Considerations

No specific lifestyle or dietary restrictions are required throughout the study.

#### 5.4 Screen Failures

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened. Rescreened participants will be assigned a new participant number.

For participants who have abnormal laboratory values at Screening that may correct or are using a prohibited concomitant medication that will be discontinued, or undergoing a prohibited procedure that will be completed, Screening period may be extended up to 2 weeks. In other situations when a participant has been screen-failed, the site should contact the Medical Monitor to discuss whether the participant may be rescreened.

## 6 Study Intervention(s)

Study intervention is any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant per the study protocol.

## 6.1 Study Intervention(s) Administration

**Table 4 Study Intervention** 

| Study Intervention Name: | Bintrafusp alfa (M7824) |
|---|---|
| <b>Dose Formulation:</b> | Sterile concentrate solution for infusion |
| Unit Dose Strength(s)/Dosage Level(s): | 10 mg/mL in single-use glass vials |
| Route of Administration: | Intravenous infusion |
| <b>Dosing Instructions:</b> | Flat dose of 1200 mg over 1 hour (-10 minutes/+ 20 minutes, i.e., over 50 to 80 minutes) once every 2 weeks |
| Sourcing | Provided centrally by the Sponsor |
| Packaging and Labeling: | Each vial will be packaged and labeled per all applicable regulatory requirements and Good Manufacturing Practice Guidelines. |

# 6.2 Study Intervention(s) Preparation, Handling, Storage, and Accountability

The Investigator, institution, or the head of the medical institution (where applicable), is responsible for study intervention accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).

- Upon receipt of the study intervention(s), the Investigator or designee must confirm appropriate temperature conditions have been maintained during transit and any discrepancies are reported and resolved before use. Also, the responsible person will check for accurate delivery. Further guidance and information for study intervention accountability are provided in the Pharmacy Manual.
- Only participants enrolled in the study may receive study intervention(s) and only authorized site staff may supply it. All study intervention(s) must be stored in a secure, environmentally-controlled, and monitored (manual or automated) area, in accordance with the labeled storage conditions, and with access limited to the Investigator and authorized site staff.
- Dispensing will be recorded on the appropriate accountability forms so that accurate records will be available for verification at each monitoring visit.
- Study intervention(s) accountability records at the study site will include the following:
  - Confirmation of receipt, in good condition and in the defined temperature range.

- The inventory provided for the clinical study and prepared at the site.
- The dose(s) each participant used during the study.
- The disposition (including return, if applicable) of any unused study intervention(s).
- Dates, quantities, batch numbers, vials numbers, expiry dates, formulations, and the participant numbers.
- The Investigator site will maintain records, which adequately documents that participants were provided the doses specified in this protocol, and all study intervention(s) provided were fully reconciled.
- Unused study intervention(s) must not be discarded or used for any purpose other than the present study. No study intervention that is dispensed to a participant may be re-dispensed to a different participant.
- A Study Monitor will periodically collect the study intervention(s) accountability forms.
- Destruction of used and unused study intervention(s) should be performed at the site if allowed by local law only after Sponsor authorization. If that is not possible, the Sponsor/designee will be responsible.
- Further guidance and information for the final disposition of unused study intervention(s) are provided in the Pharmacy Manual.
- Bintrafusp alfa should be stored in a refrigerator (2°C to 8°C) until use. Bintrafusp alfa must not be frozen and should be stored in the original packaging.
- Additional instructions for the preparation, handling, storage, and disposal of bintrafusp alfa will be provided in the Pharmacy Manual.

# 6.3 Measures to Minimize Bias: Study Intervention Assignment and Blinding

## 6.3.1 Study Intervention Assignment

The Sponsor or delegate will assign a unique participant identifier number to participants in chronological order at the time of Prescreening informed consent signature. Participant identifiers will be comprised of digits representing the study number, the site number, and the participant number, which is allocated sequentially. Enrollment will utilize an Interactive Voice/Web Response System.

## 6.3.2 Blinding

Not applicable.

## 6.4 Study Intervention Compliance

In this study, participants will receive study intervention at the study site. Well-trained medical staff will monitor and perform the study intervention administration. The information of each study

intervention administration, including the date, time, and dose of study intervention, will be recorded on the electronic case report form (eCRF). The Investigator will make sure that the information entered into the eCRF regarding study intervention administration is accurate for each participant. Any reason for noncompliance should be documented.

Noncompliance is defined as a participant missing > 1 infusion of study intervention for nonmedical reasons and barring any extenuating circumstances in the opinion of the Investigator. Extenuating circumstances should be documented, and when possible, discussed with the Sponsor in advance. If 1 infusion is missed and the interval between the subsequent infusion and the last administered treatment is longer than 4 weeks for nonmedical reasons, the criterion of insufficient compliance may be met as well. Participants who miss  $\geq 2$  doses must be discussed with Medical Monitor (see Section 6.8).

Consequences of noncompliance may lead to discontinuation of study intervention as described in Section 7.1. In case of overdose, see Section 8.4.

## 6.5 Concomitant Therapy

Record in the eCRF all concomitant therapies (e.g., medicines or nondrug interventions) used from the time the participant signs the Prescreening informed consent until completion of the study, including any changes. For prescription and over-the-counter medicines, vaccines, vitamins, and herbal supplements, record the name, reason for use, dates administered, and dosing information.

Any additional concomitant therapy that becomes necessary during the study and any change to concomitant drugs must be recorded in the corresponding section of the eCRF, noting the name, dose, duration, and indication of each drug.

Contact the Medical Monitor for any questions on concomitant or prior therapy.

#### 6.5.1 Permitted Medicines

The only permitted medications are the following:

- 1. Any medications (other than prohibited in Section 6.5.2) that are considered necessary for the participants' welfare and will not interfere with the study intervention may be given at the Investigator's discretion.
- 2. Other drugs to be used for non-steroid premedication when indicated (e.g., antihistamine and acetaminophen; steroids are not allowed to be used for premedication).
- 3. Other drugs, including steroids, as indicated, may be used for the treatment of anaphylactic reactions, IRRs, and severe hypersensitivity reactions/flu-like symptoms and irAEs (see Section 6.9).
- 4. Blood transfusions and erythroid growth factors are permitted as clinically indicated.

Any medicines that are considered necessary to protect the participant's welfare in emergencies may be given at the Investigator's discretion, regardless if it results in a protocol deviation.

#### 6.5.2 Prohibited Medicines

The following treatments must not be administered during the 28-day Screening period and for the duration of study intervention. If the administration of a nonpermitted concomitant drug becomes necessary during the study, the participant will be withdrawn from study intervention (the Sponsor may be contacted to discuss whether the study intervention must be discontinued).

- Immunotherapy, immunosuppressive drugs (e.g., chemotherapy or systemic corticosteroids), or other experimental pharmaceutical products are prohibited. Exceptions are allowed for short-term treatment of allergic reactions or for the treatment of irAEs, specifically:
  - Short-term administration of systemic steroid (i.e., for allergic reactions or the management of irAEs) is allowed.
  - Steroids with no or minimal systemic effect (topical, intranasal, intraocular, inhalation) are allowed.
  - Hormone replacement with corticosteroids for adrenal insufficiency is allowed if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or equivalent prednisone per day.
- Prophylactic use of corticosteroids for IRRs is prohibited.
- Concomitant local or regional treatment (radio/chemo-embolization) is prohibited.
- Other systemic anticancer therapy.
- Live vaccines are prohibited. Administration of inactivated vaccines is allowed (e.g., inactivated influenza vaccines).
- Any traditional Chinese medication used as anticancer treatment (regardless of the type of cancer) is prohibited. Traditional Chinese medication for indications other than anticancer treatment, such as supportive care, may be administered at the discretion of the Investigator. List of prohibited Chinese medications is provided in the Appendix 7.
- Herbal remedies with immunostimulating properties (e.g., mistletoe extract) or known to potentially interfere with major organ function (e.g., hypericin).

Medications other than those specifically excluded in this study (see above) may be administered for the management of symptoms associated with the administration of bintrafusp alfa as required. These might include analgesics, antinausea medications, antihistamines, diuretics, antianxiety medications, and medication for pain management, including narcotic agents.

#### 6.5.3 Other Interventions

#### **Permitted Procedures**

• Palliative organ-sparing radiotherapy may be administered only for specific clinical indications during the study. The assessment of PD will be made according to RECIST 1.1 and not based on the necessity for palliative radiotherapy.

#### **Prohibited Procedures**

• Major surgery within 4 weeks before the start of the study. Discuss with the Medical Monitor if unplanned major surgery is required on study to plan for timing of re-treatment. Any diagnostic biopsies collected for clinical reasons during the study should be documented as a concomitant procedure including the outcome of available pathology reports.

#### 6.6 Dose Selection and Modification

Participants will receive an intravenous infusion of bintrafusp alfa at a dose of 1200 mg over 1 hour (-10 minutes/+ 20 minutes, i.e., over 50 to 80 minutes) once every 2 weeks as detailed in the Schedule of Activities (Table 1).

Dose modification of bintrafusp alfa is not allowed.

## 6.7 Study Intervention After the End of the Study

After a participant has completed the study, has withdrawn consent, or has been withdrawn early, symptom guided appropriate treatment will be administered, if required, in accordance with the study site's standard of care and generally accepted medical practice and depending on the participant's individual medical needs. Participants will be followed for survival and AEs as specified in the Schedule of Activities (Table 1).

On withdrawal from the study, participants may receive whatever care they and their physicians agree upon.

## **6.8** Special Precautions

Any treatment-emergent adverse event (TEAE) that is assessed as potentially related to bintrafusp alfa, may require permanent or transient discontinuation of bintrafusp alfa treatment.

Single laboratory values out of the normal range that do not have any clinical correlation do not necessarily need treatment interruption. Questions or concerns with regard to management and/or follow-up of TEAEs should be discussed with the Medical Monitor.

Immune-related AEs, IRRs including hypersensitivity, anemia, TGF-β inhibition mediated skin reactions, and bleeding events are managed and followed up in their respective sections as indicated below. Permanent study intervention discontinuation may be recommended, so the relevant section must be reviewed:

- For suspected irAEs, general management by NCI-CTCAE v5.0 toxicity grading is listed in Section 6.9.2. Recommended guidance and management for specific irAEs as per published guidelines is provided in Appendix 5.
- IRR and hypersensitivity reaction guidance are presented in Section 6.9.1.
- Anemia guidance is presented in Section 6.9.4.

- Potential TGF-β inhibition mediated skin AEs guidance and management are provided in Section 
- Guidance and management of bleeding events are discussed in Section 6.9.5.

### General guidance:

- In any case, if  $\geq 2$  doses are missed due to AE, the Medical Monitor should be consulted.
- Inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks is an indication for permanent treatment discontinuation (except for use of steroids as hormone substitution).
- Persistent Grade 2 or 3 adverse reactions (excluding endocrinopathies controlled with hormone replacement therapy) that do not recover to Grade 0 to 1 within 12 weeks after last dose of study intervention is an indication for permanent treatment discontinuation.

In general, the following applies for TEAEs related to bintrafusp alfa that are not covered by the recommendations for irAE management in Appendix 5:

#### **Grade 4 treatment-related TEAEs**

Any Grade 4 treatment-related TEAEs require permanent treatment discontinuation, except:

- Endocrinopathies that have been controlled by hormone replacement,
- Isolated laboratory values out of normal range that do not have any clinical correlation. Discuss with Medical Monitor regarding work-up, management, and treatment continuation versus hold versus discontinuation for isolated Grade 4 laboratory abnormalities
- If alternative explanation is identified for Grade 4 non-tumor bleeding.

See Appendix 5 for guidance on specific Grade 4 irAEs, as most require permanent treatment discontinuation.

#### **Grade 3 treatment-related TEAEs**

- 1. Participants with any severe or Grade 3 treatment-related adverse reactions that recur should be permanently discontinued. Exceptions may be considered for the following after discussion with Medical Monitor:
  - Transient Grade 3 flu-like symptoms or fever that is controlled with medical management
  - Transient Grade 3 fatigue, local reactions, headache, nausea, emesis that resolves to < Grade 1 or baseline
  - Tumor flare phenomenon defined as local pain, irritation, or rash localized at sites of known or suspected tumors
  - Any Grade  $\geq$  3 drug-related amylase or lipase abnormality that is not associated with symptoms or clinical manifestations of pancreatitis

- Grade 3 Hgb decrease (< 8.0 g/dL) that is clinically manageable with blood transfusions or erythroid growth factor use
- Increases in ECOG PS  $\geq$  3 that resolves to  $\leq$  2 by Day 1 of the next infusion (i.e., infusions should not be given if the ECOG PS is  $\geq$  3 on the day of treatment and should be delayed until ECOG PS  $\leq$  2)
- KA and cutaneous squamous cell carcinoma (cSCC)
- Grade 3 non-tumor bleeding requiring intervention or hospitalization if alternative explanation can be identified (such as concomitant use of antithrombotic agents, traumatic event, etc).
- 2. See Appendix 5 for guidance on specific Grade 3 irAEs as many require permanent treatment discontinuation, including pneumonitis and nephritis.
  - AST or ALT > 5 times ULN or total bilirubin > 3 times ULN must be permanently discontinued, except for participants with liver metastases (e.g., who begin treatment with Grade 2 AST or ALT). These participants should be discontinued if AST or ALT increases by ≥ 50% relative to baseline and lasts for at least 1 week.
- 3. Persistent Grade 3 adverse reactions (excluding endocrinopathies controlled with hormone replacement therapy) that do not recover to Grade 0 to 1 within 12 weeks after last dose of treatment.

#### **Grade 2 treatment-related TEAEs**

- 1. If a Grade 2 treatment-related TEAE resolves to Grade  $\leq 1$  by the day before the next infusion, study intervention may be continued.
- 2. If a Grade 2 treatment-related TEAE does not resolve to Grade ≤ 1 by the day before the next infusion, but it is manageable and/or not clinically relevant, the Medical Monitor should be consulted to assess if it is clinically reasonable to administer the following infusion.

Note that treatment recommendations regarding continuation, hold, or discontinuation by grade are different depending on the specific toxicity (see Appendix 5). Toxicity grading is assigned based on NCI-CTCAE v5.0.

## 6.9 Management of Adverse Events of Special Interest

Adverse events of special interest (AESI) are serious or nonserious AEs specific to the known mechanism of action of the study intervention that are of clinical interest.

For this study, AESIs include the following:

- Infusion-related reactions including hypersensitivity
- Immune-related AEs



- TGF-β inhibition mediated skin reactions
- Anemia
- Bleeding AEs

## 6.9.1 Infusion-related Reactions Including Hypersensitivity

Infusion-related reactions, including hypersensitivity, are defined in this section. Infusion-related reactions are AESIs and identified risks for bintrafusp alfa.

#### **Infusion-Related Reactions**

Infusion-related reactions are defined as any signs or symptoms experienced by participants during the infusion of pharmacologic or biologic agents or any event occurring during or within 1 day of study intervention administration. They are identified based on a list of Medical Dictionary for Regulatory Activities (MedDRA) preferred terms and criteria on the timely relationship to an infusion. Events are divided into reactions versus signs and symptoms:

- Reactions are considered when onset is on the day of infusion (during or after the infusion) or the day after the infusion (irrespective of resolution date) for IRR, drug hypersensitivity, anaphylactic reaction, hypersensitivity, and Type 1 hypersensitivity.
- Signs and symptoms of IRR and hypersensitivity/allergic reactions are considered when onset is on the day of infusion (during or after the infusion) and resolved completely with the end date within 2 days after onset of (but not limited to) pyrexia, chills, flushing, hypotension, dyspnea, wheezing, back pain, abdominal pain, and urticaria.

#### **Management of Infusion-Related Reactions**

Premedication prior to bintrafusp alfa administration is optional and at the discretion of the Investigator. If an Investigator chooses to administer premedications, premedication with an antihistamine and with paracetamol (acetaminophen) (e.g., 25 to 50 mg diphenhydramine and 500 to 650 mg paracetamol [acetaminophen] intravenous or oral equivalent) approximately 30 to 60 minutes prior to each dose of bintrafusp alfa is recommended.

If Grade  $\geq 2$  IRRs are seen during the first 2 infusions, premedication should be continued/implemented for future infusions.

An assessment for possible IRR should be triggered based upon the development of specific symptoms within 24 hours of an infusion.

Management of symptoms should follow the guidelines as shown in Table 5.

#### Table 5 Treatment Modification of Bintrafusp alfa for Symptoms of **Infusion-Related Reactions Including Hypersensitivity**

#### NCI-CTCAE v5.0 Grade

## **Treatment Modification**

#### Grade 1 - mild

- Mild transient reaction; infusion interruption not indicated; intervention not indicated.
- · Increase monitoring of vital signs as medically indicated as long as participants are deemed medically stable by the attending Investigator.

#### Grade 2 - moderate

- Therapy or infusion interruption indicated but if responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDs, narcotics, IV fluids); prophylactic medications indicated for  $\leq$  24 hours.
- Stop the infusion of the study intervention caused
- Increase monitoring of vital signs as medically indicated as participants are deemed medically stable by the attending Investigator.
- If symptoms resolve quickly or decrease to Grade 1, resume infusion at 50% of original rate with close monitoring of any worsening, otherwise dosing held until resolution of symptoms with mandated premedication for the next scheduled visit.
- If worsens to Grade 3 or 4, follow treatment modification guidelines accordingly.

#### Grade 3 or Grade 4 - severe or life-threatening

- Grade 3: Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical
- Grade 4: Life-threatening consequences; urgent intervention indicated.
- Stop the infusion of study intervention caused IRR immediately and disconnect infusion tubing from the participant with additional appropriate medical measures and closely monitor until deemed medically stable by the attending Investigator. Hospitalization and/or close monitoring is recommended.
- Administration of glucocorticoids may be required.
- Restart the medication taking out the drug that is the cause of IRRs from the next scheduled visit.

IRR=infusion-related reaction, IV=intravenous, NCI-CTCAE=National Cancer Institute Common Terminology Criteria for Adverse Events, NSAID=nonsteroidal anti-inflammatory drug.

Once the bintrafusp alfa infusion is interrupted or rate reduced to 50% of previous infusion rate, it must remain decreased for all subsequent infusions. For Grade 3 or 4 IRRs, bintrafusp alfa discontinuation is mandated. For all types and grades of infusion reactions, details about drug physical constitution, method of preparation, and infusion must be recorded.

In the event of a Grade 2 IRR that does not improve or worsens after implementation of the treatment modifications indicated in Table 5 (including reducing the infusion rate by 50%), the Investigator may consider treatment with corticosteroids and the infusion should be stopped for that day. At the next infusion, the Investigator may consider the addition of H2 blocker antihistamines (e.g., famotidine or ranitidine), in addition to the above provided recommended optional premedication regimen, for selected participants. However, prophylactic steroids are not permitted. At the next dose, if the participant has a second IRR Grade  $\geq 2$  on the slower infusion rate, with the addition of further medication to premedication, the infusion should be stopped, and the Investigator may consider withdrawal of this participant from the study intervention.

### **Hypersensitivity Reaction**

If a hypersensitivity reaction occurs, the participant must be treated according to the best available medical practice. A complete guideline for the emergency treatment of anaphylactic reactions according to the Working Group of the Resuscitation Council United Kingdom and can be found at https://www.resus.org.uk/pages/reaction.pdf. Participants should be instructed to report any delayed reactions to the Investigator immediately.

Symptoms may include, but are not limited to:

- Impaired airway
- Decreased oxygen saturation (< 92%)
- Confusion
- Lethargy
- Hypotension
- Pale/clammy skin
- Cyanosis

Management of hypersensitivity includes:

- Epinephrine injection and intravenous dexamethasone.
- Participant should be placed on cardiac, blood pressure, heart rate, and oxygen saturation monitoring immediately.
- Alert intensive care unit for possible transfer if required.

#### **Prophylaxis of Flu-Like Symptoms**

For prophylaxis of flu-like symptoms, a nonsteroidal anti-inflammatory drug, e.g., ibuprofen 400 mg or comparable nonsteroidal anti-inflammatory drug dose, may be administered 2 hours before and 8 hours after the start of each intravenous infusion.

### 6.9.2 Immune-related Adverse Events

Immune-related AEs are specific to immunotherapies and vary by organ system. Immune-related AEs are considered AESIs.

In general, the spectrum of irAEs is similar for bintrafusp alfa compared with other checkpoint inhibitors. Effective risk management of these toxicities (irAEs) primarily caused due to inhibition of PD-L1 and PD-1 pathways is based on key recommendations (Champiat 2016). Participant education for on-time reporting of symptoms of potential irAEs and prompt clinical assessment is critical for effective management and quicker resolution of immune-mediated toxicities, thus preventing progression into severe forms of toxicity that otherwise may become life-threatening and difficult to manage or warrant permanent discontinuation from the study.

The following irAEs are important identified risks for bintrafusp alfa

- Immune-related hepatitis
- Immune-related pneumonitis
- Immune-related colitis
- Immune-related nephritis and renal dysfunction
- Immune-related endocrinopathies (thyroid disorders, adrenal insufficiency, Type 1 diabetes mellitus, pituitary disorders)
- Immune-related rash
- Other immune-related events (myositis, myocarditis, encephalitis).

The following irAEs are important potential risks for bintrafusp alfa:

- Guillain-Barré syndrome
- Uveitis
- Pancreatitis
- Myasthenia gravis/myasthenic syndrome.

The Medical Monitor may be involved as needed for follow-up. Details of the diagnostic work-up will be requested by the study team.

Recommended guidance and management for specific irAEs as per published guidelines are provided in Appendix 5. These recommendations are in accordance with the joint ASCO Clinical Practice Guidelines (Brahmer 2018) and National Comprehensive Cancer Network (NCCN 2018) guidelines.

Treatment of irAEs is mainly dependent upon severity as defined by NCI-CTCAE v5.0. In general, management by NCI-CTCAE v5.0 grading is listed below:

- Grade 1: study intervention should be continued with close monitoring, with the exception of some neurologic, hematologic, and cardiac toxicities.
- Grade 2: study intervention may be suspended for most Grade 2 toxicities, with consideration of resuming when symptoms revert to Grade 1 or less. Corticosteroids may be administered (initial dose of 0.5 to 1 mg/kg/day of prednisone or equivalent).
- Grade 3: study intervention is generally suspended and the high-dose corticosteroids (prednisone 1 to 2 mg/kg/day or methylprednisolone 1 to 2 mg/kg/day) treatment should be initiated. Corticosteroids should be tapered over the course of at least 4 to 6 weeks. Some refractory cases may require infliximab or other immunosuppressive therapy.
- Grade 4: in general, permanent discontinuation of study intervention is recommended, with the exception of endocrinopathies that have been controlled by hormone replacement.

Permanent treatment discontinuation is required in case of immune-related Grade 4 rash/inflammatory dermatitis, nephritis, autoimmune hemolytic anemia, hemolytic uremic syndrome, aplastic anemia, immune thrombocytopenia, acquired thrombotic thrombocytopenic purpura, inflammatory arthritis, myositis, and polymyalgia-like syndrome.

For Grade 4 immune-related lymphopenia, permanent treatment discontinuation will be required, if lymphopenia is considered immune-related in nature, no clear alternative explanation exists for the event, and Grade 4 lymphopenia does not resolve within 14 days. Permanent treatment discontinuation is not required when the AE is manifested by a single laboratory value out of normal range without any clinical correlates. In this case, treatment should be held until the etiology is determined. If the event is not considered immune-related and resolves to Grade  $\leq 1$ , restarting treatment may be considered.

For Grade 1 immune-related pneumonitis: continue treatment. If clinically indicated, monitor participants weekly or more frequently as needed with history, physical examination, and pulse oximetry. If symptoms appear and/or changes in the physical examination are noted, treat as Grade 2.

For myositis: in case of management with rituximab, treatment should be discontinued.

For organ/system specific management guidelines, see the guideline tables in Appendix 5.

Recommended guidance and management for specific irAEs are provided in the current NCCN guideline available at http://www.nccn.org.

## **6.9.3** TGF-β Inhibition Mediated Skin Reactions

TGF- $\beta$  inhibition mediated skin reactions, including hyperkeratosis, KA, and/or cSCCs, are important identified risks and AESI for bintrafusp alfa.

Skin assessments are performed at Screening and every 6 weeks for all participants per Schedule of Activities (Table 1). Baseline skin assessments include a detailed medical history of genetic or iatrogenic skin conditions, skin type, significant UV exposure/sun damage of skin, geographical location, and occupational or environmental exposure to radiation or chemicals.

Skin AEs appear to be related to both mechanisms of bintrafusp alfa; anti-PD-L1 and anti-TGF-β:

1. Immune-related skin AEs possibly mediated by PD-L1 inhibition (e.g., rash or maculo-papular rash, distributed typically on trunk and uniformly on limbs).

Immune-related skin AEs should be managed according to the recommended guidance and management for specific irAEs as per published guidelines (see Appendix 5). Treatment typically include use of emollients, non-sedating antihistamines for pruritus, targeted use of potent topical steroids to most inflamed lesions; oral corticosteroids in highly symptomatic case.

2. Skin AEs, possibly due to TGF-β inhibition, including hyperkeratosis, KA and/or cSCC, are important identified risks for bintrafusp alfa. The distribution of lesions tends to be in sun-exposed areas.

Management guidelines for potential TGF-β inhibition mediated skin reactions are:

- 1. Discontinuation or interruption is not required in most cases. Continuation of treatment should be evaluated by the Investigator.
- 2. Emollients may continue to be used.
- 3. Diagnostic and treatment plan should be developed in collaboration between Investigator and dermatologist. In general, treatment of TGF-β inhibition mediated skin lesions such as hyperkeratosis, KA and cSCC should be based on local guidelines/standard of care. Lesion evaluation should include excision biopsy of one representative lesion to confirm diagnosis.
- 4. Treatment and follow-up for KA and cSCC will depend on number and localization of lesions.
  - For single lesions: Full excision may be recommended.
  - In case of multiple lesions or location not suitable for full excision, other treatment options may be offered by the dermatologist, such as:
  - Mohs surgery, cryotherapy, or other standard treatment options depending on the pathology.
  - Use of retinoids, if recommended by dermatologist, may be considered after discussion with Medical Monitor.
- 5. Close clinical follow-up for re-evaluation, resolution, or potential recurrence should be implemented.
- 6. Spontaneous resolution of KA lesions without surgical intervention has been observed, typically occurring within weeks after discontinuing bintrafusp alfa.
- 7. The number and localization of lesions, diagnosis (including histopathological diagnosis), treatment, and outcome should be appropriately documented in the eCRF.

Consult with study Medical Monitor, as needed, for management of TGF-β inhibition mediated skin reactions.

#### 6.9.4 Anemia

Anemia is an AESI (refer to IB) and important identified risk for bintrafusp alfa. Notably, there are many reasons for anemia in patients with advanced cancer, therefore, a thorough investigation of new anemia cases of unspecified etiology is requested.

For new anemia events, items queried may include, but are not limited to, detailed relevant past medical and treatment history, bruising tendency, history of blood transfusions and/or dependency, and a request for an updated eCRF including details such as concomitant medications, all laboratory data, updated dosing information and, recent tumor evaluation scans.

General guidance for anemia management and evaluation:

- 1. Participants must enter the study with Hgb values at least 9 g/dL; routine blood test parameters are required as in the Schedule of Activities (Table 1).
- 2. All relevant hematologic testing for anemias should be done prior to a blood transfusion, if clinically feasible.
- 3. Transfusion should be performed at the discretion of the Investigator based on clinical assessment and considered when the participant experiences significant anemia. An attempt should be made to initiate work-up (as specified below) for the cause of anemia prior to transfusion, if clinically feasible, to not confound this work-up. In general, blood transfusions and erythroid growth factors are permitted as clinically indicated.

Guidance for evaluation of suspected anemias is provided in Table 6.

#### Table 6 Evaluation Guidance of Suspected Anemia Adverse Events

#### Baseline Anemia Evaluation (Prior to Transfusion, if feasible)

CBC with differential (e.g., Hgb, hematocrit, MCV, reticulocytes counts, ANC).

Peripheral blood smear for cell morphological assessment.

Complete metabolic panel including liver panel-LFTs, bilirubin, LDH, renal function, and other chemistries, if indicated:

- 1. Coagulation factors (PT, PTT, INR)
- 2. Urinalysis including culture
- 3. Iron panel (TIBC, ferritin, Fe)
- 4. Serum folate, B12 values
- 5. TSH/hormonal panel
- 6. Fecal-occult blood testing
- 7. Erythropoietin

#### Further Recommendation Based on Suspected Etiology (in Addition to Baseline Anemia Testing)

| Consider hematology consultation. Consider blood transfusion at clinical discretion. |
|---|
| Consider blood transfusion at clinical discretion. Consider surgical/interventional radiology consultation. Consider imaging, as clinically indicated (e.g., FAST scan, CT scan, MRI, angiography). Consider endoscopy (upper/lower). |
| Hematology consultation. Consider bone marrow aspiration/morphologic evaluation. |

ANC=absolute neutrophil count, CBC=complete blood count, CT=computed tomography, FAST=Focused assessment with sonography for trauma, Fe=iron, Hgb=hemoglobin, INR=international normalized ratio, LDH=lactate dehydrogenase, LFT=liver function test, MCV=mean corpuscular volume, MRI=magnetic resonance imaging, PT=prothrombin time, PTT=partial thromboplastin time, TIBC=total iron binding capacity, TSH=thyroid-stimulating hormone.

## 6.9.5 Bleeding Events

Bleeding events are AESIs and considered an important identified risk for bintrafusp alfa (refer to the IB).



### 6.9.5.1 Mucosal/Non-Tumor Bleeding

Participants treated with bintrafusp alfa were commonly reported with mild to moderate mucosal AEs such as epistaxis, hemoptysis, gingival bleeding and hematuria. In general, these reactions resolve without discontinuation of treatment.

For Grade 2 non-tumor bleeding, see Section 6.8 for general management of Grade 2 treatment-related TEAEs.

For Grade 3 non-tumor bleeding, study intervention must be permanently discontinued unless an alternative explanation can be identified (such as concomitant use of antithrombotic agents, traumatic event, etc.). In case of alternative explanations for the Grade 3 bleeding event, study intervention should be held until the event recovers to Grade  $\leq 1$ .

For Grade 4 non-tumor bleeding, treatment must be permanently discontinued if no alternative explanation is identified.

## 6.9.5.2 Tumor Bleeding

Participants treated with bintrafusp alfa were reported in lower frequencies, with Grade  $\geq 3$  hemorrhages including tumor bleeding. For Grade  $\geq 2$  tumor bleeding, study intervention must be held until the event recovers to Grade  $\leq 1$ . Treatment should be permanently discontinued if the Investigator considers the participant to be at risk for additional severe bleeding.

#### 6.9.6 Other Potential Risks

## 6.9.6.1 Impaired Wound Healing

Impaired wound healing is considered an important potential risk (a theoretical risk-based on literature findings) for bintrafusp alfa, given the role of TGF- $\beta$  in wound healing. Management should be discussed with the Medical Monitor for participants requiring surgery during the study. It is recommended to hold study intervention for approximately 4 weeks after major surgery for observation. Postoperative wound healing will be closely monitored.

## 6.9.6.2 Embryofetal Toxicity

Embryofetal toxicities are a known risk of the PD-1/PD-L1 targeting class and are considered important potential risks for bintrafusp alfa. Animal models link the PD-1/PD-L1 signaling pathway with maintenance of pregnancy through induction of maternal immune tolerance to fetal tissue. An appropriate contraception warning is provided as part of the inclusion criteria. Pregnant and breastfeeding women are not allowed in the bintrafusp alfa study, and adequate contraceptive measures are recommended during the study to minimize or eliminate the potential risk to the developing fetus.

Respective safety measures comprise of inclusion/exclusion criteria for participation in clinical studies with bintrafusp alfa, guidance for prevention, monitoring, and medical management of potential risks, as well as guidance on study intervention interruption or discontinuation.

## 7 Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

## 7.1 Discontinuation of Study Intervention

Participants may be discontinued from study intervention for any of the following reasons, one reinitiating course of treatment may be allowed (see Section 7.1.2.1).

- A participant may discontinue from the study intervention at any time at his/her own request (i.e., withdrawal of consent), and without giving a reason.
- Occurrence of an exclusion criterion, which is clinically relevant and affects the participant's safety, if discontinuation is considered necessary by the Investigator and/or Sponsor.
- A participant may be discontinued at any time at the discretion of the Investigator for safety, behavioral, compliance, or administrative reasons (See Section 6.8 and Section 6.9 for TEAEs and AESIs that require treatment discontinuation, respectively).
- PD per RECIST 1.1 plus subsequent confirmation (repeat imaging 4 to 6 weeks after initial determination of PD), with the exception that participants receiving treatment may continue past PD if the participant's ECOG PS has remained at least stable, and, if in the opinion of the Investigator, the participant may benefit from continued treatment (see Section 7.1.3). A participant with significant symptomatic disease progression and/or clinical deterioration should be discontinued prior to confirmation of PD per RECIST 1.1.
- Unacceptable toxicity
- Some TEAEs and AESIs require withdrawal from treatment. See Section 6.8 and Section 6.9 for additional details.
- Drug must not be given to a known pregnant participant (see Appendix 3).
- Use of a prohibited concomitant drug, as defined in Section 6.5.2, where the predefined consequence is withdrawal from the study intervention.

In case of discontinuation from the study intervention:

- The day of End-of-Treatment Visit will correspond to the day of withdrawal (or within 7 days).
- An attempt should be made to perform all assessments scheduled for the End-of-Treatment Visit if possible. If not possible, the most clinically relevant assessments and appropriate eCRFs for the End-of-Treatment Visit should be prioritized as feasible.
- Participants will be asked to continue Safety Follow-up and Survival Follow-up, which includes the collection of data on survival, and subsequent anticancer therapy. After completion of the follow-up period or after the End-of-Treatment Visit, whichever is applicable, the appropriate eCRF section for Study Termination must be completed.
- If the participant is enrolled into a new study or any new therapy post-withdrawal from study intervention, the Safety Follow-up Visit should be scheduled prior to the start of the new treatment irrespective of the 28-day Safety Follow-up period.

The Schedule of Activities specifies the data to collect at study intervention discontinuation and follow-up, and any additional evaluations that need to be completed.

### 7.1.1 Temporary Discontinuation

See Section 6.8 and Section 6.9 for guidance on temporary discontinuation from study intervention.

## 7.1.2 Rechallenge

#### 7.1.2.1 Reinitiation

One reinitiating course of treatment at the same dose and schedule and treatment duration up to 24 months is allowed at the discretion of the Investigator and agreement of the Medical Responsible for:

• Participants who are experiencing SD, PR, or CR at the time of discontinuation, and then subsequently develop disease progression after stopping therapy, but prior to the End of the Study.

#### OR

• Participants who are discontinued due to an AE that are subsequently well managed or resolved after stopping therapy, but prior to the End of the Study.

The participant should reinitiate treatment at the treatment phase visit where they left off according to the Schedule of Activities (Table 1). Participants who reinitiate treatment should stay on study and should be treated and monitored according the Schedule of Activities for the rest of the study.

Prior to reinitiation, the Investigator will need to confirm that the benefit of reinitiating treatment outweighs any risk involved, such as that which led to initial treatment discontinuation. For participants with only SD at the time of discontinuation, the Investigator should confirm that no other reasonable treatment options are available. In addition, to be eligible for reinitiation, the participant must not have previously withdrawn consent for this study and should have been followed up with regular eCRF documented evaluation scans up to reinitiation of treatment.

A new baseline scan must be performed prior to reinitiation of study intervention. Additionally, relevant safety laboratory assessments, including both full hematology and full chemistry results within 2 weeks, must be available and verified. The clinical Investigator will determine whether additional evaluation and work-up are required on a case-by-case basis. A discussion with the study team is warranted to determine whether PK/biomarker testing is indicated upon restarting treatment.

### 7.1.3 Treatment Beyond Progression

## 7.1.3.1 Treatment Beyond Initial Progression

Participants will receive bintrafusp alfa as outlined in the Schedule of Activities until disease progression. Bintrafusp alfa may continue past the initial determination of disease progression according to RECIST v1.1 as long as the following criteria are met:

- Treatment with bintrafusp alfa is ongoing.
- No new unacceptable treatment or disease-related toxicity.
- Tolerance of study interventions.
- At least stable ECOG PS.
- Treatment beyond progression will not delay an imminent intervention to prevent serious complications of disease progression (e.g., CNS metastases).

A radiographic assessment should be performed within 4 to 6 weeks of original PD to determine whether there has been a decrease in the tumor size, or continued PD. The assessment of clinical benefit should be balanced by clinical judgment as to whether the participant is clinically deteriorating and unlikely to receive any benefit from continued treatment with bintrafusp alfa.

## 7.1.3.2 Treatment Beyond Confirmed Progression

After confirmed PD, if the Investigator feels that the participant continues to achieve clinical benefit by continuing treatment, the participant should remain on the study and continue to receive monitoring according to the Schedule of Activities. The decision to continue treatment beyond confirmed PD should be discussed with the Medical Monitor and documented in the study records.

Participants who continue beyond progression will be evaluated for further tumor response as per the protocol schedule. Treatment should be discontinued permanently upon documentation of further, unequivocal, disease progression unless there are no alternative therapeutic options and the benefit-risk assessment is favorable in consultation between the Investigator and the Medical Monitor. In case of continuation of treatment beyond PD, treatment will be discontinued once any other criteria for withdrawal are met.

# 7.1.3.3 Continuation of Study Intervention After Local Treatment of Disease Progression

If disease progression is due to brain metastasis, participants may continue study interventions after the local treatment of the brain lesions provided that the above criteria are met in addition to the following:

- Tumor assessment showing disease progression has been performed and was documented according to RECIST 1.1 prior to the procedure.
- Brain metastases have been treated locally and are clinically stable for at least 2 weeks prior to reinitiation of study interventions.

- There are no ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable).
- Participants must be either off steroids or on a stable or decreasing dose of  $\leq 10$  mg daily prednisone (or equivalent).
- Benefit-risk assessment to continue study intervention is favorable under consideration of any alternative treatment options as assessed by the Investigator.

In addition, if disease progression is mainly due to a metastatic lesion which in the opinion of the Investigator may be surgically removed, participants may continue study interventions after the local treatment of such a lesion provided that:

- Tumor assessment showing disease progression has been performed and was documented according to RECIST 1.1. prior to the procedure.
- It has been at least 2 weeks and the participant has fully recovered from the surgery.
- Benefit-risk assessment to continue study intervention is favorable under consideration of any alternative treatment options as assessed by the Investigator.

## 7.2 Participant Discontinuation/Withdrawal from the Study

A participant may withdraw from the study at any time, at his/her own request or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, compliance, or administrative reasons.

At the time of discontinuing from the study, if possible, a discontinuation visit will be conducted, as listed in the Schedule of Activities. The Schedule of Activities specifies the data to collect at study discontinuation and follow-up, and any additional evaluations that need to be completed.

If the participant withdraws consent for future involvement in the study, any data collected up to that point may still be used, but no future data can be generated, and any biological samples collected will be destroyed (refer to the Main ICF).

A participant has the right at any time to request destruction of any biological samples taken. The Investigator must document this in the site study records.

## 7.3 Lost to Follow-Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions will be taken if a participant fails to return to the clinic for a required study visit:

• The site will attempt to contact the participant and reschedule the missed visit as soon as possible, counsel the participant on the importance of maintaining the assigned visit schedule, and ascertain if the participant wants to or should continue in the study.

- Before a participant is deemed "lost to follow-up", the Investigator or designee will make every effort to regain contact with the participant: 1) where possible, make 3 telephone calls; 2) if necessary, send a certified letter (or an equivalent local method) to the participant's last known mailing address, and 3) if a participant has given the appropriate consent, contact the participant's general practitioner or caretaker (where allowed by local regulations) for information. These contact attempts should be documented in the participant's medical record.
- If the participant continues to be unreachable, he/she will be considered to have withdrawn from the study.

## 8 Study Assessments and Procedures

Study assessments and procedures and their timing are summarized in the Schedule of Activities.

**No** protocol waivers or exemptions are allowed.

Immediate safety concerns should be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.

Adherence to the study design requirements, including those specified in the Schedule of Activities, is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The Investigator will maintain a screening log to record details of all participants screened, to confirm eligibility, and if applicable, record reasons for screening failure.

Prior to performing any study assessments that are not part of the participant's routine medical care, the Investigator will obtain written informed consent as specified in Appendix 2.

Procedures conducted as part of the participant's routine medical care (e.g., blood count) and obtained before signing of the Main ICF may be used for screening or baseline purposes provided the procedures met the protocol-specified criteria and were performed within the time frame defined in the Schedule of Activities.

## 8.1 Efficacy Assessments and Procedures

Contrast-enhanced computed tomography (CT) imaging of chest/abdomen/pelvis covering the area from the superior extent of the thoracic inlet to well below the symphysis pubis is the first choice of imaging modality. If a participant should not receive iodinated contrast medium, or due to radiation protection reasons, magnetic resonance imaging (MRI) of the same area, using gadolinium enhancement according to local procedure as permitted in conjunction with unenhanced CT of the chest from the thoracic inlet to the inferior costophrenic recess should be done. Regarding MRI for new lesions, in case of doubt, possible new lesions should be followed up on serial MRI before new disease is definitively confirmed. Alternatively, biopsy can be done. The same method should be used per participant throughout the study and preferably the same machines. Brain enhanced MRI (preferably) or enhanced brain CT and/or bone scans should be performed at baseline only for participants suspected to have metastases in these sites. A central

imaging laboratory will be used to read and interpret all CT/MRI/bone scan data; however, treatment decisions will be made by the treating Investigator.

Baseline scans are taken within 28 days prior to treatment. Disease must be measurable with at least 1 uni-dimensionally measurable lesion outside the CNS by RECIST 1.1 assessed by the Investigator. All the scans performed at baseline that are required for RECIST 1.1 assessment need to be repeated at subsequent visits for tumor assessment using the same method, except for brain or bone scans that are negative at baseline. For brain or bone scans that are negative at baseline, no follow-up scans are performed unless there are new symptoms or biochemical changes which suggest PD in these regions. In general, lesions detected at baseline need to be followed using the same imaging methodology and preferably the same imaging equipment at subsequent tumor evaluation visits.

Assessments previously obtained as part of routine clinical care may be used as the baseline assessment if performed within 28 days prior to start of treatment and satisfies tumor assessment requirements as noted in this section.

Participants will be evaluated every 8 weeks within the first 12 months of the participant's first dose, then every 12 weeks through Long-term Follow-up, as scheduled in Table 1.

Confirmation of CR or PR should be performed preferably at the regularly scheduled assessment intervals, but no sooner than 4 weeks after the initial documentation. Confirmation of PR can be confirmed at an assessment later than the next assessment after the initial documentation of PR provided PD does not occur between.

Diagnosis of disease progression based solely on nodal enlargement within 8 weeks of coronavirus vaccination should be made with extreme caution, particularly if in axillary and/or supraclavicular nodes on the ipsilateral side to vaccination and verified with hindsight if possible.

Tumor responses according to RECIST 1.1 will be assessed by the Investigator and an IRC and documented in the eCRF (all measurements should be recorded in metric notation).

## 8.2 Safety Assessments and Procedures

The safety profile of the study intervention will be assessed through the recording, reporting and analysis of baseline medical conditions, AEs, physical examination findings, vital signs, electrocardiograms (ECGs), and laboratory tests.

Comprehensive assessment of any potential toxicity experienced by each participant will be conducted starting when the participants give informed consent and throughout the study. The Investigator will report any AEs, whether observed by the Investigator or reported by the participant. During Prescreening, only AEs associated with study procedures should be recorded. The reporting period is specified in Section 8.3.1.

The safety assessments will be performed according to the Schedule of Activities (Table 1). Periodic evaluations of the study data will be conducted by the study team to ensure safety and the validity and scientific merit of the study (see Section 8.2.4).

Ongoing events at the 12-week Safety Follow-up Visit should continue to be monitored and documented until resolution or resolution with sequelae. All serious adverse events (SAEs) ongoing at the End-of-Treatment Visit must be monitored and followed up by the Investigator until stabilization or until the outcome is known, unless the participant is documented as "lost to follow-up". Reasonable attempts to obtain this information must be made and documented. It is also the responsibility of the Investigator to ensure that any necessary additional therapeutic measures and follow-up procedures are performed.

If a liver function test is elevated in an HBV- or HCV-positive participant, HBV deoxyribonucleic acid (DNA) or HCV ribonucleic acid (RNA) must be monitored to exclude the possibility of reactivation of viral hepatitis. In case of viral reactivation, follow the HBV and HCV management guidelines.

## 8.2.1 Physical Examinations

- Vital signs, physical examinations, and ECOG PS will be conducted at Screening and at subsequent visits as indicated in the Schedule of Activities (Table 1). These should be documented in the eCRF.
- A complete physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, and neurological systems.
- A brief physical examination (at all other scheduled visits other than Screening) will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen.
- Investigators should pay special attention to clinical signs related to previous serious illnesses.
- General status, such as asthenia or appetite, should be evaluated at baseline. Pre-existing symptoms of underlying conditions and/or signs of infection should be investigated as clinically indicated.
- Abnormal findings are to be re-assessed at subsequent visits.

## 8.2.2 Vital Signs

- Height (at Screening Visit only) and weight will be measured and recorded.
- Vital signs including body temperature, pulse rate, respiratory rate, and blood pressure will be assessed and recorded in the eCRF.
- Vital signs will be measured in a semi-supine position after 5 minutes rest and will include temperature, systolic and diastolic blood pressure, and pulse and respiratory rate.
- Blood pressure and pulse measurements will be assessed with a completely automated device. Manual techniques will be used only if an automated device is not available.
- Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones).

## 8.2.3 Electrocardiograms

Single 12-lead ECGs will be obtained as outlined in the Schedule of Activities (Table 1) using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.

## 8.2.4 Clinical Safety Laboratory Assessments

- Blood and urine samples will be collected for the clinical laboratory tests listed in Appendix 6 at the time points listed in the Schedule of Activities (Table 1). All samples should be clearly identified.
- Additional tests may be performed at any time during the study, as determined necessary by the Investigator or required by local regulations.
- The tests will be performed by the local laboratory.
- The Sponsor must receive a list of the local laboratory normal ranges before shipment of study intervention(s). Any changes to the ranges during the study must be forwarded to the Sponsor or designated organization.
- The Investigator must review each laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the eCRF. The laboratory reports must be filed with the source documents.
- If a participant has a clinically significant abnormal laboratory test value that is not present at baseline, the test should be closely monitored until the test value has returned to the normal range or the Investigator has determined that the abnormality is chronic or stable.
- The report of the results must be retained as a part of the participant's medical record or source documents. Pregnancy testing (serum or highly sensitive urine test, as required by local regulations) will be conducted at monthly intervals during study intervention administration and at the time points specified in the Schedule of Activities (Table 1), including at the end of relevant systemic exposure of the study intervention.
- HIV testing is not mandatory. History of HIV infection will be collected, if known, as part of the medical history. If a test is performed at any point in Screening or while on study, a site must consent the participant for HIV testing as per local standard guidance.

#### 8.3 Adverse Events and Serious Adverse Events

The definitions of an AE and a SAE are in Appendix 4.

# 8.3.1 Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

The AE reporting period for safety surveillance begins when the participant is initially included in the study (date of first signature of informed consent/date of first signature of first informed consent) and continues until the 28-day Safety Follow-up Visit, defined as 28 days ( $\pm$  5 days) after the last study intervention administration. After this visit, all SAEs and nonserious

treatment-related AEs should be documented until the last Safety Follow-up Visit, defined as 12 weeks (± 2 weeks) after the last study intervention. Ongoing events at the 12-week Safety Follow-up Visit should continue to be monitored and documented until resolution or resolution with sequelae, unless the participant is documented as "lost to follow-up".

During Prescreening, only AEs associated with study procedures should be recorded.

Any SAE assessed as related to study intervention must be recorded and reported, as indicated in Appendix 4, whenever it occurs, irrespective of the time elapsed since the last administration of study intervention.

The method of recording, evaluating, and assessing causality of AEs (including SAEs) and the procedures for completing and transmitting SAE reports are in Appendix 4.

## 8.3.2 Method of Detecting Adverse Events and Serious Adverse Events

At each study visit, the participant will be queried on changes in his or her condition. During the reporting period, any unfavorable changes in the participant's condition will be recorded as AEs, regardless if reported by the participant or observed by the Investigator.

Complete, accurate and consistent data on all AEs experienced for the duration of the reporting period (defined below) will be reported on an ongoing basis in the appropriate section of the eCRF. All SAEs must be additionally documented and reported using the appropriate Report Form as specified in Appendix 4.

## **8.3.3** Follow-up of Adverse Events and Serious Adverse Events

Adverse events are recorded and assessed continuously throughout the study, as specified in Section 8.3.1 and are assessed for their outcome at the 28-day Safety Follow-up Visit.

All SAEs ongoing at the at the 28-day Safety Follow-up Visit must be monitored and followed up by the Investigator until stabilization or until the outcome is known, unless the participant is documented as "lost to follow-up". Reasonable attempts to obtain this information must be made and documented. It is also the responsibility of the Investigator to ensure that any necessary additional therapeutic measures and follow-up procedures are performed. Further information on follow-up procedures is given in Appendix 4.

#### **Monitoring of Specific Adverse Events**

If monitoring is warranted for certain treatment-related TEAEs for safety issues, the treating physician or Investigator is requested to follow the participant during the post-treatment Long-term Follow-up phase until the end of study period or the participant is "lost to follow-up" and report the management and outcome of AEs to the Sponsor.

## **8.3.4** Regulatory Reporting Requirements for Serious Adverse Events

The Sponsor will send appropriate safety notifications to Health Authorities in accordance with applicable laws and regulations.

The Investigator must comply with any applicable site-specific requirements related to the reporting of SAEs (particularly deaths) involving study participants to the Independent Ethics Committee/Independent Review Board (IEC/IRB) that approved the study.

In accordance with International Council for Harmonisation Good Clinical Practice, the Sponsor/designee will inform the Investigator of findings that could adversely affect the safety of participants, impact the conduct of the study, or alter the IEC's/IRB's approval/favorable opinion to continue the study. In line with respective regulations, the Sponsor/designee will inform the Investigator of AEs that are both serious and unexpected and considered to be related to the administered product ("suspected unexpected serious adverse reactions" or SUSARs). The Investigator should place copies of Safety Reports in the Investigator Site File. National regulations regarding Safety Report notifications to Investigators will be considered.

When specifically required by regulations and guidelines, the Sponsor/designee will provide appropriate Safety Reports directly to the concerned lead IEC/IRB and will maintain records of these notifications. When direct reporting is not clearly defined by national or site-specific regulations, the Investigator will be responsible for promptly notifying the concerned IEC/IRB of any Safety Reports provided by the Sponsor/designee and of filing copies of all related correspondence in the Investigator Site File.

For studies covered by the European Directive 2001/20/EC, the Sponsor's responsibilities regarding the reporting of SAEs/SUSARs/Safety Issues will be carried out in accordance with that Directive and with the related Detailed Guidance documents.

## 8.3.5 Pregnancy

Only pregnancies the Investigator considers to be related to the study intervention (e.g., resulting from a drug interaction with a contraceptive method) are AEs. However, all pregnancies with an estimated conception date during the period defined in Section 8.3.1 must be recorded in the AE page/section of the eCRF for both pregnancies in female participants and pregnancies in female partners of male participants. The Investigator must notify the Sponsor/designee in an expedited manner of any pregnancy using the Pregnancy Report Form, which must be transmitted by the same process specified for SAE reporting in Appendix 4, section on Reporting Serious Adverse Events.

Investigators must actively follow-up, document and report on the outcome of all these pregnancies, even if the participants are withdrawn from the study.

The Investigator must notify the Sponsor/designee of these outcomes using the Pregnancy Report Form. If an abnormal outcome occurs, the SAE Report Form will be used if the participant sustains an event and the Parent-Child/Fetus AE Report Form if the child/fetus sustains an event. Any

abnormal outcome (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) must be reported in an expedited manner, as specified in Section 8.3.1, while normal outcomes must be reported within 45 days after delivery.

In the event of a pregnancy in a participant occurring during the study, the participant must be discontinued from study intervention. The Sponsor/designee must be notified without delay and the participant must be followed as indicated above.

#### 8.4 Treatment of Overdose

For this study, any dose of bintrafusp alfa greater than 2 times (i.e., > 2400 mg) of the planned dose administered within a 24-hour time period will be considered an overdose.

Of note: In the dose-escalation study (EMR200647-001), participants safely received up to 30 mg/kg bintrafusp alfa every 2 weeks (including those with doses > 2400 mg) with no observed maximum tolerated dose (refer to the IB). Safety at significantly higher doses has not been clinically evaluated.

- In case of overdose with clinical correlation, symptomatic treatment must be used; there are no known antidotes for the compound.
- In the event of an overdose, the study intervention infusion should be discontinued, and participants should be observed closely for any signs of toxicity. Supportive treatment should be provided if clinically indicated.

Even if it not associated with an AE or a SAE, any overdose is recorded in the eCRF and reported to drug safety in an expedited manner. Overdoses are reported on a SAE Report Form, following the procedure in Appendix 4, section on Reporting Serious Adverse Events.

If an AE occurs resulting from an overdose, it should follow SAE reporting criteria as indicated in Appendix 4.

#### 8.5 Pharmacokinetics

- Whole blood samples of approximately 3.5 mL will be collected for measurement of serum concentrations of bintrafusp alfa, as specified in the Schedule of Activities. The actual date and time (24-hour clock time) of each sample will be recorded to calculate actual time elapsed since the prior dose administration.
- The quantification of bintrafusp alfa in serum will be performed using a validated immunoassay method. Concentrations will be used to evaluate the PK of bintrafusp alfa.
- Remaining samples collected for analyses of bintrafusp alfa concentration may also be used to
  evaluate immunogenicity, safety or efficacy aspects related to concerns arising during or after
  the study.

Details on processes for collection and shipment of these samples are in the Laboratory Manual. Retention time and possible analyses of samples after the end of study are specified in the respective ICF.

Pharmacokinetic and antidrug antibody (ADA) samples will be collected according to Table 2. Pharmacokinetic and ADA samples collected at the same time points may be used interchangeably if the dedicated sample has insufficient quantity as the participants will have consented to all collections and tests.

The PK parameters will be summarized using descriptive statistics (Table 7). Individual as well as mean concentration-time plots will be depicted.

The following PK parameters will be calculated, when appropriate:

Table 7 **Pharmacokinetic Parameters** 

| Symbol | Definition |
|---|---|
| CEOI | The concentration observed immediately at the end of infusion |
| Ctrough | The concentration observed immediately before next dosing (corresponding to predose or trough concentration for multiple dosing) |

#### 8.6 **Pharmacodynamics**

Not applicable.

#### 8.7 **Pharmacogenetics**

- Where local regulations and IRB/IEC allow, a blood sample will be collected for DNA analysis from consenting participants. Participation in pharmacogenetic research is optional. Participants who do **not** wish to participate in the pharmacogenetic research may still participate in the study.
- In the event of DNA extraction failure, a replacement sample for pharmacogenetic testing may be requested from the participant. Additional informed consent will not be required to obtain a replacement sample.
- Appendix 8 provides further information on pharmacogenetic research.







## 8.9 Immunogenicity Assessments

- Whole blood samples of approximately 5 mL will be collected for detection of antibodies against bintrafusp alfa in serum, as specified in the Bintrafusp alfa Pharmacokinetic, Immunogenicity Sampling (Table 2). Samples will be collected prior to any bintrafusp alfa administration on the same study day.
- The detection of antibodies to bintrafusp alfa will be performed using a validated assay method with tiered testing of screening, confirmatory and titration. Confirmed positive antibodies may be tested for the presence of neutralizing antibodies and may be further characterized.
- Remaining samples collected for analysis of anti-bintrafusp alfa antibodies may also be used to evaluate bintrafusp alfa concentration during or after the study.
- Details on processes for collection and shipment of these samples are in the Laboratory Manual. Retention time and possible analyses of samples after the end of study are specified in the respective Main ICF.



| CCI | | |
|-----|------|------|
| CCI | | |
| | | <br> |
| | <br> | |



## 9.3 Populations for Analyses

The analysis populations are specified below. The final decision to exclude participants from any analysis population will be made by the team after careful consideration during a data review meeting prior to database lock.

For purposes of analysis, the analysis populations are defined in Table 10.

Table 10Analysis Populations

| Screening (SCR) | All participants, who provided informed consent, regardless of the participant's study intervention status in the study. |
|---|---|
| Safety (SAF) | All participants, who were administered at least 1 infusion of bintrafusp alfa. |
| Full analysis Set (FAS) | All participants, who were administered at least 1 infusion of bintrafusp alfa. |
| Pharmacokinetic (PK) | All participants who complete at least 1 infusion of bintrafusp alfa, and who provide at least 1 sample with a measurable concentration of bintrafusp alfa. |
| Immunogenicity | All participants who were administered at least 1 infusion of bintrafusp alfa and have at least one valid ADA result. |

## 9.4 Statistical Analyses

Full details of all planned analyses will be described in the study Integrated Analysis Plan (IAP). Major modifications of planned analyses will be reflected in a protocol amendment or in the clinical study report (CSR).

In general, continuous variables will be summarized using number (n), mean, median, standard deviation, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages. Proportions are calculated based on the number of participants in the analysis set of interest, unless otherwise specified in the IAP.

## 9.4.1 Efficacy Analyses

Analysis of efficacy variables will also be performed on the Full Analysis Set (FAS) as well as subgroup of interest as listed in Table 3, including but not restricted to PD-L1 expression.

Statistical analysis methods for primary and key secondary efficacy endpoints are summarized in Table 11. Further details will be specified in the IAP.

Table 11 Statistical Analysis Methods for Efficacy Analysis

| Endpoint | Statistical Analysis Methods | | |
|---|---|--|--|
| Primary | | | |
| Confirmed objective response according to RECIST 1.1 assessed by an IRC | The ORR will be determined as the proportion of participants with a confirmed objective response of PR or CR. Confirmation of the response according to RECIST 1.1 will be required no sooner than 4 weeks after the initial documentation of CR or PR. The 95% CI for the ORR will be calculated using the Clopper-Pearson method. | | |
| Key Secondary | | | |
| DOR assessed by an IRC | DOR is defined as the time from first documentation of a confirmed objective response (CR or PR) according to RECIST1.1 to the date of first documentation of objective response of disease progression (PD) or death due to any cause whichever occurs first. The censoring rules for DOR are as described below for PFS. Kaplan-Meier estimates will be provided; | | |
| Endpoint | Statistical Analysis Methods | |
|---|---|--|
| | Median DOR and the 95% CI for the median will be calculated according to Brookmeyer and Crowley (Brookmeyer 1982); Swimmer plots will be provided. | |
| Durable response assessed by an IRC | A durable response is defined as an objective response (CR or PR) according to RECIST 1.1, determined by an IRC, with a duration of at least 6 months. Participants for whom the DOR is censored will be treated as failures (successes) in the analysis of durable response if the censored DOR is before (at least) 6 months. The DRR is defined as the percentage of participants with durable response. The 95% CI for the DRR will be calculated using the Clopper-Pearson method. | |
| PFS according to<br>RECIST 1.1 assessed by<br>an IRC | PFS according to RECIST 1.1, is defined as the time from first administration of study intervention until date of the first documentation of PD or death due to any cause in the absence of documented PD, whichever occurs first. PFS data will be censored on the date of the last adequate tumor assessment for participants who do not have an event (PD or death), for participants who start new anticancer treatment prior to an event, or for participants with an event after 2 or more missing tumor assessments. Participants who do not have a baseline tumor assessment or who do not have any post-baseline tumor assessments will be censored on the date of first administration of study intervention unless death occurred on or before the time of the second planned tumor assessment, in which case the death will be considered an event. Kaplan-Meier estimates will be provided; Median PFS and the 95% CI for the median will be calculated according to Brookmeyer and Crowley (Brookmeyer 1982). | |
| Overall survival | Overall survival is defined as the time from first administration of study intervention to the date of death due to any cause. Participants last known to be alive will be censored at date of last contact. Kaplan-Meier estimates will be provided; Median OS and the 95% CI for the median will be calculated according to Brookmeyer and Crowley (Brookmeyer 1982). | |
| Confirmed Objective response, DOR, DRR, and PFS according to RECIST 1.1 assessed by Investigator | Definition and analyses to be performed on the efficacy endpoints as assessed by Investigator will be similar to the endpoints as assessed by the Investigator, see above. | |

CI= confidence interval, CR=complete response, DOR=duration of response, DRR=durable response rate, IRC=Independent Review Committee, ORR=objective response rate, OS=overall survival, PD=progressive disease, PFS= progression-free survival, PR=partial response, RECIST 1.1=Response Evaluation Criteria in Solid Tumors Version 1.1.

# 9.4.2 Safety Analyses

All safety analyses will be performed on the Safety Analysis population (SAF).

The on-treatment period is defined as the time from the first study intervention administration to the last study intervention administration date +30 days or the earliest date of subsequent anticancer drug therapy minus 1 day, whichever occurs first, unless otherwise stated.

Data collected after reinitiation of treatment will be summarized according to the specifications in the IAP.

Safety endpoints include AEs, AESIs, clinical laboratory assessments, vital signs, physical examination, and ECOG PS as described in Section 8.2.

The definitions, procedures for recording, evaluating, follow-up, and reporting of AEs are described in Appendix 4.

TEAEs are those events with onset dates occurring during the on-treatment period or if the worsening of an event is during the on-treatment period. The incidence of TEAEs, regardless of attribution, and TEAEs defined as possibly related to bintrafusp alfa will be summarized by MedDRA preferred term and system organ class and described in terms of intensity and relationship to bintrafusp alfa. Any AEs with an onset or worsening date after the on-treatment period will be reported separately.

See Table 12 for safety endpoints and statistical analysis methods. The specifics for safety analysis will be defined in the IAP and finalized before database lock.

 Table 12
 Safety Endpoints and Statistical Analysis Methods

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | Not applicable |
| Secondary | The safety endpoints will be tabulated using descriptive statistics. |
| Occurrence of TEAEs | Participants will be analyzed according to the actual treatment they receive. |
| and treatment-related | The safety endpoints will be analyzed using descriptive statistics. |
| AEs | The incidence of TEAEs, SAEs, treatment-related AEs, AESIs, and irAEs will be summarized by preferred term and system organ class for each treatment arm, and described in terms of severity and relationship to treatment. |
| | The worst on-treatment grades for chemistry and hematology laboratory results will be summarized. |
| | Shifts in toxicity grading from Baseline to highest grade during the on-treatment period will be displayed. |
| | For laboratory tests without an NCI-CTCAE grade definition results will be presented categorically (e.g., below, within, or above normal limits). |
| | Further details of safety analyses (including AEs, clinical laboratory assessments, vital signs, physical examination, ECG parameters, and ECOG PS) will be provided in the IAP. |

AE=adverse event, AESI=adverse event of special interest, ECG=electrocardiogram, ECOG PS=Eastern Cooperative Oncology Group performance status, IAP=Integrated Analysis Plan, irAE=immune-related adverse event, NCI-CTCAE=National Cancer Institute Common Terminology Criteria for Adverse Events, SAE=serious adverse event, TEAE=treatment-emergent adverse event.

# 9.4.3 Other Analyses

Analysis of efficacy variables may be performed on subgroups of interest as needed. The detailed subgroups will be outlined in the IAP.

Serum concentrations of bintrafusp alfa will be determined by a validated method at the times listed in the Bintrafusp alfa Pharmacokinetic, Immunogenicity Sampling (Table 2). Samples for ADA assessments will be collected per the Schedule of Activities. The immunogenicity testing strategy is in accordance with current regulatory guidance documents and industry best practices.

PK, immunogenicity and biomarker will be specified in the IAP finalized before database lock. The PopPK analysis and exposure-response may be performed using

combined data from several bintrafusp alfa clinical studies and will be specified in a separate IAP. Integrated analyses across studies, such as the PopPK analysis, exposure-response and biomarker analyses will be presented separately from the main CSR.

## 9.4.4 Sequence of Analyses

The planned efficacy analyses are specified below. Details of all planned analyses will be defined in the IAP:

- The interim analysis on unconfirmed response as assessed by the Investigator will be performed 4 months after the accrual of the first 15 participants.
- The primary analysis on objective response as assessed by an IRC will be performed 8 months after the accrual of the last participant. At the same time, the analysis of durable response of at least 6 months assessed by an IRC will be performed to support the ORR data. The analysis of DOR and PFS will be performed as well to support efficacy assessment of bintrafusp alfa.
- A final analysis will be performed for evaluation of OS 24 months after accrual of last participant.
- If the study continues after the cutoff date for final analysis, subsequent analyses may be performed.

### 10 References

Adams S, Schmid P, Rugo HS, et al. Pembrolizumab monotherapy for previously treated metastatic triple-negative breast cancer: cohort A of the phase II KEYNOTE-086 study. Ann Oncol. 2019;30(3):397-404.

Brahmer JR, Lacchetti C, Schneider BJ, et al. Management of immune-related adverse events in patients treated with immune checkpoint inhibitor therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Oncol Pract. 2018;14(4):247-49.

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics. 1982;38:29-41.

Champiat S, Lambotte O, Barreau E, et al. Management of immune checkpoint blockade dysimmune toxicities: A collaborative position paper. Ann Oncol. 2016;27(4):559-74.

Desruisseau S, Palmari J, Giusti C, et al. Determination of TGF[beta]1 protein level in human primary breast cancers and its relationship with survival. Br J Cancer. 2006;94:239-46.

Dirix LY, Takacs I, Jerusalem G, et al. Avelumab, an anti-PD-L1 antibody, in patients with locally advanced or metastatic breast cancer: a phase 1b JAVELIN Solid Tumor study. Breast Cancer Res Treat. 2018;167(3):671-86.

Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45:228-47.

Emens LA, Cruz C, Eder JP, et al. Long-term clinical outcomes and biomarker analyses of Atezolizumab therapy for patients with metastatic triple-negative breast cancer: A Phase 1 Study. JAMA Oncol. 2019;5(1):74-82.

FDA Guidance on Cancer Clinical Trial Eligibility Criteria: Patients with HIV, Hepatitis B Virus, or Hepatitis C Virus Infections, March 2019.

Gobbi H, Arteaga CL, Jensen RA, et al. Loss of expression of transforming growth factor beta type II receptor correlates with high tumour grade in human breast in-situ and invasive carcinomas. Histopathology. 2000;36:168-77.

Gorsch SM, Memoli VA, Stukel TA, et al. Immunohistochemical Staining for Transforming Growth Factor  $\beta 1$  Associates with Disease Progression in Human Breast Cancer. Cancer Res. 1992;52:6949-52.

Goudie DR, D'Alessandro M, Merriman B, et al. Multiple self-healing squamous epithelioma is caused by a disease-specific spectrum of mutations in TGFBR1. Nat Genet. 2011;43(4):365-9.

Hammond ME, Hayes DF, Dowsett M, et al. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer. J Clin Oncol. 2010a;28(16):2784-95.

Hammond ME, Hayes DF, Dowsett M, et al. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer (unabridged version). Arch Pathol Lab Med. 2010b;134(7):e48-72.

Ismail-Khan R, Bui MM. A Review of triple-negative breast cancer. Cancer Control. 2010;17:173-6.

Locke G, Zhang Y, Ojalvo LS, et al. Identification of a tumor biomarker in advanced triplenegative breast cancer that predicts response to bintrafusp alfa (M7824), a bifunctional fusion protein targeting transforming growth factor-β and programmed death ligand 1. Cancer Res. 2019a;80(suppl; abstr P3-09-13).

Locke G, Zhang Y, Ojalvo LS, et al. Identification of a tumor biomarker in advanced triple-negative breast cancer that predicts response to bintrafusp alfa (M7824), a bifunctional fusion protein targeting transforming growth factor-β and programmed death ligand 1. Presented at: 2019 San Antonio Breast Cancer Symposium, December 10–14, 2019b; San Antonio, TX, USA [abstract 1132].

Mittendorf EA, Philips AV, Meric-Bernstam F, et al. PD-L1 expression in triple-negative breast cancer. Cancer Immunol Res. 2014;2(4):361-70.

Morris JC, Tan AR, Olencki TE, et al. Phase I study of GC1008 (fresolimumab): a human anti-transforming growth factor-beta (TGFβ) monoclonal antibody in patients with advanced malignant melanoma or renal cell carcinoma. PLoS One. 2014;9(3):e90353.

National Comprehensive Cancer Network® guidelines. Hepatobiliary cancers. Version 3. 2018. Available at: https://www.nccn.org/patients/guidelines/hepatobiliary/4/.

Padua D, Zhang XH, Wang Q, et al. TGFbeta primes breast tumors for lung metastasis seeding through angiopoietin-like 4. Cell. 2008;133(1):66-77.

Spira A, Awada A, Isambert N, et al. Bintrafusp alfa (M7824), a bifunctional fusion protein targeting transforming growth factor-β and programmed death ligand 1, in advanced triplenegative breast cancer: preliminary results from a phase 1 cohort. Cancer Res. 2019;80(suppl; abstr P3-09-06).

Schmid P, Adams S, Rugo HS, et al. Atezolizumab and Nab-Paclitaxel in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2018;379:2108-21.

Schmid P, Adams S, Rugo HS, et al. IMpassion130: updated overall survival (OS) from a global, randomized, double-blind, placebo-controlled, Phase III study of atezolizumab (atezo) + nab-paclitaxel (nP) in previously untreated locally advanced or metastatic triple-negative breast cancer (mTNBC). J Clin Oncol. 2019;37:1003-1003.

Thuault S, Valcourt U, Petersen M, et al. Transforming growth factor-beta employs HMGA2 to elicit epithelial-mesenchymal transition. J Cell Biol. 2006;174(2):175-83.

Wolff AC, Hammond ME, Hicks DG, et al. Recommendations for human epidermal growth factor receptor 2 testing in breast cancer: American Society of Clinical Oncology/College of American Pathologists clinical practice guideline update. J Clin Oncol. 2013;31(31):3997-4013.

Wu J, Zhang S, Shan J, et al. Elevated HMGA2 expression is associated with cancer aggressiveness and predicts poor outcome in breast cancer. Cancer Lett. 2016;376(2):284-92.

# 11 Appendices

# **Appendix 1** Abbreviations

| Appendix 1 Appreviations | |
|--------------------------|------------------------------------------|
| ADA | Antidrug antibody |
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALT | Alanine aminotransferase |
| anti-PD-L1 | Anti-programmed death-ligand 1 |
| ART | Antiretroviral therapy |
| ASCO | American Society of Clinical Oncology |
| AST | Aspartate aminotransferase |
| CI | Confidence interval |
| CNS | Central nervous system |
| CR | Complete response |
| CrCL | Creatinine clearance |
| CRO | Contract Research Organization |
| cSCC | Cutaneous squamous cell carcinoma |
| CSR | Clinical study report |
| CT | Computed tomography |
| DNA | Deoxyribonucleic acid |
| DOR | Duration of response |
| DRR | Durable response rate |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HBV | Hepatitis B virus |
| HCV | Hepatitis C virus |
| HER2 | Human epidermal growth factor receptor 2 |
| Hgb | Hemoglobin |
| HIV | Human immunodeficiency virus |
| HMGA2 | High Mobility Group AT-Hook 2 |

| Harmonal rankacament thereny |
|--------------------------------------------------------------------------|
| Hormonal replacement therapy Integrated Analysis Plan |
| Integrated Analysis Plan Investigator's Prochure |
| Investigator's Brochure |
| Informed consent form |
| International Council for Harmonisation |
| Independent Ethics Committee |
| Immunohistochemistry |
| Immune-related adverse event |
| Independent Review Board |
| Independent Review Committee |
| Infusion-related reaction |
| Keratoacanthoma |
| Medical Dictionary for Regulatory Activities |
| Magnetic resonance imaging |
| National Comprehensive Cancer Network |
| National Cancer Institute Common Terminology Criteria for Adverse Events |
| Objective response rate |
| Overall survival |
| Progressive disease |
| programmed death-1 |
| Programmed death-ligand 1 |
| Progression-free survival |
| Pharmacokinetic(s) |
| Population pharmacokinetic |
| Partial response |
| Performance status |
| Response Evaluation Criteria in Solid Tumors Version 1.1 |
| Ribonucleic acid |
| Recommended Phase II dose |

| SAE | Serious adverse event |
|-------|-----------------------------------------------|
| SD | Stable Disease |
| SUSAR | Suspected unexpected serious adverse reaction |
| TEAE | Treatment-emergent adverse event |
| TGF-β | Transforming growth factor-β |
| TMB | Tumor mutational burden |
| TNBC | Triple Negative Breast Cancer |
| ULN | Upper limit of normal |
| WOCBP | Woman of childbearing potential |

# **Appendix 2** Study Governance

#### **Financial Disclosure**

Investigators and Sub-Investigators will provide the Sponsor with sufficient, accurate financial information, as requested, for the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. This information is required during the study and for 1 year after completion of the study.

#### **Informed Consent Process**

- The Investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative (where allowed by local laws and regulations) and answer all questions on the study.
- Participants must be informed that their participation is voluntary.
- Participants or their legally-authorized representative (where allowed by local laws and regulations) will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50; the Japanese ministerial ordinance on GCP; local regulations; ICH guidelines; Health Insurance Portability and Accountability Act (HIPAA) requirements, where applicable; and the IRB/IEC or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- If the ICF is updated during their participation in the study, participants must be re-consented to the most current, approved version.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.
- The original signed and dated consent will remain at the Investigator's site and must be safely archived so that it can be retrieved at any time for monitoring, auditing and inspection purposes.
- Participants who are rescreened are required to sign a new ICF.

#### **Data Protection**

- The Sponsor will assign a unique identifier to participants after obtaining their informed consent. All participant records or datasets transferred to the Sponsor will contain the identifier only; participant names or any identifiable information will not be transferred.
- The Sponsor must inform participants that their personal study-related data will be used per local data protection and privacy laws. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other Sponsor-appointed, authorized personnel, by appropriate IRB/IEC members, and by regulatory authority inspectors. All such persons will strictly maintain participants' confidentiality.

## **Study Administrative**

The Coordinating Investigator listed on the title page represents all Investigators for decisions and discussions on this study, per ICH GCP. The Coordinating Investigator will provide expert medical input and advice on the study design and execution and is responsible for the review and signoff of the clinical study report.

The study will appear in the following clinical studies registries: ClinicalTrials.gov and EudraCT.

This study requires a significant logistic and administrative structure for its efficient execution. Details of structures and associated procedures will be defined in a separate Investigator Site File.

This will be prepared under the supervision of the Clinical Trial Leader in close collaboration with the responsible units at the Sponsor.

The Sponsor will coordinate the study and will provide the support for a Contract Research Organization (CRO) for some activities of the study. Sponsor Global Clinical Operations will perform oversight of the activities performed by the CRO.

The Clinical Trial Supplies department of the Sponsor will supply the study medication of bintrafusp alfa, which will be distributed to the sites by Fisher Clinical Services.

Participant enrollment will be managed by an interactive voice response system or an interactive web response system.

Safety laboratory assessments will be performed locally by investigational sites. Pharmacokinetic (PK), CCI and pharmacogenetic (PGx) assessments will be performed under the responsibility and/or supervision of the Sponsor.

The Global Drug Safety Department, Merck KGaA, Darmstadt, Germany, or its designated representatives will supervise drug safety and the timely reporting of adverse events (AEs) and serious adverse events (SAEs).

Quality assurance of the study conduct will be performed by the Development Quality Assurance Department, Merck KGaA, Darmstadt, Germany.

The department of Global Biostatistics will supervise the statistical analyses (with the exception of the PK data analyses that will be outsourced to a CRO).

## **Regulatory and Ethical Considerations**

This study will be conducted in accordance with the protocol and the following:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
- Applicable ICH GCP Guidelines

## • Applicable laws and regulations

The Investigator must submit the protocol, protocol amendments (if applicable), ICF, Investigator Brochure, and other relevant documents (e.g., advertisements) to an IRB/IEC and the IRB/IEC must review and approve them before the study is initiated.

Any protocol amendments (i.e., changes to the protocol) will be documented in writing and require IRB/IEC approval before implementation of changes, except for changes necessary to eliminate an immediate hazard to study participants. When applicable, amendments will be submitted to the appropriate Health Authorities.

The Investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/IEC annually or more frequently per the IRB's/IEC's requirements, policies, and procedures.
- Notifying the IRB/IEC of SAEs or other significant safety findings, as required by IRB/IEC procedures
- Providing oversight of the study conduct at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

The protocol and any applicable documentation will be submitted or notified to the Health Authorities in accordance with all local and national regulations for each site.

#### **Review Committee**

The Independent Review Committee (IRC) will be involved in the study. The IRC will be composed of a minimum of 3 members. The role of the IRC will be to review radiographic image findings for the determination of the best overall response (objective response) and date of disease progression for each participant. The full membership, mandate, and processes of the IRC will be detailed in the IRC charter.

## **Emergency Medical Support**

The Sponsor or designee will provide Emergency Medical Support cards to participants for use during the study. These provide the means for participants to identify themselves as participating in a clinical study. Also, these give health care providers access to any information about this participation that may be needed to determine the course of medical treatment for the participant. The information on the Emergency Medical Support card may include the process for emergency unblinding (if applicable).

The first point of contact for all emergencies will be the clinical study Investigator caring for the participant. Consequently, the Investigator agrees to provide his or her emergency contact information on the card. If the Investigator is available when an event occurs, they will answer any

questions. Any subsequent action (e.g., unblinding) will follow the standard process established for Investigators.

When the Investigator is not available, the Sponsor provides the appropriate means to contact a Sponsor (or designee) physician. This includes provision of a 24-hour contact number at a call center, whereby the health care providers will be given access to the appropriate Sponsor (or designee) physician to assist with the medical emergency.

## **Clinical Study Insurance and Compensation to Participants**

Insurance coverage will be provided for each country participating in the study. Insurance conditions shall meet good local standards, as applicable.

## **Clinical Study Report**

After study completion, the Sponsor will write a clinical study report in consultation with the Coordinating Investigator.

#### **Publication**

The results of this study may be published or presented at scientific meetings. If this is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows Merck to protect proprietary information and to provide comments.

The Sponsor will comply with the requirements for publication of study results. Per standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a Coordinating Investigator will be designated by agreement.

Authorship will be determined by agreement and in line with International Committee of Medical Journal Editors authorship requirements.

## **Dissemination of Clinical Study Data**

After completion of the study, a CSR will be written by the Sponsor in consultation with the Coordinating Investigator following the guidance in ICH Topic E3 and will be submitted in accordance with local regulations.

Any and all scientific, commercial, and technical information disclosed by the Sponsor in this protocol or elsewhere should be considered the confidential and proprietary property of the Sponsor. The Investigator shall hold such information in confidence and shall not disclose the information to any third party except to such of the Investigator's employees and staff who had been made aware that the information is confidential and who are bound to treat it as such and to whom disclosure is necessary to evaluate that information. The Investigator shall not use such information for any purpose other than for determining mutual interest in performing the study and, if the parties decide to proceed with the study, for the purpose of conducting the study.

The Investigator understands that the information developed from this clinical study will be used by the Sponsor in connection with the development of the study intervention and therefore may be disclosed as required to other clinical Investigators, to the USA Food and Drug Administration, and to other government agencies. The Investigator also understands that, to allow for the use of the information derived from the clinical study, the Investigator has the obligation to provide the Sponsor with complete test results and all data developed in the study.

No publication or disclosure of study results will be permitted except under the terms and conditions of a separate written agreement.

## **Data Quality Assurance**

All participant study data will be recorded on printed or electronic CRFs or transmitted to the Sponsor or designee electronically (e.g., laboratory data). The Investigator is responsible for verifying that data entries are complete, accurate, legible, and timely by physically or electronically signing the eCRF. Details for managing CRFs are in the Operations Manual.

The Investigator must maintain accurate documentation (source data) that supports the information in the eCRF.

The Investigator must permit study-related monitoring, quality assurance audits, IRB/IEC review, and regulatory agency inspections and provide direct access to the study file and source data.

Monitoring details describing strategy (e.g., risk-based initiatives in operations and quality such as Risk Management and Mitigation Strategies and Analytical Risk-Based Monitoring), methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are in the Monitoring Plan or contracts.

The Sponsor or designee is responsible for data management of this study, including quality checking of the data and maintaining a validated database. Database lock will occur once quality control and quality assurance procedures have been completed. PDF files of the CRFs will be provided to the Investigators at study completion.

Study monitors will perform ongoing source data verification to confirm that data in the eCRF are accurate, complete, and verifiable; that the safety and rights of participants are being protected; and that the study is being conducted per the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

Records and documents, including signed ICFs, pertaining to the conduct of this study must be retained by the Investigator for 15 years after study completion, unless local regulations, institutional policies, or the Sponsor requires a longer retention. No records may be destroyed during the retention period without the Sponsor's written approval. No records may be transferred to another location or party without the Sponsor's written notification.

## **Source Documents**

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected.

The Investigator must keep a paper or electronic file (medical file and original medical records) at the site for each study participant. The file must identify each participant, contain the following demographic and medical information for the participant, and should be as complete as possible:

Participant's full name, date of birth, sex, height, and weight

- Medical history and concomitant diseases
- Prior and concomitant therapies (including changes during the study)
- Study identifier (i.e., the Sponsor's study number) and participant's study number.
- Dates of entry into the study (i.e., signature date on the informed consent) and each visit to the site
- Any medical examinations and clinical findings predefined in the protocol
- All AEs
- Date that the participant left the study, including any reason for early withdrawal from the study or study intervention, if applicable.

All source data must be filed (e.g., CT or MRI scan images, ECG recordings, and laboratory results). Each document must have the participant number and the procedure date; ideally, printed by the instrument used for the procedure. As necessary, medical evaluation of these records should be performed, documented, signed and dated by the Investigator.

Data recorded on printed or electronic CRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

The study monitors will use printouts of electronic files for source data verification. These printouts must be signed and dated by the Investigator and kept in the study file.

Source documents are stored at the site for the longest possible time permitted by the applicable regulations, and/or as per ICH GCP guidelines, whichever is longer. The Investigator ensures that no destruction of medical records is performed without the Sponsor's written approval.

Definition of what constitutes source data is found in eCRF guidelines.

## **Study and Site Closure**

The Sponsor reserves the right to close the study site or terminate the study at any time and for any reason. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a site closure visit has been completed.

The Investigator may initiate site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or Investigator may include:

- Failure of the Investigator to comply with the protocol, the requirements of the IRB/IEC or local Health Authorities, the Sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the Investigator
- Discontinuation of further development of the Sponsor's compound

#### **Contraception** Appendix 3

Contraceptive use by males and females will be consistent with local regulations on contraception methods for those participating in clinical studies.

## Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile, as specified below.

If fertility is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before the first dose of study intervention, consider additional evaluation.

#### A WOCBP is **not**:

- 1. Premenarchal
- 2. A premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy.

Documentation can come from the site personnel's review of the female's medical records, medical examination, or medical history interview.

For a female with permanent infertility due to an alternate medical cause other than the above, (e.g., Mullerian agenesis, androgen insensitivity), Investigator discretion applies to determine study entry.

## 3. A postmenopausal female:

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
  - o A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in a female not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, more than 1 FSH measurement is required in the postmenopausal range.
- A female on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if she wishes to continue her HRT during the study. Otherwise, she must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### CONTRACEPTIVES ALLOWED DURING THE STUDY

## **Highly Effective Methods That Have Low User Dependency**

- Implantable progestogen-only hormone contraception associated with inhibition of ovulation
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion
- Vasectomized partner: a highly effective contraceptive method provided that the partner is the sole sexual partner of a WOCBP and the absence of sperm has been confirmed. Otherwise, use an additional highly effective method of contraception. The spermatogenesis cycle is approximately 90 days.

Highly Effective Methods That Are User Dependent

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation

- Oral
- Intravaginal
- Transdermal
- Injectable

Progestogen-only hormone contraception associated with inhibition of ovulation

- Oral
- Injectable

Sexual abstinence: a highly effective method only if defined as refraining from intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study.

#### **Notes:**

Contraceptive use by men or women is consistent with local regulations on the use of contraceptive methods for clinical study participants.

Highly effective methods are those with a failure rate of < 1% per year when used consistently and correctly.

Typical use failure rates differ from those when used consistently and correctly.

Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method (LAM) are not acceptable methods of contraception for this study. Male condom and female condom cannot be used together (due to risk of failure with friction).



# Appendix 4 Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definitions**

#### **Adverse Event**

An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, regardless if it is considered related to the medicinal product.

For surgical or diagnostic procedures, the condition/illness leading to such a procedure is considered as the AE rather than the procedure itself.

The Investigator is required to grade the severity or toxicity of each AE.

Investigators will reference the NCI-CTCAE, v5.0 (publication date: 27 November 2017), a descriptive terminology that can be used for AE reporting.

A general grading (severity/intensity; hereafter referred to as severity) scale is provided at the beginning of the above referenced document, and specific event grades are also provided.

If the severity for an AE is not specifically graded by NCI-CTCAE, the Investigator is to use the general NCI-CTCAE definitions of Grade 1 through Grade 5, using his or her best medical judgment.

The 5 general grades are:

- Grade 1 or Mild
- Grade 2 or Moderate
- Grade 3 or Severe
- Grade 4 or Life-threatening
- Grade 5 or Death

Any clinical AE with severity of Grade 4 or 5 must also be reported as an SAE. However, a laboratory abnormality of Grade 4, such as anemia or neutropenia, is considered serious only if the condition meets one of the serious criteria specified below.

If death occurs, the primary cause of death or event leading to death should be recorded and reported as an SAE. "Fatal" will be recorded as the outcome of this specific event and death will

not be recorded as separate event. Only, if no cause of death can be reported (e.g., sudden death, unexplained death), the death per se might then be reported as an SAE.

Investigators must also systematically assess the causal relationship of AEs to study intervention (including any other non-study interventions, radiation therapy, etc.) using the following definitions. Decisive factors for the assessment of causal relationship of an AE to the study intervention include, but may not be limited to, temporal relationship between the AE and the study intervention, known side effects of study intervention, medical history, concomitant medication, course of the underlying disease, and study procedures.

Unrelated: Not reasonably related to the study intervention. AE could not medically

(pharmacologically/clinically) be attributed to the study intervention under study in this clinical study protocol. A reasonable alternative explanation must be available.

Related: Reasonably related to the study intervention. AE could medically

(pharmacologically/clinically) be attributed to the study intervention under study in

this clinical study protocol.

## Abnormal Laboratory Findings and Other Abnormal Investigational Findings

Abnormal laboratory findings and other abnormal investigational findings (e.g., on an ECG trace) should not be reported as AEs unless they are associated with clinical signs and symptoms, lead to study intervention discontinuation or are considered otherwise medically important by the Investigator. If a laboratory abnormality fulfills these criteria, the identified medical condition (e.g., anemia or increased ALT) must be reported as the AE rather than the abnormal value itself.

## **Serious Adverse Events**

An SAE is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening. Life-threatening refers to an event in which the participant is at risk of death at the time of the event, not an event that hypothetically might have caused death if it was more severe.
- Requires inpatient hospitalization or prolongs an existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly or birth defect
- Is otherwise considered to be medically important. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered as SAEs when, based upon appropriate medical judgment, they may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

For the purposes of reporting, any suspected transmission of an infectious agent via a study intervention is also considered an SAE, as specified below for reporting SAEs.

#### Events that Do Not Meet the Definition of an SAE

Elective hospitalizations to administer, or to simplify study intervention or procedures (e.g., an overnight stay to facilitate intravenous therapy) are not considered SAEs. However, all events leading to unplanned hospitalizations or unplanned prolongation of an elective hospitalization (i.e., undesirable effects of any administered treatment) must be documented and reported as SAEs.

#### Events Not to Be Considered as AEs/SAEs

Medical conditions present at the initial study visit that do not worsen in severity or frequency during the study are defined as Baseline Medical Conditions, and are not to be considered AEs.

## AE/SAEs Observed in Association with Disease Progression

Progression of the disease/disorder being studied assessed by measurement of lesions on radiographs or other methods as well as associated clinical signs or symptoms (including laboratory abnormalities) should not be reported as an (S)AE, unless the participant's general condition is more severe than expected for the participant's condition and/or unless the outcome is fatal within the adverse event reporting period, as defined in Section 8.3.2.

## **Adverse Events of Special Interest**

Infusion-related reactions including hypersensitivity, irAEs, TGF-β inhibition mediated skin reactions, anemia, and bleeding AEs are all considered as AESIs for bintrafusp alfa.

## Other Adverse Events to be Reported Following a Specialized Procedure

Not applicable.

## Recording and Follow-Up of AE and/or SAE

It is important that each AE report include a description of the event, its duration (onset and resolution dates and also onset and resolution times, when it is important to assess the time of AE onset relative to the recorded study intervention administration time), its severity, its causal relationship with the study intervention, any other potential causal factors, any treatment given or other action taken, including dose modification or discontinuation of the study intervention, and its outcome. In addition, serious cases should be identified, and the appropriate seriousness criteria documented.

Specific guidance is in the eCRF Completion and Monitoring Conventions provided by the Sponsor.

## **Reporting Serious Adverse Events**

#### **Serious Adverse Events**

In the event of any new SAE occurring during the reporting period, the Investigator must immediately (within a maximum of 24 HOURS after becoming aware of the event) inform the Sponsor or its designee using the electronic SAE report form in the Electronic Data Capture (EDC) system.

Reporting of SAEs using a paper report form is required as a back-up method only for an EDC system failure. Names, addresses, and telephone and fax numbers will be included on the paper form. All information from the paper form must be transcribed into the electronic form as soon as the system becomes available.

In exceptional circumstances, an SAE (or follow-up information) may be reported by telephone; in these cases, an electronic SAE report form must be completed immediately thereafter.

Relevant pages from the eCRF may be provided in parallel (e.g., medical history, concomitant drugs). Additional documents may be provided by the Investigator, if available (e.g., laboratory results, hospital report, autopsy report).

The Investigator must respond to any request for follow-up information (e.g., additional information, outcome, final evaluation, other records where needed) or to any question the Sponsor/designee may have on the AE within the same timelines as those noted above for initial reports. This is necessary to ensure prompt assessment of the event by the Sponsor or designee and (as applicable) to allow the Sponsor to meet strict regulatory timelines associated with expedited safety reporting obligations.

Requests for follow-up will usually be made via the study monitor, although in exceptional circumstances the drug safety department may contact the Investigator directly to obtain further information or to discuss the event.

## **Appendix 5** The Recommendations for irAE Management

This appendix provides recommendations to the Investigators for the management of irAEs. The contents are based on the NCCN irAE management guidelines (in Accordance with the Joint American Society of Clinical Oncology Clinical Practice Guidelines and National Comprehensive Cancer Network, Brahmer JR, 2018) and FDA recommendations to require permanent treatment discontinuation for Grade 4 irAEs (unless otherwise indicated in the tables below). Differences with ASCO/NCCN irAE management guidelines as recommended by the FDA are shown in bold and underlined text in the tables below. Critical instructions include the requirement that treatment must be permanently discontinued for the following Grade 4 irAEs toxicities: Rash/inflammatory dermatitis, nephritis, autoimmune hemolytic anemia, hemolytic uremic syndrome, aplastic anemia, immune thrombocytopenia, acquired TTP, and in certain circumstances, lymphopenia.

## **Table of Tables**

| Table A1 | Management of Skin irAEs in Patients Treated With ICPis96 |
|---|---|
| Table A2 | Management of GI irAEs in Patients Treated With ICPis101 |
| Table A3 | Management of Lung irAEs in Patients Treated With ICPis105 |
| Table A4 | Management of Endocrine irAEs in Patients Treated With ICPis106 |
| Table A5 | Management of Musculoskeletal irAEs in Patients Treated With ICPis |
| Table A6 | Management of Renal irAEs in Patients Treated With ICPis115 |
| Table A7 | Management of Nervous System irAEs in Patients Treated With ICPis |
| Table A8 | Management of Hematologic irAEs in Patients Treated With ICPis |
| Table A9 | Management of Cardiovascular irAEs in Patients Treated With ICPis |
| Table A10 | Management of Ocular irAEs in Patients Treated With ICPis131 |

## Table A1 Management of Skin irAEs in Patients Treated With ICPis

#### 1.0 Skin Toxicities

#### 1.1 Rash/inflammatory dermatitis

Definition: Erythema multiforme minor (a targetoid reaction in the skin and mucous membranes usually triggered by infections, such as herpes simplex viruses, but can be associated with an immune-related drug eruption and if progresses to erythema multiforme major, it and can be a harbinger of SCAR, such as SJS), lichenoid (resembling the flat-topped, polygonal, and sometimes scaly or hypertrophic lesions of lichen-planus), eczematous (inflammatory dermatitis characterized by pruritic, erythematous, scaly, or crusted papules or plaques on the skin, which is vulnerable to superinfection, psoriasiform [resembling the well-demarcated, erythematous, and scaly papules and plaques of psoriasis], morbilliform [a nonpustular, nonbullous measles-like exanthematous rash of the skin often referred to as "maculopapular" and without systemic symptoms or laboratory abnormalities, excluding occasional isolated peripheral eosinophilia], palmoplantar erythrodysesthesia [hand-foot syndrome; redness, numbness, burning, itching, and superficial desquamation of the palms and soles], neutrophilic dermatoses [e.g, Sweet syndrome], and others)

Diagnostic work-up

Pertinent history and physical examination

Rule out any other etiology of the skin problem, such as an infection, an effect of another drug, or a skin condition linked to another systemic disease or unrelated primary skin disorder

If needed, a biologic checkup, including a blood cell count and liver and kidney tests

Directed serologic studies if an autoimmune condition is suspected, such as lupus or dermatomyositis: a screening antinuclear antibody test, SS-A/Anti-Ro, SS-B/Anti-La if predominantly photodistributed/photosensitivity, antihistone, double-stranded DNA, and other relevant serologies. Consider expanding serologic studies or diagnostic work-up if other autoimmune conditions are considered based on signs, symptoms Skin biopsy Consider clinical monitoring with use of serial clinical photography

Review full list of patient medications to rule out other drug-induced cause for photosensitivity

| Grading | Management |
|---|---|
| Grading according to CTCAE is a challenge for skin. Instead, severity may be based on BSA, tolerability, morbidity, and duration | |
| G1: Symptoms do not affect the quality of life or controlled with topical regimen and/or oral antipruritic | Continue ICPi Treat with topical emollients and/or mild-moderate potency topical corticosteroids Counsel patients to avoid skin irritants and sun exposure |
| G2: Inflammatory reaction that affects quality of life and requires intervention based on diagnosis | Consider holding ICPi and monitor weekly for improvement. If not resolved, interrupt treatment until skin AE has reverted to Grade 1 Consider initiating prednisone (or equivalent) at dosing 1 mg/kg, tapering over at least 4 weeks In addition, treat with topical emollients, oral antihistamines, and medium- to high-potency topical corticosteroids |
| G3: As G2 but with failure to respond to indicated interventions for a G2 dermatitis | Hold ICPi therapy and consult with dermatology to determine appropriateness of resuming Treat with topical emollients, oral antihistamines, and high-potency topical corticosteroids Initiate (methyl)prednisolone (or equivalent) 1-2 mg/kg, tapering over at least 4 weeks |
| G4: All severe rashes unmanageable with prior interventions and intolerable | Permanently discontinue ICPi Systemic corticosteroids: IV (methyl)prednisolone (or equivalent) dosed at 1-2 mg/kg with slow tapering when the toxicity resolves |

| 1.0 Skin Toxicities | |
|---|---|
| | Monitor closely for progression to severe cutaneous adverse reaction Should admit patient immediately with direct oncology involvement and with an urgent consult by dermatology |

#### 1.2 Bullous dermatoses

Definition: Including bullous pemphigoid or other autoimmune bullous dermatoses, bullous drug reaction Diagnostic work-up

Physical examination

Rule out any other etiology of the skin problem, such as an infection, an effect of another drug, or a skin condition linked to another systemic disease

If needed, a biologic checkup, including a blood cell count, liver, and kidney tests; consider serum antibody tests to rule out bullous pemphigoid or, under the guidance of dermatology, sending patient serum for indirect immunofluorescent testing to rule out other autoimmune blistering diseases

Referral to dermatology for blisters that are not explained by infectious or transient other causes (e.g, herpes simplex, herpes zoster, bullous impetigo, bullous insect bite, friction or pressure blister)

Consider skin biopsy (both hematoxylin and eosin evaluation of lesional skin and direct immunofluorescence evaluation of perilesional skin)

| | blisters are < 10% BSA, asymptomatic, and oninflammatory (such as the case with friction blisters |
|---|---|
| G1: Asymptomatic, blisters covering < 10% BSA and no associated erythema | r pressure blisters), cessation of ICPi is not necessary,<br>nd only observation and/or local wound care is<br>carranted. |
| del<br> mu | /hen symptomatic bullae or erosions, which are eroofed vesicles or bullae, are observed on the skin or nucosal surfaces, the cutaneous irAE is by definition busidered at least G2 |
| Se | ee G2 management recommendations |
| intervention based on diagnosis not meeting criteria for Grade > 2 Blisters covering 10%-30% BSA | old ICPi therapy and consult with dermatology for ork-up and to determine appropriateness of resuming tention given to general local wound care, which icludes plain petrolatum ointment and bandages or lain petrolatum ointment gauze and bandage over any pen erosions, which are left over on the skin after the lister has popped or if the roof of the blister easily oughs off ounsel patients to avoid skin irritants and verexposure to sun, wear protective clothing, use unscreens fork-up for autoimmune bullous disease as above nitiate Class 1 high-potency topical corticosteroid (e.g., obetasol, betamethasone or equivalent) and reassess very 3 days for progression or improvement ow threshold to initiate treatment with prednisone (or quivalent) at 0.5-1 mg/kg dosing and taper over at least 4 weeks lonitor patients with G2 irAEs closely for progression or involvement of greater BSA and/or mucous membrane involvement. Consider following patients osely using serial photography rimer on monitoring for complicated cutaneous diverse drug reactions: |

| 1.0 Skin 7 | Toxicities |
|---|---|
| | Review of systems: Skin pain (like a sunburn), fevers, malaise, myalgias, arthralgias, abdominal pain, ocular discomfort or photophobia, sores or discomfort in the nares, sores or discomfort in the oropharynx, odynophagia, hoarseness, dysuria, sores or discomfort in the vaginal area for women or involving the meatus of the penis for men, sores in the perianal area, or pain with bowel movements |
| | Physical examination: Include vital signs and a full skin examination specifically evaluating all skin surfaces and mucous membranes (eyes, nares, oropharynx, genitals, and perianal area). Assess for lymphadenopathy, facial or distal extremity swelling (may be signs of DIHS/DRESS). Assess for pustules or blisters or erosions in addition to areas of "dusky erythema," which may feel painful to palpation. To assess for a positive Nikolsky sign, place a gloved finger tangentially over erythematous skin and apply friction parallel to the skin surface. Nikolsky sign is positive if this results in detached or sloughing epidermis demonstrating poor attachment of the epidermis to the dermis, which is the case in some autoimmune disorders (eg, pemphigus) and SJS/TEN |
| G3: Skin sloughing covering > 30% BSA with associated pain and limiting self-care ADL | Hold ICPi therapy and consult with dermatology to determine appropriateness of resuming Administer IV (methyl)prednisolone (or equivalent) 1-2 |
| | mg/kg, tapering over at least 4 weeks If bullous pemphigoid is diagnosed, it may be possible to avoid long-term use of systemic corticosteroids and treat with rituximab, as an alternative approach to treating the irAE |
| | Seek infectious disease consultation if patient might have secondary cellulitis or if patient has other infection risk factors, such as neutropenia, etc. |
| G4: Blisters covering > 30% BSA with associated fluid | Permanently discontinue ICPi |
| or electrolyte abnormalities | Admit patient immediately and place under supervision of a dermatologist |
| | Administer IV (methyl)prednisolone (or equivalent) 1-2 mg/kg with tapering over at least 4 weeks when the toxicity resolves |
| | If bullous pemphigoid is diagnosed, it may be possible to avoid long-term use of systemic corticosteroids and treat with rituximab as an alternative approach to treating the irAE |
| 1.3 SCARs, including SJS, TEN, acute generalized exa | Seek infectious disease consultation if patient might have secondary cellulitis or if patient has other infection risk factors, such as neutropenia, etc |

## 1.3 SCARs, including SJS, TEN, acute generalized exanthematous pustulosis, and DRESS/DIHS

Definition: Severe changes in either structure or functions of skin, the appendages or the mucous membranes due to a drug

Diagnostic work-up

Total body skin examination with attention to examining all mucous membranes as well as complete review of systems

Rule out any other etiology of the skin problem, such as an infection, an effect of another drug, or a skin condition linked to another systemic disease

#### 1.0 Skin Toxicities

A biologic checkup, including a CBC with differential test, and liver and kidney function tests, including urinalysis, in addition to the blood work; if the patient is febrile, blood cultures should be considered as well

Skin biopsies to assess for full-thickness epidermal necrosis, as is seen in SJS/TEN, as well as other possible etiologies like paraneoplastic pemphigus or other autoimmune blistering dermatoses or other drug reactions, such as acute generalized exanthematous pustulosis

Consider following patients closely using serial clinical photography

If mucous membrane involvement or blistering is observed on the skin, consider early admission to a burn center for further monitoring and management Primer on monitoring for complicated cutaneous adverse drug reactions:

Review of systems: Skin pain (like a sunburn), fevers, malaise, myalgias, arthralgias, abdominal pain, ocular discomfort or photophobia, sores or discomfort in the nares, sores or discomfort in the oropharynx, odynophagia, hoarseness, dysuria, sores or discomfort in the vaginal area for women or involving the meatus of the penis for men, sores in the perianal area, or pain with bowel movements

Physical examination: Include vital signs and a full skin examination specifically evaluating all skin surfaces and mucous membranes (eyes, nares, oropharynx, genitals, and perianal area). Assess for lymphadenopathy, facial or distal extremity swelling (may be signs of DIHS/DRESS). Assess for pustules or blisters or erosions in addition to areas of "dusky erythema", which may feel painful to palpation. To assess for a positive Nikolsky sign, place a gloved finger tangentially over erythematous skin and apply friction parallel to the skin surface. Nikolsky sign is positive if this results in detached or sloughing epidermis demonstrating poor attachment of the epidermis to the dermis, which is the case in some autoimmune disorders (e.g., pemphigus) and SJS/TEN

| · | |
|---|---|
| Grading | Management |
| All Grades | In cases of suspected SJS or any mucous membrane involvement, discontinue ICPi treatment and monitor closely for improvement, regardless of grade |
| G1: NA | For SCARs, there is no G1 category; if lower BSA is involved with bullae or erosions, there should remain a high concern that this reaction will progress to G3 or G4 |
| G2: Morbilliform ("maculopapular") exanthem covering 10%-30% BSA with systemic symptoms, lymphadenopathy, or facial swelling | Hold ICPi and monitor patients closely every 3 days with G2 irAEs for progression to involvement of greater BSA and/or mucous membrane involvement Consider following patients closely using serial photography |
| | Initiate therapy with topical emollients, oral antihistamines, and medium- to high-strength topical corticosteroids |
| | Consider initiation of prednisone (or equivalent) 0.5-1 mg/kg tapered over at least 4 weeks |
| G3: Skin sloughing covering < 10% BSA with mucosal involvement associated signs (e.g, erythema, purpura, epidermal detachment, mucous membrane detachment) | Hold ICPi therapy and consult with dermatology Treat skin with topical emollients and other petrolatum emollients, oral antihistamines, and high-strength topical corticosteroids; dimethicone may also be offered as an alternative to petrolatum |
| | Administer IV (methyl)prednisolone (or equivalent) 0.5-<br>1 mg/kg and convert to oral corticosteroids on<br>response, wean over at least 4 weeks |
| | Admit to burn and/or consult wound services with attention to supportive care, including fluid and electrolyte balance, minimizing insensible water losses, and preventing infection |
| | Given the immune mechanism of action of these medicines, use of immune suppression is warranted and should be offered |

| 1.0 Skin Toxicities | |
|---|---|
| | For mucous membrane involvement of SJS or TEN, appropriate consulting services should be offered to guide management in preventing sequelae from scarring (e.g., ophthalmology; ear, nose, and throat; urology; gynecology; etc, as appropriate) |
| G4: Skin erythema and blistering/sloughing covering | Permanently discontinue ICPi |
| ≥ 10% to > 30% BSA with associated signs (e.g, erythema, purpura, epidermal detachment, mucous membrane detachment) and/or systemic symptoms and concerning associated blood work abnormalities (e.g, liver function test elevations in the setting of DRESS/DIHS) | Admit patient immediately to a burn unit or ICU with consulted dermatology and wound care services Consider further consultations based on management of mucosal surfaces (e.g, ophthalmology; urology; gynecology; ear, nose, and throat surgery; etc) Initiate IV (methyl)prednisolone (or equivalent) 1-2 mg/kg, tapering when toxicity resolves to normal |
| | IVIG or cyclosporine may also be considered in severe or corticosteroid-unresponsive cases |
| | Consider pain/palliative consultation and/or admission in patients presenting with DRESS manifestations |

Additional considerations: The usual prohibition of corticosteroids for SJS is not relevant here, as the underlying mechanism is a T-cell immunodirected toxicity

Adequate suppression is necessary with corticosteroids or other agents and may be prolonged in cases of DRESS/DIHS

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate

Abbreviations: ADL, activities of daily living; AE, adverse event; BSA, body surface area; CBC, complete blood count; CTCAE, Common Terminology Criteria for Adverse Events; DIHS, drug-induced hypersensitivity syndrome; DRESS, drug reaction with eosinophilia and systemic symptoms; G, Grade; ICPi, immune checkpoint inhibitor; ICU, intensive care unit; irAE, immune-related adverse event; IV, intravenous; IVIG, intravenous immunoglobulin; NA, not applicable; SCAR, severe cutaneous adverse reactions; SJS, Stevens-Johnson syndrome; TEN, toxic epidermal necrolysis.

## Table A2 Management of GI irAEs in Patients Treated With ICPis

#### 2.0 GI Toxicities

#### 2.1 Colitis

Definition: A disorder characterized by inflammation of the colon Diagnostic work-up

G2

Work-up of blood (CBC, comprehensive metabolic panel, TSH, ESR, CRP), stool (culture, Clostridium difficile, parasite, CMV or other viral etiology, ova and parasite) should be performed

Consider testing for lactoferrin (for patient stratification to determine who needs more urgent endoscopy) and calprotectin (to follow-up on disease activity)

Screening laboratories (HIV, hepatitis A and B, and blood quantiferon for TB) to prepare patients to start infliximab should be routinely done in patients at high risk for those infections and appropriately selected patients based on infectious disease expert's evaluation

Imaging (e.g, CT scan of abdomen and pelvis and GI endoscopy with biopsy) should be considered as there is evidence showing that the presence of ulceration in the colon can predict a corticosteroid-refractory course, which may require early infliximab

Consider repeating endoscopy for patients who do not respond to immunosuppressive agents; repeating endoscopy for disease monitoring can be considered when clinically indicated and when planning to resume therapy

#### G3-4

All the work-up listed for G2 (blood, stool, imaging, and scope with biopsy) should be completed immediately Consider repeating endoscopy for patients who do not respond to immunosuppressive agents; repeating endoscopy for disease monitoring should only be considered when clinically indicated and when planning to resume ICPi

| Grading (based on CTCAE for diarrhea, as most often used clinically) | Management |
|---|---|
| All patients | Counsel all patients to be aware of and inform their health care provider immediately if they experience: Abdominal pain, nausea, cramping, blood or mucus in stool or changes in bowel habits, fever, abdominal distention, obstipation, constipation For G2 or higher, consider permanently discontinuing CTLA-4 agents and may restart PD-1, PD-L1 agents if patient can recover to G1 or less; concurrent immunosuppressant maintenance therapy should be considered only if clinically indicated in individual cases |
| G1: Increase of fewer than four stools per day over baseline; mild increase in ostomy output compared with baseline | Continue ICPi; alternatively, ICPi may be held temporarily and resumed if toxicity does not exceed G1 Monitor for dehydration and recommend dietary changes Facilitate expedited phone contact with patient/caregiver May obtain gastroenterology consult for prolonged G1 cases |
| G2: Increase of four to six stools per day over baseline; moderate increase in ostomy output compared with baseline | Should hold ICPi temporarily until patient's symptoms recover to G1; can consider permanently discontinuing CTLA-4 agents and may restart PD-1, PD-L1 agents if patient can recover to G1 or less Concurrent immunosuppressant maintenance therapy (10 mg prednisone equivalent dose) may be offered only if clinically indicated in individual cases May also include supportive care with medications such as Imodium if infection has been ruled out Should consult with gastroenterology for G2 or higher |

| 2.0 GI Toxicities | |
|---|---|
| | Administer corticosteroids, unless diarrhea is transient, starting with initial dose of 1 mg/kg/day prednisone or equivalent |
| | When symptoms improve to G1 or less, taper corticosteroids over at least 4-6 weeks before resuming treatment, although resuming treatment while on low-dose corticosteroid may also be an option after an evaluation of the risks and benefits |
| | EGD/colonoscopy, endoscopy evaluation should be highly recommended for cases Grade ≥ 2 to stratify |
| | patients for early treatment with infliximab based on the endoscopic findings and to determine the safety of resuming PD-1, PD-L1 therapy |
| | Stool inflammatory markers can be considered (lactoferrin and calprotectin) in cases of G2 or higher to differentiate functional versus inflammatory diarrhea, and use calprotectin to monitor treatment response if provider prefers |
| | Repeat colonoscopy is optional for cases of G2 or higher for disease activity monitoring to achieve complete remission, especially if there is a plan to resume ICPi |
| G3: Increase of seven or more stools per day over baseline, incontinence, hospitalization indicated, severe increase in ostomy output compared with baseline, | Should consider permanently discontinuing CTLA-4 agents and may restart PD-1, PD-L1 agents if patient can recover to G1 or less. |
| limiting self-care ADL | Administer corticosteroids (initial dose of 1-2 mg/kg/d prednisone or equivalent) |
| | Consider hospitalization or outpatient facility for patients with dehydration or electrolyte imbalance |
| | If symptoms persist ≥ 3-5 days or recur after improvement, consider administering IV corticosteroid or noncorticosteroid (e.g, infliximab) |
| | Consider colonoscopy in cases where patients have been on immunosuppression and may be at risk for opportunistic infections as an independent cause for diarrhea (i.e, CMV colitis) and for those who are anti-TNF or corticosteroid refractory |
| G4: Life-threatening consequences; urgent intervention | Permanently discontinue treatment |
| indicated | Should admit patient when clinically indicated; patients managed as outpatients should be very closely monitored |
| | Administer 1-2 mg/kg/d methylprednisolone or equivalent until symptoms improve to G1, and then start taper over 4-6 weeks |
| | Consider early infliximab 5-10 mg/kg if symptoms refractory to corticosteroid within 2-3 days Consider lower GI endoscopy if symptoms are refractory despite treatment or there is concern of new infections |
| Additional considerations | |

#### Additional considerations

The use of vedolizumab may be considered in patients refractory to infliximab and/or contraindicated to TNF-a blocker. The decision should be made on an individual basis from gastroenterology and oncology evaluation. This is based on case series showing promising results

Patients with hepatitis and irAE colitis are rare, and management should include permanently discontinuing ICPi and offering other immunosuppressant agents that work systemically for both conditions

#### 2.0 GI Toxicities

Currently, enteritis alone as the cause of diarrhea is uncommon and requires small bowel biopsy as the evaluation tool. It may be managed similar as colitis, including corticosteroid and/or infliximab, etc

#### 2.2 Hepatitis

Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma Diagnostic work-up

Monitor patient for abnormal liver blood tests: AST, ALT, and bilirubin prior to each infusion and/or weekly if G1 liver function test elevations. No treatment is recommended for G1 liver function test abnormality For G2 or higher:

Work-up for other causes of elevated liver enzymes should be tested, viral hepatitis, alcohol history, iron study, thromboembolic event, liver ultrasound, cross-sectional imaging for potential liver metastasis from primary malignancy. If suspicion for primary autoimmune hepatitis is high, can consider ANAs, antismooth muscle antibodies, antineutrophil cytoplasmic antibodies. If patients with elevated alkaline phosphatase alone, g-glutamyl transferase should be tested. For isolated elevation of transaminases, consider checking CK for other etiologies

| Grading | Management |
|---|---|
| All patients | Counsel all patients to be aware of and inform their health care provider immediately if they experience: Yellowing of skin or whites of the eyes Severe nausea or vomiting |
| | Pain on the right side of the abdomen Drowsiness Dark urine (tea colored) Bleeding or bruising more easily than normal Feeling less hungry than usual |
| G1: Asymptomatic (AST or ALT > ULN to 3.0 x ULN and/or total bilirubin > ULN to 1.5 x ULN) | Continue ICPi with close monitoring; consider alternate etiologies Monitor laboratories one to two times weekly Manage with supportive care for symptom control |
| G2: Asymptomatic (AST or ALT > 3.0 to $\leq$ 5 x ULN and/or total bilirubin > 1.5 to $\leq$ 3 x ULN) | Hold ICPi temporarily and resume if recover to G1 or less on prednisone ≤ 10 mg/d For Grade 2 hepatic toxicity with symptoms, may administer corticosteroid 0.5-1 mg/kg/d prednisone or equivalent if the abnormal elevation persists with significant clinical symptoms in 3-5 days Increase frequency of monitoring to every 3 days Infliximab might not be the most appropriate treatment option in the situation of immune-mediated hepatitis given the potential risk of idiosyncratic liver failure (Note: No clear evidence shows the liver toxicity from infliximab from other studies) In follow-up, may resume ICPi treatment followed by taper only when symptoms improve to G1 or less and corticosteroid ≤ 10 mg/d; taper over at least 1 month Patients should be advised to stop unnecessary medications and any known hepatotoxic drugs |
| G3: Symptomatic liver dysfunction, fibrosis by biopsy, compensated cirrhosis, reactivation of chronic hepatitis (AST or ALT 5-20 x ULN and/or total bilirubin 3-10x3 ULN) | Permanently discontinue ICPi Immediately start corticosteroid 1-2 mg/kg methylprednisolone or equivalent If corticosteroid refractory or no improvement after 3 days, consider mycophenolate mofetil or azathioprine (if using azathioprine should test for thiopurine methyltransferase deficiency) Laboratories at daily or every other day; consider inpatient monitoring for patients with AST/ALT > 8 x ULN and/or elevated TB 3 x ULN |

| 2.0 GI Toxicities | |
|---|---|
| | Increase frequency of monitoring to every 1-2 days |
| | Infliximab might not be the most appropriate treatment option in the situation of immune-mediated hepatitis given the potential risk of liver failure (Note: No clear evidence shows that the liver toxicity from infliximab from other studies); alternatives include non—TNF-a agents as systemic immunosuppressants If no improvement is achieved with corticosteroids or for patients on combination therapy with a novel agent, with standard chemotherapy, or with targeted therapy, refer to hepatologist for further pathologic evaluation of hepatitis Corticosteroid taper can be attempted around 4-6 |
| | weeks; re-escalate if needed; optimal duration unclear |
| G4: Decompensated liver function (e.g., ascites, | Permanently discontinue ICPi |
| coagulopathy, encephalopathy, coma; AST or ALT > 20 x ULN and/or total bilirubin > 10 x ULN) | Administer 2 mg/kg/d methylprednisolone equivalents |
| | If corticosteroid refractory or no improvement after 3 days, consider mycophenolate mofetil |
| | Monitor laboratories daily; consider inpatient monitoring |
| | Avoid the use of infliximab in the situation of immune-mediated hepatitis |
| | Hepatology consult if no improvement was achieved with corticosteroid |
| | Corticosteroid taper can be attempted around 4-6 weeks when symptoms improve to G1 or less; reescalate if needed; optimal duration unclear |
| | Consider transfer to tertiary care facility if necessary |
| All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations is moderate. | |

Abbreviations: ADL, activities of daily living; ALT, alanine aminotransferase; ANA, antinuclear antibody; AST, aspartate aminotransferase; CBC, complete blood count, CK, creatine kinase; CMV, cytomegalovirus; CRP, C-reactive protein; CT, computed tomography; CTCAE, Common Terminology Criteria for Adverse Events; CTLA-4, cytotoxic T-cell lymphocyte-associated antigen-4; EGD, esophagogastroduodenoscopy; ESR, erythrocyte sedimentation rate; G, Grade; GI, gastrointestinal; HIV, human immunodeficiency virus; ICPi, immune checkpoint inhibitor; irAE, immune-related adverse event; IV, intravenous; PD-1; programmed death 1; PD-L1, programmed death-ligand 1; TB, tuberculosis; TNF, tumor necrosis factor; TSH, thyroid-stimulating hormone; ULN, upper limit of

CCI CCI

normal.

## Table A3 Management of Lung ir AEs in Patients Treated With ICPis

#### 3.0 Lung Toxicities

#### 3.1 Pneumonitis

Definition: Focal or diffuse inflammation of the lung parenchyma (typically identified on CT imaging)

No symptomatic, pathologic, or radiographic features are pathognomonic for pneumonitis

Diagnostic work-up

Should include the following: CXR, CT, pulse oximetry

For G2 or higher, may include the following infectious work-up: nasal swab, sputum culture and sensitivity, blood culture and sensitivity, urine culture and sensitivity

| Grading | Management |
|---|---|
| G1: Asymptomatic, confined to one lobe of the lung or < 25% of lung parenchyma, clinical or diagnostic observations only | Continue ICPi If clinically indicated. Monitor participants weekly or more frequently as needed with history, physical examination and pulse oximetry; may also offer CXR. May offer one repeat CT scan in 3-4 weeks; in patients who have had baseline testing, may offer a repeat spirometry/DLCO in 3-4 weeks If symptoms appear and/or changes in the physical exam are noted, treat as G2 |
| G2: Symptomatic, involves more than one lobe of the lung or 25%-50% of lung parenchyma, medical intervention indicated, limiting instrumental ADL | Hold ICPi until resolution to G1 or less Prednisone 1-2 mg/kg/d and taper by 5-10 mg/wk over 4-6 weeks Consider bronchoscopy with BAL Consider empirical antibiotics Monitor every 3 days with history and physical examination and pulse oximetry, consider CXR; no clinical improvement after 48-72 hours of prednisone, treat as G3 |
| G3: Severe symptoms, hospitalization required, involves all lung lobes or 50% of lung parenchyma, limiting self-care ADL, oxygen indicated G4: Life-threatening respiratory compromise, urgent intervention indicated (intubation) | Permanently discontinue ICPi Empirical antibiotics; (methyl)prednisolone IV 1-2 mg/kg/d; no improvement after 48 hours, may add infliximab 5 mg/kg or mycophenolate mofetil IV 1 g twice a day or IVIG for 5 days or cyclophosphamide; taper corticosteroids over 4-6 weeks Pulmonary and infectious disease consults if necessary Bronchoscopy with BAL ± transbronchial biopsy Patients should be hospitalized for further management |

#### Additional considerations

GI and Pneumocystis prophylaxis with PPI and Bactrim may be offered to patients on prolonged corticosteroid use (> 12 weeks), according to institutional guidelines

Consider calcium and vitamin D supplementation with prolonged corticosteroid use

The role of prophylactic fluconazole with prolonged corticosteroid use (> 12 weeks) remains unclear, and physicians should proceed according to institutional guidelines

Bronchoscopy + biopsy; if clinical picture is consistent with pneumonitis, no need for biopsy

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate.

Abbreviations: ADL, activities of daily living; BAL, bronchoalveolar lavage; CT, computed tomography; CXR, chest X-ray; DLCO, diffusing capacity of lung for carbon monoxide; G, Grade; GI, gastrointestinal; ICPi, immune checkpoint inhibitor; irAE, immune-related adverse event; IV, intravenous; IVIG, intravenous immunoglobulin; PPI, proton pump inhibitor.



#### Table A4 Management of Endocrine irAEs in Patients Treated With ICPis

| 4.0 | End | locrine | Toxicity |
|-----|-----|---------|----------|

Counsel patients to inform their health care provider immediately if they experience any changes in their health since their last visit, especially any of the following:

Headaches that will not go away or unusual headache

patterns

Vision changes

Rapid heartbeat

Increased sweating

Extreme tiredness or weakness

Muscle aches

Weight gain or weight loss

Dizziness or fainting

Feeling more hungry or thirsty than usual

Hair loss

Changes in mood or behavior, such as decreased sex

drive, irritability, or forgetfulness Feeling cold

Constipation

Voice gets deeper

Urinating more often than usual

Nausea or vomiting

Abdominal pain

## 4.1 Thyroid

#### 4.1.1 Primary hypothyroidism

Definition: Elevated TSH, normal or low FT4

Diagnostic work-up

TSH and FT4 every 4-6 weeks as part of routine clinical monitoring on therapy or for case detection in

| symptomatic patients | |
|---|---|
| Grading | Management |
| G1: TSH < 10 mIU/L and asymptomatic G2: Moderate symptoms; able to perform ADL; TSH persistently > 10 mIU/L | Should continue ICPi with close follow-up and monitoring of TSH, FT4 May hold ICPi until symptoms resolve to baseline |
| | Consider endocrine consultation |
| | Prescribe thyroid hormone supplementation in symptomatic patients with any degree of TSH elevation or in asymptomatic patients with TSH levels that persist > 10 mlU/L (measured 4 weeks apart) |
| | Monitor TSH every 6-8 weeks while titrating hormone replacement to normal TSH FT4 can be used in the short term (2 weeks) to ensure adequacy of therapy in those with frank hypothyroidism where the FT4 was initially low |
| | Once adequately treated, should monitor thyroid function (at least TSH) every 6 weeks while on active ICPi therapy or as needed for symptoms to ensure appropriate replacement; repeat testing annually or as indicated by symptoms once stable |
| G3-4: Severe symptoms, medically significant or life-<br>threatening consequences, unable to perform ADL | Hold ICPi until symptoms resolve to baseline with appropriate supplementation Endocrine consultation |

| 4.0 Endocrine Toxicity | |
|---|---|
| | May admit for IV therapy if signs of myxedema (bradycardia, hypothermia) Thyroid supplementation and reassessment as in G2 |

#### Additional considerations

For patients without risk factors, full replacement can be estimated with an ideal body weight–based dose of approximately 1.6  $\mu g/kg/d$ 

For elderly or fragile patients with multiple comorbidities, consider titrating up from low dose, starting at 25-50 mg Extreme elevations of TSH can be seen in the recovery phase of thyroiditis and can be watched in asymptomatic patients to determine whether there is recovery to normal within 3-4 weeks

Under guidance of endocrinology, consider tapering hormone replacement and retesting in patients with a history of thyroiditis (initial thyrotoxic phase)

Adrenal dysfunction, if present, must always be replaced before thyroid hormone therapy is initiated

## 4.1.2 Hyperthyroidism

Definition: Suppressed TSH and high normal or elevated FT4 and/or triiodothyronine

Diagnostic work-up

Monitor TSH, FT4 every 4-6 weeks from the start of therapy or as needed for case detection in symptomatic patients

Consider TSH receptor antibodies if there are clinical features and suspicion of Grave disease (e.g, ophthalmopathy)

Close monitoring of thyroid function every 2-3 weeks after diagnosis to catch transition to hypothyroidism in patients with thyroiditis and hyperthyroidism

| Grading | Management |
|---|---|
| G1: Asymptomatic or mild symptoms | Can continue ICPi with close follow-up and monitoring of TSH, FT4 every 2-3 weeks until it is clear whether there will be persistent hyperthyroidism (see below) or hypothyroidism (see 4.1.1) |
| | Consider holding ICPi until symptoms return to baseline |
| | Consider endocrine consultation |
| | b-Blocker (e.g, atenolol, propranolol) for symptomatic relief |
| | Hydration and supportive care |
| | Corticosteroids are not usually required to shorten duration |
| | For persistent hyperthyroidism (> 6 weeks) or clinical suspicion, work-up for Graves disease (TSI or TRAb) and consider thionamide (methimazole or PTU) Refer to endocrinology for Graves disease |
| G3-4: Severe symptoms, medically significant or life-<br>threatening consequences, unable to perform ADL | Hold ICPi until symptoms resolve to baseline with appropriate therapy Endocrine consultation |
| | b-Blocker (e.g, atenolol, propranolol) for symptomatic relief |
| | For severe symptoms or concern for thyroid storm, hospitalize patient and initiate prednisone 1-2 mg/kg/d or equivalent tapered over 1-2 weeks; consider also use of SSKI or thionamide (methimazole or PTU). |

#### Additional considerations

Thyroiditis is transient and resolves in a couple of weeks to primary hypothyroidism or normal. Hypothyroidism can be treated as above. Graves disease is generally persistent and is due to increased thyroid hormone production that can be treated with antithyroid medical therapy. Physical examination findings of ophthalmopathy or thyroid bruit are diagnostic of Graves and should prompt early endocrine referral.



| 4.0 Endocrine Toxicity | |
|---|---|
| 4.2 Adrenal – primary adrenal insufficiency | |
| Definition: Adrenal gland failure leading to low morning cortisol, high morning ACTH, as well as hyponatremia and hyperkalemia with orthostasis and volume depletion due to loss of aldosterone | |
| Diagnostic work-up for patients in whom adrenal insufficiency is suspected: | |
| Evaluate ACTH (AM), cortisol level (AM) | |
| Basic metabolic panel (Na, K, CO <sub>2</sub> , glucose) Consider ACTH stimulation test for indeterminate | |
| results | |
| If primary adrenal insufficiency (high ACTH, low cortisol) is found biochemically: | |
| Evaluate for precipitating cause of crisis such as infection Perform an adrenal CT for metastasis/hemorrhage | |
| Grading | Management |
| G1: Asymptomatic or mild symptoms | Consider holding ICPi until patient is stabilized on replacement hormone |
| | Endocrine consultation |
| | Replacement therapy with prednisone (5-10 mg daily) or hydrocortisone (10-20 mg orally every morning, 5-10 mg orally in early afternoon) |
| | May require fludrocortisone (0.1 mg/d) for mineralocorticoid replacement in primary adrenal insufficiency |
| | Titrate dose up or down as symptoms dictate |
| G2: Moderate symptoms, able to perform ADL | Consider holding ICPi until patient is stabilized on replacement hormone |
| | Endocrine consultation |
| | Initiate outpatient treatment at two to three times maintenance |
| | (if prednisone, 20 mg daily; if hydrocortisone, 20-30 mg in the morning, and 10-20 mg in the afternoon) to manage acute symptoms. |
| | Taper stress-dose corticosteroids down to maintenance doses over 5-10 days |
| | Maintenance therapy as in G1. |
| G3-4: Severe symptoms, medically significant or life-<br>threatening consequences, unable to perform ADL | Hold ICPi until patient is stabilized on replacement hormone |
| | Endocrine consultation |
| | See in clinic or, for after hours, make an emergency department referral for normal saline (at least 2 L) and IV stress-dose corticosteroids on presentation hydrocortisone 100 mg or dexamethasone 4 mg (if the diagnosis is not clear and stimulation testing will be needed) |
| | Taper stress-dose corticosteroids down to maintenance doses over 7-14 days after discharge |
| Additional considerations | Maintenance therapy as in G1 |

### Additional considerations

Primary and secondary adrenal insufficiency can be distinguished by the relationship between ACTH and cortisol. If the ACTH is low with low cortisol, then management is as per 4.3.


### 4.0 Endocrine Toxicity

Patients on corticosteroids for management of other conditions will have low morning cortisol as a result of iatrogenic, secondary adrenal insufficiency. ACTH will also be low in these patients. A diagnosis of adrenal insufficiency is challenging to make in these situations (see next section on hypophysitis).

Emergent therapy for someone with suspected adrenal insufficiency is best done with dexamethasone as a stimulation test can still be performed. If the diagnosis is already confirmed, can use hydrocortisone 100 mg.

All patients need education on stress dosing and a medical alert bracelet for adrenal insufficiency to trigger stress-dose corticosteroids by EMS.

Endocrine consultation prior to surgery or any procedure for stress-dose planning.

### 4.3 Pituitary - hypophysitis

Definition: Inflammation of the pituitary with varying effects on hormone function. Most commonly presenting with central adrenal insufficiency. May also have central hypothyroidism, diabetes insipidus, and hypogonadism. Diagnostic work-up

Diagnosis: Low ACTH with a low cortisol. Low or normal TSH with a low FT4. Hypernatremia and volume depletion with diabetes insipidus. Low testosterone or estradiol with low LH and FSH.

### Testing

Evaluate ACTH, cortisol (AM), TSH, FT4, electrolytes

Consider evaluating LH, FSH, and testosterone levels in males or estrogen in premenopausal females with fatigue, loss of libido, and mood changes Consider MRI of the brain with or without contrast with pituitary/sellar cuts in patients with multiple endocrine abnormalities ± new severe headaches or complaints of vision changes

| Grading | Management |
|---|---|
| G1: Asymptomatic or mild symptoms | Consider holding ICPi until patient is stabilized on replacement hormones Endocrine consultation Hormonal supplementation as in G1 |
| G3-4: Severe symptoms, medically significant or life-<br>threatening consequences, unable to perform ADL | Hold ICPi until patient is stabilized on replacement hormones Endocrine consultation Hormonal supplementation as in G1 Consider initial pulse dose therapy with prednisone 1-2 mg/kg oral daily (or equivalent) tapered over at least 1-2 weeks |

### Additional considerations

Be aware of the need to start corticosteroids first when planning hormone replacement therapy for multiple deficiencies

All patients need instruction on doubling doses for illness (stress dosing) and a medical alert bracelet for adrenal insufficiency to trigger stress-dose corticosteroids by EMS

Corticosteroid use can cause isolated central adrenal insufficiency

Work-up cannot be done with a simple AM cortisol in a patient on corticosteroids for other conditions Laboratory confirmation of adrenal insufficiency should not be attempted until treatment with corticosteroids for other disease is ready to be discontinued. For long-term exposure, consult endocrinology for recovery and weaning protocol using hydrocortisone.

### 4.4 Diabetes

Definition: T2DM is a combination of insulin resistance and insufficiency that may require oral or insulin therapy. It may be new onset or exacerbated during therapy for nonimmunologic reasons, such as corticosteroid exposure. Autoimmune T1DM results from islet cell destruction and is often acute onset, with ketosis and an insulin requirement

Diagnostic work-up

Monitor patients for hyperglycemia or other signs and symptoms of new or worsening DM, including measuring glucose at baseline and with each treatment cycle during induction for 12 weeks, then every 3-6 weeks thereafter. To guide the work-up in new-onset hyperglycemia, clinicians should consider a patient's medical background, exposure history, and risk factors for each subtype of DM.



| 4.0 Endocrine Toxicity |
|------------------------|
|------------------------|

Laboratory evaluation in suspected T1DM should include testing for ketosis in urine and an assessment of the anion gap on a metabolic panel. Anti-glutamic acid decarboxylase, anti-islet cell, or anti-insulin antibodies are highly specific for autoimmune diabetes. Insulin and C-peptide levels can also assist in the diagnosis.

| riigiliy specific for autofilifiurie diabetes. Irisuilif and C-peptide levels can also assist in the diagnosis. | |
|---|---|
| Grading | Management |
| G1: Asymptomatic or mild symptoms; fasting glucose value > ULN (160 mg/dL); fasting glucose value > ULN (8.9 mmol/L); no evidence of ketosis or laboratory evidence of T1DM | Can continue ICPi with close clinical follow-up and laboratory evaluation May initiate oral therapy for those with new-onset T2DM Screen for T1DM if appropriate, for example, acute onset with prior normal values or clinical concern for ketosis |
| G2: Moderate symptoms, able to perform ADL, fasting glucose value > 160-250 mg/dL; fasting glucose value > 8.9-13.9 mmol/L, ketosis or evidence of T1DM at any glucose level | May hold ICPi until glucose control is obtained Titrate oral therapy or add insulin for worsening control in T2DM Should administer insulin for T1DM (or as default therapy if there is confusion about type) Urgent endocrine consultation for any patient with T1DM; in the absence of endocrinology, internal medicine may suffice Consider admission for T1DM if early outpatient evaluation is not available or signs of ketoacidosis are present |
| G3-4: Severe symptoms, medically significant or life-threatening consequences, unable to perform ADL G3: > 250-500 mg/dL (> 13.9-27.8 mmol/L) G4: > 500 mg/dL (> 27.8 mmol/L) | Hold ICPi until glucose control is obtained on therapy with reduction of toxicity to G1 or less Urgent endocrine consultation for all patients Initiate insulin therapy for all patients Admit for inpatient management: Concerns for developing DKA, Symptomatic patients regardless of diabetes type, New-onset T1DM unable to see endocrinology |

### Additional considerations

Insulin therapy can be used as the default in any case with hyperglycemia

Long-acting therapy alone is not usually sufficient for T1DM, where half of daily requirements are usually given in divided doses as prandial coverage and half as long acting.

Insulin doses will be lower in T1DM because of preserved sensitivity (total daily requirement can be estimated at 0.3-0.4 units/kg/d).

In T2DM, sliding-scale coverage with meals over a few days provides data to estimate a patient's daily requirements and can be used to more rapidly titrate basal needs.

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate.

Abbreviations: ACTH, adrenocorticotropic hormone: ADL, activities of daily living: CT, computed tomography: DKA, diabetic ketoacidosis; DM, diabetes mellitus; EMS, emergency medical services; FSH, follicle-stimulating hormone; FT4, free thyroxine; G, Grade; ICPi, immune checkpoint inhibitor; irAE, immune-related adverse event; IV.intravenous; LH, luteinizing hormone; MRI, magnetic resonance imaging; PTU, propylthiouracil; SSKI, potassium iodide; T1DM, type 1 diabetes mellitus; T2DM, type 2 diabetes mellitus; TRAb, thyroid-stimulating hormone receptor antibody; TSH, thyroid-stimulating hormone; TSI, thyroid-stimulating immunoglobulin; ULN, upper limit of normal.

### Table A5 Management of Musculoskeletal irAEs in Patients Treated With ICPis

#### 5.0 Musculoskeletal Toxicities

### 5.1 Inflammatory arthritis

Definition: A disorder characterized by inflammation of the joints

Clinical symptoms: Joint pain accompanied by joint swelling; inflammatory symptoms, such as stiffness after inactivity or in the morning, lasting > 30 minutes to 1 hour; improvement of symptoms with NSAIDs or corticosteroids but not with opioids or other pain medications may also be suggestive of inflammatory arthritis.

Diagnostic work-up

G1

Complete rheumatologic history and examination of all peripheral joints for tenderness, swelling, and range of motion; examination of the spine Consider plain x-ray/imaging to exclude metastases and evaluate joint damage (erosions), if appropriate

Consider autoimmune blood panel including ANA, RF, and anti-CCP, and anti-inflammatory markers (ESR and CRP) if symptoms persist; if symptoms are suggestive of reactive arthritis or affect the spine, consider HLA B27 testing

G2

Complete history and examination as above; laboratory tests as above

Consider US ± MRI of affected joints if clinically indicated (e.g, persistent arthritis unresponsive to treatment, suspicion for differential diagnoses such as metastatic lesions or septic arthritis)

Consider early referral to a rheumatologist, if there is joint swelling (synovitis) or if symptoms of arthralgia persist > 4 weeks

G3-4

As for G2

Seek rheumatologist advice and review

Monitoring: Patients with inflammatory arthritis should be monitored with serial rheumatologic examinations, including inflammatory markers, every 4-6 weeks after treatment is instituted.

| Grading | Management |
|---|---|
| All Grades | Clinicians should follow reports of new joint pain to determine whether inflammatory arthritis is present; question whether symptom new since receiving ICPi |
| G1: Mild pain with inflammation, erythema, or joint swelling | Continue ICPi<br>Initiate analgesia with acetaminophen and/or NSAIDs |
| G2: Moderate pain associated with signs of inflammation, erythema, or joint swelling, limiting instrumental ADL | Hold ICPi and resume upon symptom control and on prednisone ≤ 10 mg/d Escalate analgesia and consider higher doses of |
| | NSAIDS as needed If inadequately controlled, initiate prednisone or |
| | prednisolone 10-20 mg/d or equivalent for 4-6 weeks If improvement, slow taper according to response during the next 4-6 weeks; if no improvement after initial 4-6 weeks, treat as G3 |
| | If unable to lower corticosteroid dose to < 10 mg/d after 3 months, consider DMARD |
| | Consider intra-articular corticosteroid injections for large joints |
| | Referral to rheumatology |
| G3-4: Severe pain associated with signs of inflammation, erythema, or joint swelling; irreversible joint damage; disabling; limiting self-care ADL | For G3: Hold ICPi temporarily and may resume in consultation with rheumatology, if recover to G1 or less For G4: permanently discontinue ICPi Initiate oral prednisone 0.5-1 mg/kg |

| 5.0 Musculoskeletal Toxicities | |
|---|---|
| | If failure of improvement after 4 weeks or worsening in meantime, consider synthetic or biologic DMARD Synthetic: methotrexate, leflunomide |
| | Biologic: consider anticytokine therapy such as TNF-a or IL-6 receptor inhibitors. (Note: As caution, IL-6 inhibition can cause intestinal perforation; while this is extremely rare, it should not be used in patients with colitis.) Test for viral hepatitis B, C, and latent/active TB test prior to DMARD treatment Referral to rheumatology. |

### Additional considerations

Early recognition is critical to avoid erosive joint damage.

Corticosteroids can be used as part of initial therapy in inflammatory arthritis, but due to likely prolonged treatment requirements, physicians should consider starting corticosteroid-sparing agents earlier than one would with other irAEs

Oligoarthritis can be treated early on with intra-articular corticosteroids; consider early referral.

Consider PCP prophylaxis for patients treated with high dose of corticosteroids for 12 weeks, as per local guidelines.

### 5.2 Myositis

Definition: A disorder characterized by muscle inflammation with weakness and elevated muscle enzymes (CK). Muscle pain can be present in severe cases. Can be life-threatening if respiratory muscles or myocardium are involved

Diagnostic work-up

Complete rheumatologic and neurologic history regarding differential diagnosis; rheumatologic and neurologic examination, including muscle strength; and examination of the skin for findings suggestive of dermatomyositis. Muscle weakness is more typical of myositis than pain. Consider preexisting conditions that can cause similar symptoms.

Blood testing to evaluate muscle inflammation

CK, transaminases (AST, ALT), LDH, and aldolase can also be elevated

Troponin to evaluate myocardial involvement and other cardiac testing, such as echocardiogram, as needed Inflammatory markers (ESR and CRP)

Consider EMG, imaging (MRI), and/or biopsy on an individual basis when diagnosis is uncertain and overlap with neurologic syndromes, such as myasthenia gravis, is suspected

Consider paraneoplastic autoantibody testing for myositis and neurologic conditions, such as myasthenia gravis Monitoring: CK, ESR, CRP

G1: Complete examination and laboratory work-up as above

G2: Complete history and examination as above; autoimmune myositis blood panel; EMG, MRI of affected joints Early referral to a rheumatologist or neurologist

G3-4: As for G2

Urgent referral to a rheumatologist or neurologist

| Grading | Management |
|---|---|
| G1: Mild weakness with or without pain | Continue ICPi |
| | If CK is elevated and patient has muscle weakness, may offer oral corticosteroids, and treat as G2 |
| | Offer analgesia with acetaminophen or NSAIDs if there are no contraindications |
| G2: Moderate weakness with or without pain, limiting age-appropriate instrumental ADL | Hold ICPi temporarily and may resume upon symptom control, if CK is normal and prednisone dose 10 mg; if worsens, treat as per G3 NSAIDs as needed |
| | Referral to rheumatologist or neurologist |

| 5.0 Musculoskeletal Toxicities | |
|---|---|
| | If CK is elevated three times or more), initiate prednisone or equivalent at 0.5-1 mg/kg May require permanent discontinuation of ICPi in most patients with G2 symptoms and objective findings (elevated enzymes, abnormal EMG, abnormal muscle MRI or biopsy) |
| G3-4: Severe weakness with or without pain, limiting self-care ADL | For G3: Hold ICPi until G1 or less and permanently discontinue if any evidence of myocardial involvement For G4: permanently discontinue ICPi Consider hospitalization for severe weakness Referral to rheumatologist or neurologist Initiate prednisone 1 mg/kg or equivalent. Consider 1-2 mg/kg of methylprednisolone IV or higher-dose bolus if severe compromise (weakness severely limiting mobility, cardiac, respiratory, dysphagia) Consider plasmapheresis Consider IVIG therapy Consider other immunosuppressant therapy, such as methotrexate, azathioprine, or mycophenolate mofetil, if symptoms and CK levels do not improve or worsen after 4-6 weeks; rituximab is used in primary myositis but caution is advised given its long biologic duration In case of management with rituximab, ICPi treatment should be discontinued |
| A 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |

Additional considerations: Caution is advised with rechallenging

### 5.3 Polymyalgia-like syndrome

Definition: Characterized by marked pain and stiffness in proximal upper and/or lower extremities and no signs of true muscle inflammation such as CK elevation or EMG findings of myositis. No true muscle weakness, difficulty in active motion related to pain

Diagnostic work-up

G1

Complete rheumatologic history regarding differential diagnosis and examination of all joints and skin Check for symptoms of temporal arteritis, such as headache or visual disturbances; refer to ophthalmologist if present, and consider temporal artery biopsy ANA, RF, anti-CCP

CK to evaluate differential diagnosis of myositis

Inflammatory markers (ESR, CRP)

Monitoring: ESR, CRP

G2: Complete history and examination as above; autoimmune tests as required for differential diagnosis; early referral to a rheumatologist

G3-4: As for G2; see rheumatologist advice and review

| Grading | Management |
|---|---|
| G1: Mild stiffness and pain | Continue ICPi Initiate analgesia with acetaminophen and/or NSAIDs if there are no contraindications |
| G2: Moderate stiffness and pain, limiting age-<br>appropriate instrumental ADL | Consider holding ICPi and resuming upon symptom control, prednisolone < 10 mg; if worsens, treat as per G3 |
| | Initiate prednisone 20 mg/d or equivalent; if symptoms improve, start to taper dose after 3-4 weeks |
| | If no improvement or need for higher dosages after 4 weeks, escalate to G3 Consider referral to rheumatology |

### 5.0 Musculoskeletal Toxicities

G3-4: Severe stiffness and pain, limiting self-care ADL

For G3: Hold ICPi and may resume, in consultation with rheumatology, if recover to G1 or less; however, note that cases of toxicity returning upon rechallenge have been reported. ICPi should be permanently discontinued in such cases

For G4: permanently discontinue ICPi

Referral to rheumatology

Should initiate prednisone 20 mg/d or equivalent. If no improvement or need for higher dosages for prolonged time, may offer a corticosteroid-sparing agent such as methotrexate or IL-6 inhibition with tocilizumab

(Note: As caution, IL-6 inhibition can cause intestinal perforation; while this is extremely rare, it should not be used in patients with colitis or GI metastases). Consider admission for pain control

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate.

Abbreviations: ADL, activities of daily living; ALT, alanine aminotransferase; ANA, antinuclear antibodies; AST, aspartate aminotransferase; CCP, citrullinated protein antibody; CK, creatine kinase; CRP, C-reactive protein; DMARD, disease-modifying antirheumatic drug; EMG, electromyography; ESR, erythrocyte sedimentation rate; G, Grade; GI, gastrointestinal; HLA, human leukocyte antigen; ICPi, immune checkpoint inhibitor; IL, interleukin; irAE, immune-related adverse event; IV, intravenous; IVIG, intravenous immunoglobulin; LDH, lactate dehydrogenase; MRI, magnetic resonance imaging, NSAID, nonsteroidal anti-inflammatory drug; PCP, Pneumocystis pneumonia; RF, rheumatoid factor; TB, tuberculosis; TNF, tumor necrosis factor; US, ultrasound.

# Table A6 Management of Renal irAEs in Patients Treated With ICPis

| 6.0 Renal Toxicities | |
|---|---|
| Nephritis and renal dysfunction: diagnosis and monitoring | ] |
| For any suspected immune-mediated adverse reactions, | exclude other causes |
| Monitor patients for elevated serum creatinine prior to eve | ery dose |
| Routine urinalysis is not necessary, other than to rule out | |
| If no potential alternative cause of AKI identified, then one should forego biopsy and proceed directly with immunosuppressive therapy Swift treatment of autoimmune component important | |
| 6.1 Nephritis | |
| Definition: Inflammation of the kidney affecting the structu | ıre |
| Grading | Management |
| G1: Creatinine level increase > ULN - 1.5 x ULN | Consider temporarily holding ICPi, pending consideration of potential alternative etiologies (recent IV contrast, medications, fluid status) and baseline renal function. A change that is still < 1.5 ULN could be meaningful |
| G2: Creatinine | Hold ICPi |
| > 1.5 - 3.0 x baseline; > 1.5 - 3.0 x ULN | Consult nephrology |
| | Evaluate for other causes (recent IV contrast, medications, fluid status, etc); if other etiologies ruled out, administer 0.5-1 mg/kg/d prednisone equivalents If worsening or no improvement: 1 to 2 mg/kg/d prednisone equivalents and permanently discontinue treatment |
| | If improved to G1 or less, taper corticosteroids over 4-6 weeks If no recurrence of chronic renal insufficiency, discuss resumption of ICPi with patient after taking into account the risks and benefits. |
| G3: Creatinine<br>> 3.0 x baseline; > 3.0 - 6.0 x ULN | Permanently discontinue ICPi |
| G4: Life-threatening consequences; dialysis indicated; > 6.0 x ULN | Permanently discontinue ICPi Consult nephrology Evaluate for other causes (recent IV contrast, medications, fluid status, etc) Administer corticosteroids (initial dose of 1-2 mg/kg/d prednisone or equivalent) |
| Additional considerations Monitor creatinine weekly Reflex kidney biopsy should be discouraged until corticosteroid treatment has been attempted | |
| 6.2 Symptomatic nephritis: follow-up | |
| Grading | Management |
| G1 | Improved to baseline, resume routine creatinine monitoring |
| G2 | If improved to G1, taper corticosteroids over at least 3 weeks before resuming treatment with routine creatinine monitoring If elevations persist > 7 days or worsen and no other cause found, treat as G3 |
| G3 | If improved to G1, taper corticosteroids over at least 4 weeks |

# Bintrafusp alfa in HMGA2-expressing Triple Negative Breast Cancer

| 6.0 Renal Toxicities | |
|---|---|
| | If elevations persist 3-5 days or worsen, consider additional immunosuppression (e.g, mycophenolate) |
| G4 | If improved to G1, taper corticosteroids over at least 4 weeks If elevations persist 2-3 days or worsen, consider additional immunosuppression (e.g, mycophenolate) |
| All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate. | |

Abbreviations: AKI, acute kidney injury; G, Grade; ICPi, immune checkpoint inhibitor; irAE, immune-related adverse event; IV, intravenous; ULN, upper limit of normal; UTI, urinary tract infection.

### Table A7 Management of Nervous System ir AEs in Patients Treated With ICPis

### 7.0 Nervous System Toxicities

### 7.1 Myasthenia gravis

Definition: Fatigable or fluctuating muscle weakness, generally more proximal than distal. Frequently has ocular and/or bulbar involvement (ptosis, extraocular movement abnormalities resulting in double vision, dysphagia, dysarthria, facial muscle weakness). May have neck and/or respiratory muscle weakness. (Note: May occur with myositis and/or myocarditis). Respiratory symptoms may require evaluation to rule out pneumonitis, myocarditis. Miller Fisher variant of Guillain-Barré syndrome (ophthalmoparesis) and the oculobulbar myositis (ptosis, ophthalmoparesis, dysphagia, neck and respiratory weakness) with ICPi may have overlapping symptoms.

### Diagnostic work-up

AChR and antistriated muscle antibodies in blood; if AChR antibodies are negative, consider muscle specific kinase and lipoprotein-related 4 antibodies in blood Pulmonary function assessment with NIF and VC CPK, aldolase, ESR, CRP for possible concurrent myositis

Consider MRI of brain and/or spine, depending on symptoms to rule out CNS involvement by disease or alternate diagnosis

If respiratory insufficiency or elevated CPK, troponin T, perform cardiac examination with ECG and TTE for possible concomitant myocarditis

Neurologic consultation

Electrodiagnositic studies, including neuromuscular junction testing with repetitive stimulation and/or jitter studies, NCS to exclude neuropathy, and needle EMG to evaluate for myositis

| Grading | Management |
|---|---|
| All grades | All grades warrant work-up and intervention given potential for progressive myasthenia gravis to lead to respiratory compromise |
| No G1 | |
| G2: Some symptoms interfering with ADL MGFA severity class 1 (ocular symptoms and findings only) and MGFA severity class 2 (mild generalized weakness) | Hold ICPi and may resume in G2 patients (MGFA 1 and 2) only if symptoms resolve Should consult neurology Pyridostigmine starting at 30 mg orally three times a day and gradually increase to maximum of 120 mg orally four times a day as tolerated and based on symptoms Administer corticosteroids (prednisone, 1-1.5 mg/kg orally daily) if symptoms G2; wean based on symptom improvement |
| G3-4: Limiting self-care and aids warranted, weakness limiting walking, ANY dysphagia, facial weakness, respiratory muscle weakness, or rapidly progressive symptoms, or MGFA severity class 3-4 moderate to severe generalized weakness to myasthenic crisis | Permanently discontinue ICPi Admit patient, may need ICU-level monitoring Neurology consult Continue corticosteroids and initiate IVIG 2 g/kg IV over 5 days (0.4 g/kg/d) or plasmapheresis for 5 days Frequent pulmonary function assessment Daily neurologic review |

### Additional considerations

Avoid medications that can worsen myasthenia: β-blockers, IV magnesium, fluoroquinolones, aminoglycosides, and macrolides Initially a 5-day course of plasmapheresis or a 2 g/kg course of IVIG over 5 days

1-2 mg/kg methylprednisolone daily, wean based on symptom improvement

Pyridostigmine, wean based on improvement

ICPi-associated myasthenia gravis may be monophasic, and additional corticosteroid-sparing agents may not be required



### 7.0 Nervous System Toxicities

### 7.2 Guillain-Barré syndrome

Definition: Progressive, most often symmetrical muscle weakness with absent or reduced deep tendon reflexes. Often starts with sensory symptoms/neuropathic pain localized to lower back and thighs. May involve extremities (typically ascending weakness but not always), facial, respiratory, and bulbar and oculomotor nerves. May have dysregulation of autonomic nerves.

Diagnostic work-up

Neurologic consultation

MRI of spine with or without contrast (rule out compressive lesion and evaluate for nerve root enhancement/thickening)

Lumbar puncture: CSF typically has elevated protein and often elevated WBCs; even though this is not typically seen in classic Guillain-Barré syndrome, cytology should be sent with any CSF sample from a patient with cancer.

Serum antibody tests for Guillain-Barré syndrome variants (GQ1b for Miller Fisher variant a/w ataxia and ophthalmoplegia) Electrodiagnostic studies to evaluate polyneuropathy

Pulmonary function testing (NIF/VC)

Frequent neurochecks

| Grading | Management |
|---|---|
| All grades | Warrant work-up and intervention given potential for progressive Guillain-Barré syndrome to lead to respiratory compromise Note: There is no G1 toxicity |
| G1: Mild, none | NA |
| G2: Moderate, some interference with ADL, symptoms concerning to patient | Discontinue ICPi |
| G3-4: Severe, limiting self-care and aids warranted, weakness, limiting walking, ANY dysphagia, facial weakness, respiratory muscle weakness, or rapidly progressive symptoms | Permanently discontinue ICPi. Admission to inpatient unit with capability of rapid transfer to ICU-level monitoring Start IVIG (0.4 g/kg/d for 5 days for a total dose of 2 g/kg) or plasmapheresis. Corticosteroids are usually not recommended for idiopathic Guillain-Barré syndrome; however, in ICPi-related forms, a trial is reasonable (methylprednisolone 2-4 mg/kg/d), followed by slow corticosteroid taper Pulse corticosteroid dosing (methylprednisolone 1 g/d for 5 days) may also be considered for G3-4 along with IVIG or plasmapheresis Frequent neurochecks and pulmonary function monitoring Monitor for concurrent autonomic dysfunction Nonopioid management of neuropathic pain Treatment of constipation/ileus |

### Additional considerations

Slow prednisone taper after corticosteroid pulse plus IVIG or plasmapheresis May require repeat IVIG courses Caution with rechallenging for severe cases

### 7.3 Peripheral neuropathy

Definition: Can present as asymmetric or symmetric sensory, motor, or sensory motor deficit. Focal mononeuropathies, including cranial neuropathies (e.g, facial neuropathies/Bell palsy) may be present. Numbness and paresthesias may be painful or painless. Hypo- or areflexia or sensory ataxia may be present.

Diagnostic work-up

G1

Screen for reversible neuropathy causes: diabetic screen, B12, folate, TSH, HIV, consider serum protein electrophoresis, and other vasculitic and autoimmune screen Neurologic consultation

### 7.0 Nervous System Toxicities

Consider MRI of spine with or without contrast

G2: in addition to above

MRI spine advised/MRI of brain if cranial nerve Consider EMG/NCS

Consider neurology consultation

G3-4: go to Guillain-Barré syndrome algorithm

| Grading | Management |
|---|---|
| G1: Mild, no interference with function and symptoms not concerning to patient. Note: Any cranial nerve problem should be managed as moderate | Low threshold to hold ICPi and monitor symptoms for a week If to continue, monitor very closely for any symptom progression |
| G2: Moderate, some interference with ADL, symptoms concerning to patient (i.e, pain but no weakness or gait limitation) | Hold ICPi and resume once return to G1 Initial observation OR initiate prednisone 0.5-1 mg/kg (if progressing from mild) Neurontin, pregabalin, or duloxetine for pain |
| G3-4: Severe, limiting self-care and aids warranted, weakness limiting walking or respiratory problems (i.e, leg weakness, foot drop, rapidly ascending sensory changes) Severe may be Guillain-Barré syndrome and should be managed as such | Permanently discontinue ICPi Admit patient Neurologic consultation Initiate IV methylprednisolone 2-4 mg/kg and proceed as per Guillain-Barré syndrome management |

### 7.4 Autonomic neuropathy

Definition: Nerves that control involuntary bodily functions are damaged. This may affect blood pressure, temperature control, digestion, bladder function, and sexual function. A case of severe enteric neuropathy with ICPi has been reported. Can present with GI difficulties such as new severe constipation, nausea, urinary problems, sexual difficulties, sweating abnormalities, sluggish pupil reaction, and orthostatic hypertension.

### Diagnostic work-up

An evaluation by neurologist or relevant specialist, depending on organ system, with testing that may include Screening for other causes of autonomic dysfunction: diabetic screen, adrenal insufficiency, HIV, paraproteinemia, amyloidosis, botulism; consider chronic diseases such as Parkinson and other autoimmune screening AM orthostatic vitals

Consider electrodiagnostic studies to evaluate for concurrent polyneuropathy

Consider paraneoplastic Lambert-Eaton myasthenic syndrome, antineutrophil cytoplasmic antibodies, and ganglionic AChR antibody testing

| Grading | Management |
|---|---|
| G1: Mild, no interference with function and symptoms not concerning to patient | Low threshold to hold ICPi and monitor symptoms for a week; if to continue, monitor very closely for any symptom progression |
| G2: Moderate, some interference with ADL, symptoms concerning to patient | Hold ICPi and resume once return to G1 Initial observation OR initiate prednisone 0.5-1 mg/kg (if progressing from mild) Neurologic consultation |
| G3-4: Severe, limiting self-care and aids warranted | Permanently discontinue ICPi Admit patient Initiate methylprednisolone 1 g daily for 3 days followed by oral corticosteroid taper Neurologic consultation |

### 7.5 Aseptic meningitis

Definition: may present with headache, photophobia, and neck stiffness; often afebrile but may be febrile. There may be nausea/vomiting. Mental status should be normal (distinguishes from encephalitis).

Diagnostic work-up

MRI of brain with or without contrast + pituitary protocol

AM cortisol, ACTH to rule out adrenal insufficiency



### 7.0 Nervous System Toxicities

Consider lumbar puncture: measure opening pressure; check cell count and protein glucose; and perform Gram stain, culture, PCR for HSV, and other viral PCRs depending on suspicion, cytology

May see elevated WBC count with normal glucose, normal culture, and Gram stain; may see reactive lymphocytes or histiocytes on cytology

### Grading Management

- G1: Mild, no interference with function and symptoms not concerning to patient. Note: Any cranial nerve problem should be managed as moderate.
- G2: Moderate, some interference with ADL, symptoms concerning to patient (i.e, pain but no weakness or gait limitation)
- G3-4: Severe, limiting self-care and aids warranted

Hold ICPi and discuss resumption with patient only after taking into account the risks and benefits, consider empirical antiviral (IV acyclovir) and antibacterial therapy until CSF results Once bacterial and viral infection are negative, may closely monitor off corticosteroids or consider oral prednisone 0.5-1 mg/kg or IV methylprednisolone 1 mg/kg if moderate/severe symptoms

### 7.6 Encephalitis

Definition: As for aseptic meningitis, need to exclude infectious causes, especially viral (i.e, HSV). Confusion, altered behavior, headaches, seizures, short-term memory loss, depressed level of consciousness, focal weakness, speech abnormality

Diagnostic work-up

Neurologic consultation

MRI of brain with or without contrast may reveal T2/fluid-attenuated inversion recovery changes typical of what is seen in autoimmune encephalopathies or limbic encephalitis or may be normal

Lumbar puncture: check cell count and protein glucose and perform Gram stain, culture, PCR for HSV and other viral PCRs depending on suspicion, cytology, oligoclonal bands, autoimmune encephalopathy, and paraneoplastic panels.

May see elevated WBC count with lymphocytic predominance and/or elevated protein

EEG to evaluate for subclinical seizures

Blood: metabolic, CBC, ESR, CRP, ANCA (if suspect vasculitic process), thyroid panel including TPO and thyroglobulin Rule out concurrent anemia/thrombocytopenia, which can present with severe headaches and confusion

| Grading | Management |
|---|---|
| G1: Mild, no interference with function and symptoms not concerning to patient. Note: Any cranial nerve problem should be managed as moderate. G2: Moderate, some interference with ADL, symptoms concerning to patient (i.e, pain but no weakness or gait limitation) G3-4: Severe, limiting self-care and aids warranted | Hold ICPi and discuss resumption with patient only after taking into account the risks and benefits As above for aseptic meningitis suggest concurrent IV acyclovir until PCR results obtained and negative Trial of methylprednisolone 1-2 mg/kg If severe or progressing symptoms or oligoclonal bands present, consider pulse corticosteroids methylprednisolone 1 g IV daily for 3-5 days plus IVIG 2 g/kg over 5 days If positive for autoimmune encephalopathy antibody and limited or no improvement, consider rituximab or plasmapheresis in consultation with neurology. |

### 7.7 Transverse myelitis

Definition: Acute or subacute weakness or sensory changes bilateral, often with increased deep tendon reflexes

Diagnostic work-up

Neurologic consultation

MRI of spine (with thin axial cuts through the region of suspected abnormality) and MRI of brain

Lumbar puncture: cell count, protein, glucose, oligoclonal bands, viral PCRs, cytology, onconeural antibodies Blood: B12, HIV, RPR, ANA, Ro/La, TSH, aquaporin-4 IgG

Evaluation for urinary retention, constipation



# Bintrafusp alfa in HMGA2-expressing Triple Negative Breast Cancer

| 7.0 Nervous System Toxicities | |
|---|---|
| Grading | Management |
| G1: Mild, no interference with function and symptoms not concerning to patient. Note: Any cranial nerve problem should be managed as moderate. G2: Moderate, some interference with ADL, symptoms concerning to patient (i.e, pain but no weakness or gait limitation) G3-4: Severe, limiting self-care and aids warranted | Permanently discontinue ICPi Methylprednisolone 2 mg/kg Strongly consider higher doses of 1 g/d for 3-5 days Strongly consider IVIG |
| All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate. | |

Abbreviations: AChR, acetylcholine receptor; ACTH, adrenocorticotropic hormone; ADL, activities of daily living; ANA, antinuclear antibody; ANCA, antineutrophil cytoplasmic antibodies; CBC, complete blood count; CNS, central nervous system; CPK, creatine phosphokinase; CRP, C-reactive protein; CSF, cerebrospinal fluid; ECG, electrocardiogram; EEG, electroencephalogram; EMG, electromyography; ESR, erythrocyte sedimentation rate; G, Grade; GI, gastrointestinal; HIV, human immunodeficiency virus; HSV, herpes simplex virus; ICPi, immune checkpoint inhibitor; ICU, intensive care unit; IgG, immunoglobulin G; irAE, immune-related adverse event; IV, intravenous; IVIG, intravenous immunoglobulin; MGFA, Myasthenia Gravis Foundation of America; MRI, magnetic resonance imaging; NA, not applicable; NCS, nerve conduction study; NIF, negative inspiratory force; PCR, polymerase chain reaction; RPR, rapid plasma reagin, TPO, thyroid peroxidase; TSH, thyroid-stimulating hormone; TTE, transthoracic echocardiogram; VC, vital capacity; WBC, white blood cell.

### Table A8 Management of Hematologic irAEs in Patients Treated With ICPis

### 8.0 Hematologic Toxicities

### 8.1 Autoimmune hemolytic anemia

Definition: A condition in which RBCs are destroyed and removed from the blood stream before their normal lifespan is over. Symptoms include weakness, paleness, jaundice, dark-colored urine, fever, inability to do physical activity, and heart murmur.

### Diagnostic work-up

History and physical examination (with special consideration of history of new drugs and insect, spider, or snake bites)

Blood chemistry, CBC with evidence of anemia, macrocytosis, evidence of hemolysis on peripheral smear; LDH, haptoglobin, bilirubin, reticulocyte count, free Hgb DIC panel, which could include PTNIR infectious causes Autoimmune serology

Paroxysmal nocturnal hemoglobinuria screening

Direct and indirect bilirubin; LDH; direct agglutinin test; and if no obvious cause, bone marrow analysis, cytogenetic analysis to evaluate for myelodysplastic syndromes

Evaluation for viral/bacterial (mycoplasma, etc) causes of hemolysis studies

Protein electrophoresis, cryoglobulin analysis

Work-up for bone marrow failure syndrome if refractory, including B12, folate, copper, parvovirus, FE, thyroid, infection

Glucose-6-phosphate dehydrogenase

Evaluation of common drug causes (ribavirin, rifampin, dapsone, interferon, cephalosporins, penicillins, NSAIDs, quinine/quinidine, fludarabine, ciprofloxacin, lorazepam, diclofenac, etc)

Assessment of methemoglobinemia

| Grading | Management |
|---|---|
| G1: Hgb < LLN to 10.0 g/dL; < LLN to 6.2 mmol/L; < LLN to 100 g/L | Continue ICPi with close clinical follow-up and laboratory evaluation |
| G2: Hgb < 10.0 to 8.0 g/dL; < 6.2 to 4.9mmol/L; < 100 to 80 g/L | Hold ICPi and strongly consider permanent discontinuation |
| | Administer 0.5-1 mg/kg/d prednisone equivalents |
| G3: Hgb < 8.0 g/dL; < 4.9 mmol/L; < 80 g/L; transfusion | Permanently discontinue ICPi |
| indicated | Should use clinical judgment and consider admitting the patient |
| | Hematology consult |
| | Prednisone 1-2 mg/kg/d (oral or IV depending on symptoms/speed of development) |
| | If worsening or no improvement, 1-2 mg/kg/d prednisone equivalents and permanently discontinue ICPi treatment |
| | Consider RBC transfusion per existing guidelines; do not transfuse more than the minimum number of RBC units necessary to relieve symptoms of anemia or to return a patient to a safe Hgb range (7-8 g/dL in stable, noncardiac inpatients) |
| | Should offer patients supplementation with folic acid 1 mg once daily |
| G4: Life-threatening consequences, urgent intervention | Permanently discontinue ICPi |
| indicated | Admit patient |
| | Hematology consult |
| | IV prednisone corticosteroids 1-2 mg/kg/d |

# 8.0 Hematologic Toxicities If no improvement or if worsening while on corticosteroids or severe symptoms on presentation, initiate other immunosuppressive drugs, such as rituximab, IVIG, cyclosporin A, and mycophenolate mofetil RBC transfusion per existing guidelines; discuss with blood bank team prior to transfusions that a patient with possible ICPi serious AE is in house.

Additional considerations: Monitor Hgb levels on a weekly basis until the corticosteroid tapering process is complete; thereafter, less-frequent testing is needed

### 8.2 Acquired TTP

Definition: A disorder characterized by the presence of microangiopathic hemolytic anemia, thrombocytopenic purpura, fever, renal abnormalities, and neurologic abnormalities, such as seizures, hemiplegia, and visual disturbances. It is an acute or subacute condition.

Diagnostic work-up

History with specific questions related to drug exposure (e.g, chemotherapy, sirolimus, tacrolimus, opana ER antibiotics, quinine) Physical examination, peripheral smear

ADAMTS13 activity level and inhibitor titer

LDH, haptoglobin, reticulocyte count, bilirubin, urinalysis to rule out other causes

PT, activated PTT, fibrinogen

Blood group and antibody screen, direct antiglobulin test, CMV serology

Consider CT/MRI brain, echocardiogram, ECG

Viral studies

Note: This disorder is usually associated with a severe drop in platelets and hemolysis/anemia precipitously

| Grading | Management |
|---|---|
| All grades | The first step in the management of TTP is a high index of suspicion for the diagnosis and timely recognition; hematology consult should immediately be called, as delay in identification is associated with increased mortality/morbidity. |
| | Initially, the patient should be stabilized and any critical organ dysfunction stabilized |
| G1: Evidence of RBC destruction (schistocytosis) without anemia, renal insufficiency, or thrombocytopenia clinically G2: Evidence of RBC destruction (schistocytosis) without clinical consequence with G2 anemia and thrombocytopenia | Hold ICPi and discuss resumption with patient only after taking into account the risks and benefits, noting that there are currently no data to recommend restarting ICPi therapy Hematology consult Administer 0.5-1 mg/kg/d prednisone |
| G3: Laboratory findings with clinical consequences (G3 thrombocytopenia, anemia, renal insufficiency > 2) G4: Life-threatening consequences (e.g, CNS hemorrhage or thrombosis/embolism or renal failure) | For G3: Hold ICPi and discuss resumption with patient only after taking into account the risks and benefits, noting that there are currently no data to recommend restarting ICPi therapy For G4: permanently discontinue ICPi Hematology consult |
| | In conjunction with hematology, initiate PEX according to existing guidelines with further PEX dependent on clinical progress |
| | Administer methylprednisolone 1 g IV daily for 3 days, with the first dose typically administered immediately after the first PEX |
| | May offer rituximab |
| | In case of management with rituximab, ICPi treatment will be discontinued |

### 8.0 Hematologic Toxicities

### 8.3 Hemolytic uremic syndrome

Definition: A disorder characterized by a form of thrombotic microangiopathy with renal failure, hemolytic anemia, and severe thrombocytopenia. Signs and symptoms of hemolytic uremic syndrome can include:

Bloody diarrhea

Decreased urination or blood in the urine

Abdominal pain, vomiting, and occasionally fever

Pallor

Small, unexplained bruises or bleeding from the nose and mouth Fatigue and irritability

Confusion or seizures

High blood pressure

Swelling of the face, hands, feet, or entire body

Diagnostic work-up

History and physical examination (special consideration for new history of high-risk drugs, hypertension, or cardiac causes) CBC with indices

Blood smear morphology. Note that the presence of schistocytes on smear is critical for diagnosis.

Serum creatinine

ADAMTS13 (to rule out TTP)

Homocysteine/methylmalonic acid

Complement testing C3, C4, CH50 (complement inhibitory antibodies for suspected familial)

Evaluate reticulocyte count and mean corpuscular volume

Evaluation of infectious cause, including screening for EBV, CMV, HHV6

Evaluation for nutritional causes of macrocytosis (B12 and folate)

Pancreatic enzymes

Evaluation for diarrheal causes, shiga toxin, Escherichia coli 0157, etc

Direct antibody test (Coombs test), haptoglobin, LDH, and other etiologies of anemia

Evaluation for common drugs causing hemolysis (tacrolimus, cyclosporine, sirolimus, etc)

Evaluation for concurrent confusion

| Grading | Management |
|---|---|
| G1-2: Evidence of RBC destruction (schistocytosis) without clinical consequences of anemia, thrombocytopenia Grade 2 | For G1 and G2: Continue ICPi with close clinical follow-<br>up and laboratory evaluation<br>Supportive care |
| G3: Laboratory findings with clinical consequences (e.g, renal insufficiency, petechiae) G4: Life-threatening consequences (e.g, CNS thrombosis/ embolism or renal failure) | For G3 and G4: Permanently discontinue ICPi Begin therapy with eculizumab therapy 900 mg weekly for four doses, 1,200 mg week 5, then 1,200 mg every 2 weeks Red blood transfusion according to existing guidelines |

### 8.4 Aplastic anemia

Definition: Condition in which the body stops producing enough new blood cells

Diagnostic work-up

History and physical examination (close attention to medications, exposure to radiation, toxins, recent viral infections) CBC, smear, reticulocyte count

Viral studies, including CMV, HHV6, EBV, parvovirus

Nutritional assessments including B12, folate, iron, copper, ceruloplasmin, vitamin D

Serum LDH, renal function

Work-up for infectious causes

Identify marrow hypo/aplasia

Bone marrow biopsy and aspirate analysis

Peripheral blood analysis, including neutrophil count, proportion of GPI-negative cells by flow for PNH

Flow cytometry to evaluate loss of GPI-anchored proteins



CONFIDENTIAL INFORMATION

| 8.0 Hematologic Toxicities | |
|---|---|
| Type and screen patient for transfusions and notify blood bank that all transfusions need to be irradiated and filtered | |
| Grading | Management |
| G1: Nonsevere, < 0.5 polymorphonuclear cells x 10 <sup>9</sup> /L hypocellular marrow, with marrow cellularity < 25%, peripheral platelet count > 20,000, reticulocyte count | Hold ICPi and provide growth factor support and close clinical follow-up, and laboratory evaluation |
| < 20,000 | Supportive transfusions as per local guidelines |
| G2: Severe, hypocellular marrow < 25% and two of the following: ANC < 500, peripheral platelet < 20,000, and reticulocyte < 20,000 | Hold ICPi and provide growth factor support and close clinical laboratory evaluations daily |
| | Administer ATG + cyclosporine; HLA typing and evaluation for bone marrow transplantation if patient is candidate; all blood products should be irradiated and filtered |
| | Supportive care with granulocyte colony-stimulating factor may be added in addition |
| G3-4: Very severe, ANC > 200, platelet count > 20,000, reticulocyte count > 20,000, plus hypocellular marrow > 25% | For G3: Hold ICPi and monitor weekly for improvement; if not resolved, discontinue treatment until AE has reverted to G1 |
| | For G4: permanently discontinue ICPi |
| | Hematology consult, growth factor support |
| | Horse ATG plus cyclosporine |
| | If no response, repeat immunosuppression with rabbit ATG plus cyclosporine, cyclophosphamide |
| | For refractory patients, consider eltrombopag plus supportive care |
| 8.5.1 vmphopenia | |

### 8.5 Lymphopenia

Definition: An abnormally low level of lymphocytes in PB; for adults, counts of < 1,500/mm<sup>3</sup>

### Diagnostic work-up

History and physical examination (special attention for lymphocyte-depleting therapy such as fludarabine, ATG, corticosteroids, cytotoxic chemotherapy, radiation exposure, etc, as well as history of autoimmune disease, family history of autoimmune disease) Evaluation of nutritional state as cause

### Spleen size

CBC with differential, peripheral smear and reticulocyte counts

CXR for evaluation of presence of thymoma

Bacterial cultures and evaluation for infection (fungal, viral, bacterial specifically CMV/HIV)

| Grading | Management |
|---|---|
| G1-2: 500-1,000 PB lymphocyte count | Continue ICPi for G1 to G2 |
| G3: 250-499 PB lymphocyte count<br>G4: < 250 PB lymphocyte count | For G3 single laboratory values out of normal range without any clinical correlates, hold treatment until resolution to G1 |
| | For G4, for single laboratory values out of normal range without any clinical correlates, permanent treatment discontinuation is not required. Treatment should be held until the etiology is determined. Permanent treatment discontinuation will only be required, if lymphopenia is considered of immune-related in nature, no clear alternative explanation exists for the event, and grade 4 lymphopenia does not resolve within 14 days. If the event is not considered immune-related and resolves to G $\leq$ 1 restarting treatment may be |
| | considered. |

| 8.0 Hematologic Toxicities | |
|---|---|
| | Check CBC weekly for monitoring, initiation of CMV screening Consider holding ICPi |
| | Initiate <i>Mycobacterium avium</i> complex prophylaxis and <i>Pneumocystis jirovecii</i> prophylaxis, CMV screening. HIV/hepatitis screening if not already done |
| | May consider EBV testing if evidence of lymphadenopathy/hepatitis, fevers, hemolysis consistent with lymphoproliferative disease. |

### 8.6 Immune thrombocytopenia

Definition: An autoimmune disorder characterized by immunologic destruction of otherwise normal platelets

Diagnostic work-up

History and physical examination (special attention for lymphocyte-depleting therapy, such as fludarabine, ATG, corticosteroids, cytotoxic therapy) Family history of autoimmunity or personal history of autoimmune disease History of viral illness

CBC

Peripheral blood smear, reticulocyte count

Bone marrow evaluation only if abnormalities in the above test results and further investigation is necessary for a diagnosis

Patients with newly diagnosed immune thrombocytopenia should undergo testing for HIV, hepatitis C virus, hepatitis B virus, and Helicobacter pylori Direct antigen test should be checked to rule out concurrent Evan syndrome

Nutritional evaluation

Bone marrow evaluation if other cell lines affected and concern for aplastic anemia

| Grading | Management |
|---|---|
| G1: Platelet count < 100/µL<br>G2: Platelet count < 75/µL | Continue ICPi with close clinical follow-up and laboratory evaluation |
| ' | Hold ICPi but monitor for improvement; if not resolved, interrupt treatment until AE has reverted to G1 |
| | Administer prednisone 1 mg/kg/d (dosage range, 0.5-2 mg/kg/d) orally for 2-4 weeks after which time this medication should be tapered over 4-6 weeks to the lowest effective dose IVIG may be used in conjunction with corticosteroids if a more-rapid increase in platelet count is required. |
| G3: Platelet count < 50/μL | Hold ICPi but monitor for improvement; if not resolved, interrupt treatment until AE has reverted to G1 |
| G4: Platelet count < 25/μL | Permanently discontinue ICPi |
| | Hematology consult |
| | Prednisone 1-2 mg/kg/d (oral or IV depending on symptoms) |
| | If worsening or no improvement, 1-2 mg/kg/d prednisone equivalents and permanently discontinue treatment |
| | IVIG used with corticosteroids when a more-rapid increase in platelet count is required |
| | If IVIG is used, the dose should initially be 1 g/kg as a one-time dose. This dosage may be repeated if necessary |

# 8.0 Hematologic Toxicities If previous treatment with corticosteroids and/or IVIG unsuccessful, subsequent treatment may include rituximab, thrombopoietin receptor agonists, or morepotent immunosuppression (From American Society of Hematology guideline on immune thrombocytopenia; consult for further details)

### 8.7 Acquired hemophilia

Definition: Disorder caused by the development of autoantibodies (inhibitors) directed against plasma coagulation factors

### Diagnostic work-up

Full blood count to assess platelet number, fibrinogen, PT, PTT, INR; the typical finding in patients with acquired hemophilia A is a prolonged activated PTT with a normal PT

MRI, CT, and ultrasonography may be indicated to localize, quantify, and serially monitor the location and response of bleeding Medication review to assess for alternative causes

Determination of Bethesda unit level of inhibitor

| Grading | Management |
|---|---|
| G1: Mild, 5%-40% of normal factor activity in blood, 0.05-0.4 IU/mL of whole blood | Hold ICPi and discuss resumption with patient only after taking into account the risks and benefits Administer 0.5-1 mg/kg/d prednisone Transfusion support as required Treatment of bleeding disorders with hematology consult |
| G2: Moderate, 1%-5% of normal factor activity in blood, 0.01- 0.05 IU/mL of whole blood | Hematology consult Administration of factor replacement (choice based on Bethesda unit of titer) Administer 1 mg/kg/d prednisone ± rituximab (dose, 375 mg/m² weekly for 4 weeks) and/or cyclophosphamide (dose, 1-2 mg/kg/d); choice of rituximab v cyclophosphamide is patient specific and should be done with assistance of hematology consult; prednisone, rituximab, and cyclophosphamide should be given for at least 5 weeks Factors should be provided to increase level during bleeding episodes, with choice of factor based on presence or absence of inhibitor |
| G3-4: Severe, < 1% of normal factor activity in blood, < 0.01 IU/mL of whole blood | Permanently discontinue ICPi Admit patient Hematology consult Administration of factor replacement, choice based on Bethesda unit level of inhibitor Bypassing agents may be used (factor VII, factor VIII inhibitor bypass activity); caution should be taken in the elderly and those with coronary artery disease Prednisone 1-2 mg/kg/d (oral or IV depending on symptoms) ± rituximab (dose, 375 mg/m² weekly for 4 weeks) and/or cyclophosphamide (dose, 1-2 mg/kg/d). Transfusion support as required for bleeding If worsening or no improvement add cyclosporine or immunosuppression/immunoadsorption |

CCI CCI

established.

Consult and/or transfer to a specialist center is often appropriate. If consultation with or transfer to a hemophilia center is not immediately possible, then investigation and treatment should be initiated while a liaison is being

### 8.0 Hematologic Toxicities

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate.

Abbreviations: AE, adverse event; ANC, absolute neutrophil count; ATG, antithymocyte globulin; CBC, complete blood count; CMV, cytomegalovirus; CNS, central nervous system; CT, computed tomography; CXR, chest x-ray; DIC, disseminated intravascular coagulation; EBV, Epstein-Barr virus; ECG, electrocardiogram; ER, extended release; FE, ferritin; G, Grade; GPI, glycosylphosphatidylinositol; Hgb, hemoglobin; HHV6, human herpesvirus 6; HIV, human immunodeficiency virus; HLA, human leukocyte antigen; ICPi, immune checkpoint inhibitor; INR, international normalized ratio; irAE, immune-related adverse event; IV, intravenous; IVIG, intravenous immunoglobulin; LDH, lactate dehydrogenase; LLN, lower limit of normal; MRI, magnetic resonance imaging; NSAID, nonsteroidal anti-inflammatory drug; PB, peripheral blood; PEX, plasma ex-change; PNH, paroxysmal nocturnal hemoglobinuria; PT, prothrombin time; PTT, partial thromboplastin time; RBC, red blood cell; TTP, thrombotic thrombocytopenic purpura.

### Table A9 Management of Cardiovascular irAEs in Patients Treated With ICPis

### 9.0 Cardiovascular Toxicities

### 9.1 Myocarditis, pericarditis, arrhythmias, impaired ventricular function with heart failure and vasculitis

Definition: Signs and symptoms may include chest pain, arrhythmia, palpitations, peripheral edema, progressive or acute dyspnea, pleural effusion, fatigue

Diagnostic work-up

At baseline

**ECG** 

Consider troponin, especially in patient treated with combination immune therapies Upon signs/symptoms (consider cardiology consult)

**ECG** 

Troponin

BNP Echocardiogram CXR

Additional testing to be guided by cardiology and may include

Stress test

Cardiac catherization Cardiac MRI

| Grading | Management |
|---|---|
| G1: Abnormal cardiac biomarker testing, including abnormal ECG | All grades warrant work-up and intervention given potential for cardiac compromise |
| G2: Abnormal screening tests with mild symptoms | Consider the following: |
| G3: Moderately abnormal testing or symptoms with mild | For G1: Hold ICPi |
| activity | For G2, G3, and G4: Permanently discontinue ICPi |
| G4: Moderate to severe decompensation, IV medication or intervention required, life-threatening conditions | For G1-G4: High-dose corticosteroids (1-2 mg/kg of prednisone) initiated rapidly (oral or IV depending on symptoms) |
| | Admit patient, cardiology consultation |
| | Immediate transfer to a coronary care unit for patients with elevated troponin or conduction abnormalities |
| | In patients without an immediate response to high-dose corticosteroids, consider early institution of cardiac transplant rejection doses of corticosteroids (methylprednisolone 1 g every day) and the addition of either mycophenolate, infliximab, or antithymocyte globulin |

Qualifying statement: Treatment recommendations are based on anecdotal evidence and the life-threatening nature of cardiovascular complications. The appropriateness of rechallenging remains unknown. Note that infliximab has been associated with heart failure and is contraindicated at high doses in patients with moderate-severe heart failure.

### 9.2 Venous thromboembolism

Definition: A disorder characterized by occlusion of a vessel by a thrombus that has migrated from a distal site via the blood stream. Clinical signs and symptoms are variable and may include pain, swelling, increased skin vein visibility, erythema, and cyanosis accompanied by unexplained fever for DVT and dyspnea, pleuritic pain, cough, wheezing, or hemoptysis for PE

Diagnostic work-up

Evaluation of signs and symptoms of PE or DVT may include Clinical prediction rule to stratify patients with suspected venous thromboembolism Venous ultrasound for suspected DVT

CTPA for suspected PE

Can also consider D-dimer for low-risk patients based on risk stratification by clinical prediction rule for DVT/PE when CT or Doppler are not available or appropriate Ventilation/perfusion scan is also an option when CTPA is not appropriate

Consider other testing, including ECG, CXR, BNP and troponin levels, and arterial blood gas

| 9.0 Cardiovascular Toxicities | |
|---|---|
| Grading | Management |
| G1: Venous thrombosis (e.g, superficial thrombosis) | Continue ICPi |
| | Warm compress |
| | Clinical surveillance |
| G2: Venous thrombosis (e.g, uncomplicated DVT), medical intervention indicated | Hold ICPi until AE reverts back to G1 or less. If reverts to G2, use benefit-risk assessment for ICPi continuation |
| G3: Thrombosis (e.g, uncomplicated PE [venous], nonembolic cardiac mural [arterial] thrombus), medical intervention indicated | Consider consult from cardiology or other relevant specialties |
| | LMWH is suggested over VKA, dabigatran, rivaroxaban apixaban, or edoxaban for initial and long-term treatment |
| | IV heparin is an acceptable alternative for initial use, and oral anticoagulants are acceptable for the long term |
| G4: Life-threatening (e.g, PE, cerebrovascular event, | Permanently discontinue ICPi |
| arterial insufficiency), hemodynamic or neurologic instability, urgent intervention indicated | Admit patient and management according to CHEST, ACC, and/or AHA guidelines and with guidance from cardiology |
| | Respiratory and hemodynamic support |
| | LMWH is suggested over VKA, dabigatran, rivaroxaban, apixaban, or edoxaban for initial and long-term treatment |
| | IV heparin is an acceptable alternative for initial use, and oral anticoagulants are acceptable for the long term |
| | Further clinical management as indicated based on symptoms |

### Additional considerations

While it may be impossible to determine the etiology of thromboembolic disease in patients with advanced cancer and the role, if any, that ICPi treatment plays, it is reasonable to remove the potential inciting agents given the severity and life-threatening potential of G4 complications. Clinicians are to use clinical judgment and take into account the risks and benefits when deciding whether to discontinue ICPi treatment.

Anticoagulant therapy duration should continue for a minimum of 9-12 months to indefinitely in the setting of active cancer unless patient is asymptomatic, doing well, or in remission.

All recommendations are expert consensus based, with benefits outweighing harms, and strength of recommendations are moderate.

Abbreviations: BNP, brain natriuretic peptide; CT, computed tomography; CTPA, computed tomography pulmonary angiography; CXR, chest x-ray; DVT, deep vein thrombosis; ECG, electrocardiogram; G, Grade; ICPi, immune checkpoint inhibitor; irAE, immune-related adverse event; IV, intravenous; LMWH, low-molecular-weight heparin; MRI, magnetic resonance imaging; PE, pulmonary embolism; VKA, vitamin K agonist.



### Table A10 Management of Ocular irAEs in Patients Treated With ICPis

### 10.0 Ocular Toxicities

Counsel all patients to inform their health care provider immediately if they experience any of the following ocular symptoms

Blurred vision

Change in color vision Photophobia

Distortion

Scotomas

Visual field changes Double vision Tenderness

Pain with eye movement Eyelid swelling Proptosis

Evaluation, under the guidance of ophthalmology

Check vision in each eye separately

Color vision

Red reflex

Pupil size, shape, and reactivity

Fundoscopic examination

Inspection of anterior part of eye with penlight

Prior conditions

Exclude patients with history of active uveitis

History of recurrent uveitis requiring systemic immunosuppression or continuous local therapy

Additional considerations

Ocular irAEs are many times seen in the context of other organ irAEs

High level of clinical suspicion as symptoms may not always be associated with severity Best to treat after ophthalmologist eye examination

### 10.1 Uveitis/iritis

Definition: Inflammation of the middle layer of the eye Diagnostic work-up: as per above

| ļ | · · · |
|---|---|
| Grading | Management |
| G1: Asymptomatic | Continue ICPi Refer to ophthalmology within 1 week Artificial tears |
| G2: Medical intervention required, anterior uveitis | Hold ICPi temporarily until after ophthalmology consult Urgent ophthalmology referral Topical corticosteroids, cycloplegic agents, systemic corticosteroids May resume ICPi treatment once off systemic corticosteroids, which are purely indicated for ocular adverse effects or once corticosteroids for other concurrent systemic irAEs are reduced to ≤ 10 mg; continued topical/ocular corticosteroids are permitted when resuming therapy to manage and minimize local toxicity Re-treat after return to G1 or less |
| G3: Posterior or panuveitis | Permanently discontinue ICPi Urgent ophthalmology referral. Systemic corticosteroids and intravitreal/periocular/topical corticosteroids |
| G4: 20/200 or worse | Permanently discontinue ICPi<br>Emergent ophthalmology referral |

CONFIDENTIAL INFORMATION

| 10.0 Ocu | ılar Toxicities |
|---|---|
| | Systemic corticosteroids (IV prednisone 1-2 mg/kg or methylprednisolone 0.8-1.6 mg/kg) and intravitreal/periocular/topical corticosteroids per ophthalmologist opinion |
| Additional considerations: Consider use of infliximab or refractory to standard treatment | other TNF-α blockers in cases that are severe and |
| 10.2 Episcleritis | |
| Definition: Inflammatory condition affecting the episcler in the absence of an infection Diagnostic work-up: As p | al tissue between the conjunctiva and the sclera that occurs er 10.0 |
| Grading | Management |
| G1: Asymptomatic | Continue ICPi Refer to ophthalmology within 1 week Artificial tears |
| G2: Vision 20/40 or better | Hold ICPi therapy temporarily until after ophthalmology consult Urgent ophthalmology referral Topical corticosteroids, cycloplegic agents, systemic corticosteroids |
| G3: Symptomatic and vision worse than 2/40 | Permanently discontinue ICPi Urgent ophthalmology referral. Systemic corticosteroids and topical corticosteroids with cycloplegic agents |
| G4: 20/200 or worse | Permanently discontinue ICPi Emergent ophthalmology referral. Systemic corticosteroids and topical corticosteroids with cycloplegic agents |
| Additional considerations: Consider use of infliximab or refractory to standard treatment | other TNF-α blockers in cases that are severe and |
| 10.3 Blepharitis | |
| Definition: Inflammation of the eyelid that affects the ey | elashes or tear production Diagnostic work-up: As per 10.0 |
| Grading | Management |
| No formal grading system | Warm compresses and lubrication drops Continue therapy unless persistent and serious |
| All recommendations are expert consensus based, with recommendations are moderate. | n benefits outweighing harms, and strength of |

Abbreviations: ICPi, immune checkpoint inhibitor; G, Grade; irAE, immune-related adverse event; IV, intravenous, TNF, tumor necrosis factor.

# **Appendix 6** Clinical Laboratory Tests

Table 13 Protocol-Required Clinical Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | | |
|---|---|---|---|---|
| Hematology | Platelet count <sup>d</sup> | | Mean Corpuscular<br>Volume (MCV) | White blood cell (WBC) Count with Differential <sup>d</sup> : |
| | Reticulocytes ( | %) | Mean corpuscular hemoglobin concentration (MCHC) | <ul><li>Neutrophils</li><li>Lymphocytes</li><li>Monocytes</li></ul> |
| | Hemoglobind | | Mean corpuscular hemoglobin (MCH) | Eosinophils Basophils |
| | Hematocrit | | Activated partial thromboplastin time (aPTT) <sup>a</sup> | |
| | Red blood cell of | count <sup>d</sup> | Prothrombin time <sup>a</sup> | |
| | Absolute lymphocyte count <sup>d</sup> | | International normalized ratio (INR) <sup>a</sup> | |
| | Absolute neutrophil countd | | | |
| Biochemistry | Blood Urea<br>Nitrogen/Total<br>urea | Potassium | Aspartate<br>Aminotransferase <sup>d</sup> | Bilirubin (total, indirect/direct) <sup>d</sup> |
| | Creatinined | Sodium | Alanine<br>Aminotransferase <sup>d</sup> | Total Protein |
| | Glucose | Calcium | Alkaline phosphatase | Tuberculin skin test,<br>QuantiFERON-TB-Gold,<br>or T-SPOT (if positive<br>history of tuberculosis<br>exposure) |
| | Lipase | Chloride | Albumin | Lactate dehydrogenase (LDH) |
| | C-reactive protein | Amylase | | |
| Routine Urinalysis | Dipstick plus microscopic evaluation. Dipstick, including physical appearance, bilirubin, blood, color, glucose, ketones, leukocyte esterase, nitrite, pH, protein, specific gravity, urobilinogen, as locally available | | | |
| Other Screening<br>Tests | <ul> <li>FSH and estradiol (as needed if <b>not</b> a WOCBP only)</li> <li>Serum or highly sensitive urine β-hCG pregnancy test</li> <li>Free T4 and TSH</li> </ul> | | | |
| | Hepatitis Screening <sup>b</sup> : Hepatitis B surface antigen; Hepatitis B core antibody and Hepatitis C antibody | | | · |
| 20 15 | HIV; HIV virus RNA, quantitative; and CD4 lymphocyte count <sup>c</sup> | | | |

<sup>&</sup>lt;sup>a</sup> Coagulation parameters collected at baseline and as clinically indicated, thereafter (See Table 1).

<sup>&</sup>lt;sup>c</sup> Not required for all participants. Testing required for participants with known history of HIV. Participants must be adequately consented per local regulations for any HIV-related testing.



<sup>&</sup>lt;sup>b</sup> If hepatitis B surface antigen positive and hepatitis B core antibody positive, then reflex to quantitative HBV DNA (PCR); if hepatitis B core antibody positive alone, then reflex to quantitative hepatitis B DNA (PCR); if hepatitis C antibody positive, then reflex to quantitative hepatitis C RNA (PCR).

# Bintrafusp alfa (M7824) MS200647\_0020

# Bintrafusp alfa in HMGA2-expressing Triple Negative Breast Cancer

| Laboratory<br>Assessments | Parameters |
|---|---|
| d Results must be review | ewed by the Investigator within 3 days prior to dosing. |

# **Appendix 7** Prohibited Traditional Chinese Medicines

### Name of Traditional Chinese Medicine with Anticancer Indication

| | CCI | English |
|----|-----|------------------------------------------------------------------|
| 1 | CCI | Ai Di injection® |
| 2 | | De Li Shen, Delisheng, injection |
| 3 | | Kanglaite injection, or KLT |
| 4 | | Ganfule, Gan Fu Le, GanFuLe tablet/capsules |
| 5 | | Huaier, Huaier Keli, granules |
| 6 | | Jinlong capsules |
| 7 | | Cinobufacini injection |
| 8 | | Jiedu Granules |
| 9 | | Elemene injection, Elemenum emulsion, Injectio Emulsioni Elemeni |
| 10 | | Xiaoaiping tablets |
| 11 | | Chloroxoquinoline capsules |
| 12 | | Kanglixin capsules |
| 13 | | Kanglixin tablets |
| 14 | | Sodium Cantharidinate For Injection |
| 15 | | compound capsules cantharidin |
| 16 | | Java brucea fruit oil emulsion |
| 17 | | Java brucea fruit oil capsules |
| 18 | | Java brucea fruit oil injection |
| 19 | | Weimaining capsules |
| 20 | | Shenyi Capsule |
| 21 | | Shelian capsule |
| 22 | | Kangai injection |
| 23 | | Ubenimex |
| 24 | | Xianchan tablet |
| | | Immune Treatment |
| 1 | | Interleukin-2 |
| 2 | | interferon |
| 3 | | Thymosin/thymopentin |

## **Appendix 8** Pharmacogenetics

## Use/Analysis of Deoxyribonucleic acid (DNA)

Genetic variation may impact a participant's response to therapy, susceptibility to, and severity and progression of disease. Variable response to therapy may be due to genetic determinants that impact study intervention absorption, distribution, metabolism, and excretion; mechanism of action of the study intervention; disease etiology; and/or molecular subtype of the disease being treated.

DNA samples will be analyzed for genetic research. Additional analyses may be conducted if it is hypothesized that this may help further understand the clinical data.

In addition, DNA samples will be used for research related to bintrafusp alfa or TNBC. They may also be used to develop tests or assays, including diagnostic tests related to bintrafusp alfa and/or treatments of this drug class and TNBC. Pharmacogenetic research may consist of the analysis of one or more candidate genes or the analysis of genetic markers throughout the genome (as appropriate).

The results of pharmacogenetic analyses may be reported in the CSR or in a separate study summary.

Details on processes for collection and shipment of these samples can be found in the Laboratory Manual. The Sponsor will store the DNA samples in a secure storage space with adequate measures to protect confidentiality.

Retention time and possible analysis of DNA sample after the study ends are specified in the respective ICF.

# **Appendix 9** Protocol Amendment History

The information for the current amendment is on the title page.

# **Appendix 10 Sponsor Signature Page**

Study Title: A Phase II, Multicenter, Open Label Study of Bintrafusp

alfa (M7824) Monotherapy in Participants with

HMGA2-expressing Triple Negative Breast Cancer

Regulatory Agency Identifying

**Numbers:** 

CCI

, EudraCT: 2019-004833-18

Clinical Study Protocol Version: 06 July 2021/Version 2.0

I approve the design of the clinical study:

PPD PPD PPD

Signature Date of Signature

Name, academic degree: PPD , PPD

Function/Title: PPD

**Institution:** EMD Serono Research & Development Institute, Inc.

**Address:** 45A Middlesex Turnpike

Billerica, MA 01821, USA

Telephone number:

Fax number:

**E-mail address:** laureen.ojalvo@emdserono.com

# Appendix 11 Coordinating Investigator Signature Page

| Study Title: | A Phase II, Multicenter, | Open Label | Study of Bintrafusp |
|--------------|--------------------------|------------|---------------------|
|--------------|--------------------------|------------|---------------------|

alfa (M7824) Monotherapy in Participants

HMGA2-expressing Triple Negative Breast Cancer

Regulatory Agency Identifying

EudraCT: 2019-004833-18

Numbers:

**Clinical Study Protocol Version:** 

06 July 2021/Version 2.0

**Site Number:** 

I approve the design of the clinical study, am responsible for the conduct of the study at this site and understand and will conduct it per the clinical study protocol, any approved protocol amendments, International Council for Harmonisation Good Clinical Practice (Topic E6) and all applicable Health Authority requirements and national laws.

| PD | | | | | |
|---|---|---|---|---|---|
| Signature | | <u> </u> | Date of | Signature | 1 |
| Name, academic degree: Function/Title: Institution: | PPD<br>PPD | PPD | | | |
| Address: Telephone number: | PPD | | | | |
| Fax number: E-mail address: | | | | | |

# **Appendix 12 Principal Investigator Signature Page**

| Study Title: | A Phase II, Multicenter, Open Label Study of Bintrafusp alfa (M7824) Monotherapy in Participants with |
|---|---|
| | HMGA2-expressing Triple Negative Breast Cancer |
| Regulatory Agency Identifying Numbers: | EudraCT: 2019-004833-18 |
| <b>Clinical Study Protocol Version:</b> | 06 July 2021/Version 2.0 |
| Site Number: | |
| clinical study protocol, any appro | e study at this site and understand and will conduct it per the oved protocol amendments, International Council for ctice (Topic E6) and all applicable Health Authority |
| supply details about ownership interest<br>any other financial ties with the Sport<br>complying with the regulatory requirencessary information regarding ownership. | ies may require the Sponsors of clinical studies to obtain and sts in the Sponsor or Investigational Medicinal Product and nsor. The Sponsor will use any such information solely for ements. Therefore, I agree to supply the Sponsor with any ership interest and financial ties including those of my spouse rovide updates as necessary to meet Health Authority |
| Signature | Date of Signature |
| Name, academic degree: | |
| Function/Title: | |
| Institution: | |
| Address: | |
| Telephone number: | |
| Fax number: | |

E-mail address: